CLINICAL TRIAL: NCT01039688
Title: Phase 3 Randomized, Double-blind Study Of The Efficacy And Safety Of 2 Doses Of Cp-690,550 Compared To Methotrexate In Methotrexate Navie Patients With Rheumatoid Arthritis
Brief Title: Comparing The Effectiveness And Safety Of 2 Doses Of An Experimental Drug, CP-690,550, To Methotrexate (MTX) In Patients With Rheumatoid Arthritis Who Have Not Previously Received MTX
Acronym: ORAL1069
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921069; 2009-016987-34 (EudraCT Number)
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: oral JAK inhibitor; MTX; DMARD; clinical trial; joint diseases; autoimmune diseases; anti-Inflammatory agents; rheumatic diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Joint Diseases; Autoimmune Diseases; Rheumatic Diseases | interventions — tofacitinib; Antirheumatic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 5 mg BID CP-690,550 (Experimental)
  Interventions: Drug: CP-690,550
- 10 mg BID CP-690,550 (Experimental)
  Interventions: Drug: CP-690,550
- methotrexate (Active Comparator)
  Interventions: Drug: Disease-modifying antirheumatic drug

INTERVENTIONS:
Drug: CP-690,550 — Oral tablets administered at a dose of 5 mg BID for 24 months
  Arms: 5 mg BID CP-690,550
Drug: CP-690,550 — Oral tablets administered at a dose of 10 mg BID for 24 months
  Arms: 10 mg BID CP-690,550
Drug: Disease-modifying antirheumatic drug — Oral capsules,administered as 10 mg per week for 4 weeks titrated to 15 mg per week for 4 weeks, then titrated to 20 mg week for 24 months
  Other Names: DMARD, MTX
  Arms: methotrexate

SUMMARY:
This study is designed to compare the effectiveness of the experimental drug, CP-690,550, to methotrexate in preventing joint damage and improving symptoms of rheumatoid arthritis. This study will also compare the safety of CP-690,550 with methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Adults with moderate to severe RA (Rheumatoid Arthritis) who have not been treated with methotrexate.
* Diagnosis of RA based on the American College of Rheumatology 1987 revised criteria.
* Active disease as defined by both >=6 tender or painful joints on motion and >= 6 joints swollen; and either an erythrocyte sedimentation rate (ESR) > 28 mm or a C-reactive protein (CRP) concentration > 7 mg/dL

Exclusion Criteria:

* Blood dyscrasias including confirmed: Hemoglobin <9 g/dL or Hematocrit <30%; White blood cell count <3.0 x 109/L; Absolute neutrophil count <1.2 x 109/L; Platelet count <100 x 109/L
* History of any other rheumatic autoimmune disease other than Sjogren's syndrome
* No malignancy or history of malignancy
* History of infection requiring hospitalization, parenteral antimicrobial therapy, or as otherwise judged clinically significant by the investigator, within the 6 months prior to the first dose of study drug
* No chronic liver disease, recent or active hepatitis or other contraindication to methotrexate therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 956 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (174):
- United States (40):
  - Catalina Pointe Clinical Research, Inc., Tucson, Arizona
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - University of California San Diego Perlman Ambulatory Clinic, La Jolla, California
  - University of California San Diego Center for Innovative Therapy, La Jolla, California
  - Keck Hospital of USC, Lower Level Pharmacy, Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - USC Keck School of Medicine, Los Angeles, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Southeastern Arthritis Center, Gainesville, Florida
  - Southeastern Imaging and Diagnostics, Gainesville, Florida
  - Southeastern Integrated Medical, PL dba Florida Medical Research, Gainesville, Florida
  - Center for Arthritis and Rheumatic Diseases, Miami, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - Bernard F. Germain, MD, Tampa, Florida
  - Burnette & Silverfield, MDS PLC, Tampa, Florida
  - Diagnostic Rheumatology and Research, PC, Indianapolis, Indiana
  - Medical Associates Clinic, PC, Dubuque, Iowa
  - Louisiana State University Health Sciences, New Orleans, Louisiana
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - The Center for Rheumatology, Albany, New York
  - AAIR Research Center, Rochester, New York
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLP, Wyomissing, Pennsylvania
  - Medical University of South Carolina - Rheumatology, Charleston, South Carolina
  - Medical University of South Carolina Investigational Drug Services, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Arthritis Clinic, Jackson, Tennessee
  - West Tennessee Research Institute, Jackson, Tennessee
  - Austin Rheumatology Research, Austin, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - University of North Texas Health Science Center at Fort Worth, Fort Worth, Texas
  - Investigational Drug Service, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Mountain State Clinical Research, Clarksburg, West Virginia
  - United Hospital Center (Imaging Only), Clarksburg, West Virginia
- Argentina (3):
  - OMI - Organización Médica de Investigación, Buenos Aires
  - Saint Dennis Medical Group S.A., Buenos Aires
  - Consultorios Reumatológicos Pampa, Buenos Aires
- Australia (3):
  - Rheumatology Research Unit Sunshine Coast, Maroochydore, Queensland
  - The Queen Elizabeth Hospital, Department of Rheumatology, Woodville, South Australia
  - Emeritus Research, Malvern East, Victoria
- Universitair Ziekenhuis Gent - Reumatologie, Ghent, Belgium
- Brazil (6):
  - CIP - Centro Internacional de Pesquisas, Goiânia, Goiás
  - Clinica de Raios X Nabyh Salum S/S - Clinica Sao Matheus, Goiânia, Goiás
  - Centro de Estudos em Terapias Inovadoras, Curitiba, Paraná
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - CEPIC - Centro Paulista de Investigacao Clinica e Servicos Medicos Ltda, São Paulo, São Paulo
  - CCBR Brasil Centro de Pesquisas e Analises Clinicas Ltda, Rio de Janeiro
- Bulgaria (6):
  - Revmatologichno Otdelenie, MBAL - Plovdiv, Plovdiv
  - MBAL-Ruse, AD, IV Terapevtichno i kardiologichno otdelenie, Rousse
  - MBAL na Voennomeditsinska Akademia - Sofia, Klinika po Revmatologia i Kardiologia, Sofia
  - MBAL Sveti Ivan Rilski Sofia; Klinika po Revmatologia, Sofia
  - DKTs "Sveta Anna", Sofia; Konsultativen kabinet po Revmatologia, Sofia
  - MOBAL "D-r Stefan Cherkezov" AD, Revmokardiologichno otdelenie s intenziven sektor, Veliko Tarnovo
- Canada (12):
  - Rheumatology Research Associates Ltd., Edmonton, Alberta
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
  - Manitoba Clinic, Winnipeg, Manitoba
  - Burlington Rheumatology and Osteoporosis Clinic, Burlington, Ontario
  - Dr. William G. Bensen Medicine Professional Corporation, Hamilton, Ontario
  - Office of Dr. Fernando Bianchi, Hamilton, Ontario
  - MAC Research Inc., Hamilton, Ontario
  - KW Musculoskeletal Research Inc., Kitchener, Ontario
  - Rheumatology Research Associates, Ottawa, Ontario
  - Niagara Peninsula Arthritis Centre, St. Catharines, Ontario
  - Windsor Radiological Associates, Windsor, Ontario
  - Clinical Research and Arthritis Centre, Windsor, Ontario
- Chile (5):
  - Consulta Privada Dra. Lucia Ponce, Temuco, Región de la Araucanía
  - Estudios Clinicos V Region, Viña del Mar, Región de Valparaíso
  - Centro de Estudios Reumatologicos, Santiago, RM
  - Consulta Privada Dra. Marta Aliste, Santiago, RM
  - Hospital Regional de Rancagua, Rancagua
- Colombia (3):
  - Centro de Reumatologia y Ortopedia, Barranquilla, Atlántico
  - Centro Integral de Reumatologia e Inmunologia CIREI, Bogota, Cundinamarca
  - Servimed E.U, Bucaramanga, Santander Department
- Costa Rica (2):
  - Centro de Reumatología y Osteoporosis, Cartago, Cartago
  - Hospital Cima San Jose, San José
- Czechia (6):
  - Fakultni nemocnice Brno, Brno
  - Revmacentrum MUDr. Mostera, s.r.o., Brno-Židenice
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Revmatologicka ambulance, Ostrava-Poruba
  - Revmatologicky ustav, Prague
  - Revmatologicka ambulance, Prague
- Patricia Alvarez Site, Santo Domingo, Dominican Republic
- Germany (8):
  - Privat-Praxis, Rheumatologie (P515), Aachen
  - Schlosspark-Klinik, Berlin
  - Studienambulanz, Medizinische Klinik 3 Universitaetsklinikum Erlangen, Erlangen
  - Schwerpunktpraxis Rheumatologie FAE Innere Medizin, Halle
  - Schoen Klinik Hamburg-Eilbek, Abt. Rheumatologie und Klin. Immunologie, Hamburg
  - Arztpraxis, Internist - Rheumatologie, Nuremberg
  - Rheumaforschung - Studienambulanz Dr. Wassenberg, Ratingen
  - Schwerpunktpraxis fuer Rheumatologie, Rheine
- Hungary (5):
  - Drug Research Center Kft. Reumatologiai Szakrendeles, Balatonfüred
  - Revita Reumatologiai Rendelo, Budapest
  - Synexus Magyarorszag Kft., Budapest
  - Mozgasszervi Rehabilitacios Kozpont, Reumatologiai szakrendeles, Mezőkövesd
  - MAV Korhaz es Rendelointezet, Szolnok
- India (7):
  - Mahavir Hospital & Research Center, Hyderabad, Andhra Pradesh
  - Department of Rheumatology, Secunderabad, Andhra Pradesh
  - Rheumatic Disease Clinic, Ahmedabad, Gujarat
  - Shirdi Sai Hospital, Bangalore, Karnataka
  - Arthritis Research and Care Foundation, Pune, Maharashtra
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune, Maharashtra
  - Shalby Hospital, Ahmedabad
- Malaysia (3):
  - Hospital Tuanku Ja'afar, Seremban, Negeri Sembilan
  - Sunway Medical Centre, Petaling Jaya, Selangor
  - Sarawak General Hospital, Kuching
- Mexico (4):
  - Unidad de Enfermedades Reumaticas y Cronico Degenerativas SC, Torreón, Coahuila
  - Instituto Jaliscience de Investigación Clínica SA de CV, Guadalajara, Jalisco
  - Unidad de Investigacion en Enfermedades Cronico Degenerativas, Guadalajara, Jalisco
  - Hospital Universitario Jose Eleuterio Gonzalez, Monterrey, Nuevo León
- New Zealand (4):
  - Centre for Clinical Research and Effective Practice (CCREP Middlemore Hospital, Otahuhu, Auckland
  - The Canterbury Geriatric Medical Research Trust, c/- The Princess Margaret Hospital, Christchurch
  - Ryburns Building, Waikato Hospital, Hamilton
  - Timaru Hospital, Clinical Trials Unit, Timaru
- Peru (4):
  - Hospital Nacional IV Alberto Sabogal Sologuren, Callao
  - Clinica Anglo Americana, Lima
  - Centro Medico Corpac, Lima
  - Instituto Peruano del Hueso y la Articulacion SAC-Privado-Lima/Centro de Investigacion IPHAR, Lima
- Philippines (3):
  - Chong Hua Hospital, Cebu City
  - Brokenshire Integrated Health Ministries, Inc. Brokenshire Memorial Hospital, Davao City
  - Rayuma Klinik, OPD Department, Jose R. Reyes Memorial Medical Center, Manila
- Poland (5):
  - Przychodnia Medyczna Lekarskiej Spoldzielni Pracy, Gdynia
  - Centrum Leczenia Chorob Cywilizacyjnych Sp. z.o.o. SKA Oddzial Gdynia, Gdynia
  - Centrum Leczenia Chorob Cywilizacyjnych Sp. z o.o. SKA Oddzial Katowice, Katowice
  - Synexus SCM Sp. z o.o. Oddzial Warszawa, Warsaw
  - Rheuma Medicus - Specjalistyczne Centrum Reumatologii i Osteoporozy, Warsaw
- Puerto Rico (2):
  - Ponce School of Medicine, Ponce
  - Edificio Parra, Ponce
- Russia (14):
  - State Healthcare Institution Regional Clinical Hospital, Barnaul
  - State Healthcare Institution Regional Clinical Hospital for War Veterans, Kemerovo
  - Federal State Institution named after Academician E.N. Meshalkin, Novosibirsk State Research, Novosibirsk
  - Scientific Research Institute of Clinical and Experimental Lymphology of the Siberian Branch of RAMS, Novosibirsk
  - State Health Institution City Hospital # 25, City Rheumatology Center of St. Petersburg, Saint Petersburg
  - Clinical Hospital #122 named after L.G. Sokolov of the Federal Medical-Biological Agency, Saint Petersburg
  - Almazov Federal Heart, Blood and Endocrinology Centre, Saint Petersburg
  - State Healthcare Institution City Hospital # 40 of Administrative Health Resort District, Saint Petersburg
  - St. Petersburg State Institution of Healthcare Consultative-diagnostic Center #85, Saint Petersburg
  - Smolensk State Medical Academy, Clinical Research Centre of Diagnostic Medicine and Drugs, Smolensk
  - Regional State Healthcare Institution of Tomsk Regional Clinical Hospital, Tomsk
  - State Healthcare Institution, Yekaterinburg
  - Ltd. Medical Association "Novaya Bolnitsa" (X-Ray Only), Yekaterinburg
  - State Educational Institution of Higher Professional Education, Yekaterinburg
- Slovakia (5):
  - Reumatolog s.r.o., Bratislava
  - AAGS, s.r.o. , nestatne zdravotnicke zariadenie, Dunajská Streda
  - Reumatologicka ambulancia, Ecclesia, s.r.o., Nové Zámky
  - Narodny ustav reumatickych chorob, Piešťany
  - Nestatna reumatologicka ambulancia, Žilina
- South Korea (3):
  - Seoul National University Hospital, Rheumatology, Internal Medicine, Seoul
  - Yonsei University College of Medicine, Severance Hospital, Rheumatology, Internal Medicine, Seoul
  - Asan Medical Center, Rheumatology, Internal Medicine, Seoul
- Spain (5):
  - Hospital Nuestra Señora de La Esperanza, Santiago de Compostela, A Coruña
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Civil. Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen Macarena, Seville
- Sweden (3):
  - Skanes Universitetssjukhus i Malmo, Malmo
  - Sundsvalls sjukhus- Medicinkliniken, Sundsvall
  - Akademiska sjukhuset, Reumatologmottagningen, Uppsala
- Taiwan (3):
  - Chung-Ho Memorial Hospital, Kaohsiung Medical University, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
- Thailand (3):
  - Rheumatology Unit, Department of Internal Medicine, Phramongkutklao Hospital, Phayathai, Bangkok
  - Rheumatology Unit, Department of Internal Medicine, Rajavithi Hospital, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok
- Ukraine (5):
  - CRI "Clinical Territorial Medical Association "University Clinic", Department of Rheumatology, Simferopol, Autonomous Republic of Crimea
  - State Institution "Republican Clinical Hospital of the Ministry of Health of Ukraine", Kyiv
  - Municipal City Clinical Hospital #4, Department of Rheumatology, Lviv
  - Municipal Establishment "City Clinical Hospital #9 n.a. O.I. Minakov", Department of Rheumatology, Odesa
  - Vinnitsa Regional Clinical Hospital n.a. M.I. Pirogov, Vinnitsa

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Pope J, Finckh A, Silva-Fernandez L, Mandl P, Fan H, Rivas JL, Valderrama M, Montoro M. Tofacitinib Monotherapy in Rheumatoid Arthritis: Clinical Trials and Real-World Data Contextualization of Patients, Efficacy, and Treatment Retention. Open Access Rheumatol. 2024 Jun 11;16:115-126. doi: 10.2147/OARRR.S446431. eCollection 2024. PMID 38883150
- [Derived] Ciurea A, Distler O, Kwok K, Jo H, Wang L, Killeen T, Ospelt C, Frank Bertoncelj M. Joint-level responses to tofacitinib and methotrexate: a post hoc analysis of data from ORAL Start. Arthritis Res Ther. 2023 Sep 29;25(1):185. doi: 10.1186/s13075-023-03144-1. PMID 37773189
- [Derived] Charles-Schoeman C, Hyde C, Guan S, Parikh N, Wang J, Shahbazian A, Stockert L, Andrews J. Relationship Between Paraoxonase-1 Genotype and Activity, and Major Adverse Cardiovascular Events and Malignancies in Patients With Rheumatoid Arthritis Receiving Tofacitinib. J Rheumatol. 2023 Jul 15:jrheum.2023-0112. doi: 10.3899/jrheum.2023-0112. Online ahead of print. PMID 37453736
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Dougados M, Taylor PC, Bingham CO 3rd, Fallon L, Brault Y, Roychoudhury S, Wang L, Kessouri M. The effect of tofacitinib on residual pain in patients with rheumatoid arthritis and psoriatic arthritis. RMD Open. 2022 Sep;8(2):e002478. doi: 10.1136/rmdopen-2022-002478. PMID 36814062
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Dikranian AH, Gonzalez-Gay MA, Wellborne F, Alvaro-Gracia JM, Takiya L, Stockert L, Paulissen J, Shi H, Tatulych S, Curtis JR. Efficacy of tofacitinib in patients with rheumatoid arthritis stratified by baseline body mass index: an analysis of pooled data from phase 3 studies. RMD Open. 2022 May;8(1):e002103. doi: 10.1136/rmdopen-2021-002103. PMID 35577477
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Bykerk VP, Lee EB, van Vollenhoven R, Gruben DC, Fallon L, Woolcott JC, Keystone E. Identification of Distinct Disease Activity Trajectories in Methotrexate-Naive Patients With Rheumatoid Arthritis Receiving Tofacitinib Over Twenty-Four Months. Arthritis Care Res (Hoboken). 2022 Jan;74(1):131-141. doi: 10.1002/acr.24709. PMID 34057820
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Strand V, Kaine J, Alten R, Wallenstein G, Diehl A, Shi H, Germino R, Murray CW. Associations between Patient Global Assessment scores and pain, physical function, and fatigue in rheumatoid arthritis: a post hoc analysis of data from phase 3 trials of tofacitinib. Arthritis Res Ther. 2020 Oct 15;22(1):243. doi: 10.1186/s13075-020-02324-7. PMID 33059710
- [Derived] van der Heijde D, Landewe RBM, Wollenhaupt J, Strengholt S, Terry K, Kwok K, Wang L, Cohen S. Assessment of radiographic progression in patients with rheumatoid arthritis treated with tofacitinib in long-term studies. Rheumatology (Oxford). 2021 Apr 6;60(4):1708-1716. doi: 10.1093/rheumatology/keaa476. PMID 33057725
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Kivitz AJ, Cohen S, Keystone E, van Vollenhoven RF, Haraoui B, Kaine J, Fan H, Connell CA, Bananis E, Takiya L, Fleischmann R. A pooled analysis of the safety of tofacitinib as monotherapy or in combination with background conventional synthetic disease-modifying antirheumatic drugs in a Phase 3 rheumatoid arthritis population. Semin Arthritis Rheum. 2018 Dec;48(3):406-415. doi: 10.1016/j.semarthrit.2018.07.006. Epub 2018 Jul 19. PMID 30177460
- [Derived] Strand V, Kavanaugh A, Kivitz AJ, van der Heijde D, Kwok K, Akylbekova E, Soonasra A, Snyder M, Connell C, Bananis E, Smolen JS. Long-Term Radiographic and Patient-Reported Outcomes in Patients with Rheumatoid Arthritis Treated with Tofacitinib: ORAL Start and ORAL Scan Post-hoc Analyses. Rheumatol Ther. 2018 Dec;5(2):341-353. doi: 10.1007/s40744-018-0113-7. Epub 2018 May 14. PMID 29761420
- [Derived] van Vollenhoven RF, Lee EB, Fallon L, Zwillich SH, Wilkinson B, Chapman D, DeMasi R, Keystone E. Tofacitinib in Rheumatoid Arthritis: Lack of Early Change in Disease Activity and the Probability of Achieving Low Disease Activity at Month 6. Arthritis Care Res (Hoboken). 2019 Jan;71(1):71-79. doi: 10.1002/acr.23585. PMID 29696833
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Fleischmann RM, Huizinga TW, Kavanaugh AF, Wilkinson B, Kwok K, DeMasi R, van Vollenhoven RF. Efficacy of tofacitinib monotherapy in methotrexate-naive patients with early or established rheumatoid arthritis. RMD Open. 2016 Jul 26;2(2):e000262. doi: 10.1136/rmdopen-2016-000262. eCollection 2016. PMID 27493790
- [Derived] Fleischmann R, Strand V, Wilkinson B, Kwok K, Bananis E. Relationship between clinical and patient-reported outcomes in a phase 3 trial of tofacitinib or MTX in MTX-naive patients with rheumatoid arthritis. RMD Open. 2016 Apr 26;2(1):e000232. doi: 10.1136/rmdopen-2015-000232. eCollection 2016. PMID 27175296
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- [Derived] Lee EB, Fleischmann R, Hall S, Wilkinson B, Bradley JD, Gruben D, Koncz T, Krishnaswami S, Wallenstein GV, Zang C, Zwillich SH, van Vollenhoven RF; ORAL Start Investigators. Tofacitinib versus methotrexate in rheumatoid arthritis. N Engl J Med. 2014 Jun 19;370(25):2377-86. doi: 10.1056/NEJMoa1310476. PMID 24941177
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921069&StudyName=Comparing%20The%20Effectiveness%20And%20Safety%20Of%202%20Doses%20Of%20An%20Experimental%20Drug%2C%20CP-690%2C550%2C%20To%20Methotrexate%20%28MTX%29%20In%20Patients%20With%20

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 5 mg Twice Daily (BID): Participants received CP-690,550 5 milligram (mg) tablets, orally, BID, matching placebo CP-690,550 tablets, orally, BID, and matching placebo methotrexate (MTX) capsules, orally, once per week, for up to 24 months.
- CP-690,550 10 mg BID: Participants received CP-690,550 two 5 mg tablets, orally, BID, and matching placebo MTX capsules, orally, once per week, for up to 24 months.
- MTX 10, 15, or 20 mg, Weekly: Participants received MTX capsules at doses of 10 to 20 mg per week and matching placebo CP-690,550 tablets, orally, BID, for up to 24 months. MTX dose was titrated to a maximum of 20 mg/week as follows: 10 mg/once weekly for 4 weeks, if tolerated the dose was titrated to 15 mg/once weekly for 4 weeks, if tolerated the dose was titrated to 20 mg/once weekly. One dose reduction was allowed for lack of tolerance.
Period: Overall Study
Arm/Group | CP-690,550 5 mg Twice Daily (BID) | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Started | 373 | 397 | 186
Completed | 266 | 286 | 106
Not Completed | 107 | 111 | 80
Not completed — Adverse Event | 38 | 39 | 24
Not completed — Lack of Efficacy | 20 | 11 | 26
Not completed — Lost to Follow-up | 11 | 9 | 5
Not completed — Other | 13 | 25 | 12
Not completed — Withdrawal by Subject | 23 | 27 | 13
Not completed — Death | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants randomized to the study who received at least 1 dose of study drug (CP-690,550) or MTX.
Groups:
- CP-690,550 5 mg Twice Daily (BID): Participants received CP-690,550 5 mg tablets, orally, BID, matching placebo CP-690,550 tablets, orally, BID, and matching placebo MTX capsules, orally, once per week, for up to 24 months.
- Total: Total of all reporting groups
Arm/Group | CP-690,550 5 mg Twice Daily (BID) | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly | Total
Number analyzed (Participants) | 373 | 397 | 186 | 956
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (12.2) | 49.3 (12.8) | 48.8 (13.3) | 49.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 286 | 327 | 145 | 758
  Male | 87 | 70 | 41 | 198

OUTCOME MEASURES:

1. Primary Outcome: Modified Total Sharp Score (mTSS) at Month 6
Description: mTSS: sum of erosion and joint space narrowing (JSN) scores for 44 joints (16 per hand and 6 per foot). mTSS scores range from 0 (normal) to 448 (worst possible total score).
Time Frame: Month 6
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug (CP-690,550) or MTX (in MTX-naive participants) with a baseline (BL) and at least 1 nonmissing on-study assessment. Missing values due to withdrawal were imputed using linear extrapolation (LEP) of BL/post-BL value before withdrawal.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- CP-690,550 5 mg BID: Participants received CP-690,550 5 mg) tablets, orally, BID, matching placebo CP-690,550 tablets, orally, BID, and matching placebo MTX capsules, orally, once per week, for up to 24 months.
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 346 | 369 | 166
score on a scale | 20.50 (40.58) | 18.85 (39.21) | 17.54 (29.96)

2. Primary Outcome: Change From Baseline at Month 6 in mTSS
Description: mTSS: sum of erosion and JSN scores for 44 joints (16 per hand and 6 per foot). mTSS scores range from 0 (normal) to 448 (worst possible total score). An increase in mTSS from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represents improvement.
Time Frame: Month 6
Population: FAS, imputation using LEP
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- CP-690,550 5 mg BID: Participants received CP-690,550 5 mg tablets, orally, BID, matching placebo CP-690,550 tablets, orally, BID, and matching placebo MTX capsules, orally, once per week, for up to 24 months.
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 346 | 370 | 165
score on a scale | 0.20 (0.09) | 0.15 (0.08) | 0.65 (0.12)
Statistical Analysis 1: Comparison: CP-690,550 5 mg BID vs MTX 10, 15, or 20 mg, Weekly; Test type: Superiority or Other; p = 0.0014, ANCOVA — A stepdown procedure was used to control for multiple comparisons. In order for the comparison of CP-690,550 5 mg to be statistically significant versus MTX, the comparison of CP-690,550 10 mg versus MTX had to be statistically significant; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.73 to -0.18], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: CP-690,550 10 mg BID vs MTX 10, 15, or 20 mg, Weekly; Test type: Superiority or Other; p = 0.0004, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.77 to -0.23], Standard Error of Mean 0.14

3. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 70 (ACR70) Response at Month 6
Description: ACR70 response: greater than or equal to (≥) 70 percent (%) improvement in tender joints count (TJC) or swollen joints count (SJC) and ≥70% improvement in at least 3 of 5 remaining ACR core measures: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability (disability index of the Health Assessment Questionnaire [HAQ]), and 5) C-reactive protein (CRP).
Time Frame: Month 6
Population: FAS. Missing values due to participant withdrawal were imputed using nonresponder imputation (NRI) method.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 366 | 391 | 182
percentage of participants | 25.41 | 37.34 | 12.09
Statistical Analysis 1: Comparison: CP-690,550 5 mg BID vs MTX 10, 15, or 20 mg, Weekly; Test type: Superiority or Other; p < 0.0001, Normal approximation — A stepdown procedure was used to control for multiple comparisons. For comparison of 5 mg to be statistically significant, comparison of 10 mg to MTX in ACR70 and comparison of 5 mg to MTX in change from BL in mTSS had to be statistically significant; Risk Difference (RD) = 13.32, 95% CI 2-sided [6.81 to 19.82]
Statistical Analysis 2: Comparison: CP-690,550 10 mg BID vs MTX 10, 15, or 20 mg, Weekly; Test type: Superiority or Other; p < 0.0001, Normal approximation — A stepdown procedure was used to control for multiple comparisons. For comparison of 10 mg to MTX in ACR70 to be statistically significant, comparison of 10 mg to MTX in change from BL in mTSS had to be statistically significant; Risk Difference (RD) = 25.25, 95% CI 2-sided [18.51 to 31.99]

4. Primary Outcome: Absolute Blood Pressure (BP) Values (mmHg)
Description: BP: pressure exerted by the blood upon the walls of the blood vessels and especially arteries, usually measured on the radial artery using a sphygmomanometer. Systolic BP: the highest arterial blood pressure of a cardiac cycle occurring immediately after systole of the left ventricle of the heart. Diastolic BP: the lowest arterial blood pressure of a cardiac cycle occurring during diastole of the heart.
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, and 24
Population: FAS; 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
mmHg
  Baseline: systolic BP | 123.37 (15.41) | 124.30 (14.79) | 123.47 (13.73)
  Baseline: diastolic BP | 77.64 (8.97) | 77.59 (8.90) | 78.02 (8.89)
  Month 1: systolic BP: number analyzed (Participants) | 365 | 393 | 184
  Month 1: systolic BP | 123.76 (15.28) | 124.57 (14.17) | 123.41 (14.59)
  Month 1: diastolic BP: number analyzed (Participants) | 365 | 393 | 184
  Month 1: diastolic BP | 77.79 (9.11) | 78.30 (8.62) | 76.09 (9.00)
  Month 2: systolic BP: number analyzed (Participants) | 361 | 388 | 178
  Month 2: systolic BP | 123.65 (14.87) | 124.28 (13.33) | 122.59 (13.89)
  Month 2: diastolic BP: number analyzed (Participants) | 361 | 388 | 178
  Month 2: diastolic BP | 77.77 (9.08) | 78.68 (8.81) | 76.22 (9.82)
  Month 3: systolic BP: number analyzed (Participants) | 355 | 383 | 172
  Month 3: systolic BP | 124.08 (14.94) | 124.24 (14.40) | 122.61 (13.18)
  Month 3: diastolic BP: number analyzed (Participants) | 355 | 383 | 172
  Month 3: diastolic BP | 77.80 (9.19) | 78.33 (9.54) | 76.52 (7.80)
  Month 6: systolic BP: number analyzed (Participants) | 340 | 365 | 158
  Month 6: systolic BP | 123.71 (14.56) | 125.02 (14.37) | 122.28 (12.81)
  Month 6: diastolic BP: number analyzed (Participants) | 340 | 365 | 158
  Month 6: diastolic BP | 77.74 (8.70) | 78.56 (8.69) | 76.50 (8.32)
  Month 9: systolic BP: number analyzed (Participants) | 328 | 349 | 144
  Month 9: systolic BP | 123.90 (13.98) | 123.89 (13.71) | 121.94 (13.01)
  Month 9: diastolic BP: number analyzed (Participants) | 328 | 349 | 144
  Month 9: diastolic BP | 78.01 (9.11) | 77.70 (8.38) | 76.34 (8.53)
  Month 12: systolic BP: number analyzed (Participants) | 315 | 331 | 135
  Month 12: systolic BP | 125.61 (15.05) | 124.34 (13.68) | 122.22 (12.70)
  Month 12: diastolic BP: number analyzed (Participants) | 315 | 331 | 135
  Month 12: diastolic BP | 78.08 (9.14) | 78.08 (8.16) | 76.59 (8.12)
  Month 15: systolic BP: number analyzed (Participants) | 293 | 313 | 128
  Month 15: systolic BP | 124.63 (14.24) | 124.28 (13.48) | 123.71 (13.46)
  Month 15: diastolic BP: number analyzed (Participants) | 293 | 313 | 128
  Month 15: diastolic BP | 77.98 (8.77) | 78.04 (8.42) | 76.46 (8.95)
  Month 18: systolic BP: number analyzed (Participants) | 284 | 294 | 115
  Month 18: systolic BP | 124.48 (13.65) | 124.39 (12.75) | 121.57 (13.08)
  Month 18: diastolic BP: number analyzed (Participants) | 284 | 294 | 115
  Month 18: diastolic BP | 77.66 (8.90) | 78.34 (8.02) | 76.76 (8.89)
  Month 21: systolic BP: number analyzed (Participants) | 272 | 290 | 111
  Month 21: systolic BP | 123.83 (13.53) | 124.52 (12.91) | 123.29 (11.98)
  Month 21: diastolic BP: number analyzed (Participants) | 272 | 290 | 111
  Month 21: diastolic BP | 77.28 (8.24) | 78.44 (7.56) | 76.45 (8.34)
  Month 24: systolic BP: number analyzed (Participants) | 263 | 280 | 105
  Month 24: systolic BP | 124.48 (13.15) | 124.34 (12.24) | 122.47 (12.56)
  Month 24: diastolic BP: number analyzed (Participants) | 264 | 280 | 105
  Month 24: diastolic BP | 78.25 (8.15) | 78.07 (7.73) | 76.57 (8.46)

5. Primary Outcome: Change From Baseline in BP Values (mmHg)
Description: as for outcome 4
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, and 24
Population: FAS; 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 365 | 393 | 184
mmHg
  Month 1: systolic BP | 0.44 (11.70) | 0.32 (11.03) | -0.02 (11.75)
  Month 1: diastolic BP | 0.11 (7.35) | 0.78 (7.88) | -1.91 (7.96)
  Month 2: systolic BP: number analyzed (Participants) | 361 | 388 | 178
  Month 2: systolic BP | 0.41 (12.74) | 0.07 (12.84) | -0.43 (10.93)
  Month 2: diastolic BP: number analyzed (Participants) | 361 | 388 | 178
  Month 2: diastolic BP | 0.13 (8.56) | 1.18 (8.86) | -1.63 (8.07)
  Month 3: systolic BP: number analyzed (Participants) | 355 | 383 | 172
  Month 3: systolic BP | 0.91 (13.84) | -0.25 (12.71) | -0.48 (11.64)
  Month 3: diastolic BP: number analyzed (Participants) | 355 | 383 | 172
  Month 3: diastolic BP | 0.16 (8.70) | 0.70 (8.37) | -1.31 (8.08)
  Month 6: systolic BP: number analyzed (Participants) | 340 | 365 | 158
  Month 6: systolic BP | 0.34 (12.60) | 0.36 (12.15) | -0.97 (10.45)
  Month 6: diastolic BP: number analyzed (Participants) | 340 | 365 | 158
  Month 6: diastolic BP | -0.04 (8.29) | 0.87 (8.34) | -1.41 (7.95)
  Month 9: systolic BP: number analyzed (Participants) | 328 | 349 | 144
  Month 9: systolic BP | 0.35 (12.33) | -0.43 (12.52) | -1.69 (10.79)
  Month 9: diastolic BP: number analyzed (Participants) | 328 | 349 | 144
  Month 9: diastolic BP | 0.14 (9.12) | 0.04 (8.47) | -1.79 (8.42)
  Month 12: systolic BP: number analyzed (Participants) | 315 | 331 | 135
  Month 12: systolic BP | 2.32 (12.94) | -0.02 (13.17) | -1.36 (11.19)
  Month 12: diastolic BP: number analyzed (Participants) | 315 | 331 | 135
  Month 12: diastolic BP | 0.29 (9.00) | 0.37 (8.03) | -1.41 (7.25)
  Month 15: systolic BP: number analyzed (Participants) | 293 | 313 | 128
  Month 15: systolic BP | 0.93 (12.90) | -0.00 (13.57) | -0.16 (12.14)
  Month 15: diastolic BP: number analyzed (Participants) | 293 | 313 | 128
  Month 15: diastolic BP | -0.11 (8.98) | 0.41 (8.38) | -1.63 (8.78)
  Month 18: systolic BP: number analyzed (Participants) | 284 | 294 | 115
  Month 18: systolic BP | 1.09 (12.61) | 0.23 (12.45) | -2.38 (13.23)
  Month 18: diastolic BP: number analyzed (Participants) | 284 | 294 | 115
  Month 18: diastolic BP | -0.30 (8.42) | 0.59 (9.09) | -1.49 (8.82)
  Month 21: systolic BP: number analyzed (Participants) | 272 | 290 | 111
  Month 21: systolic BP | 0.49 (13.08) | 0.31 (13.68) | -0.68 (11.18)
  Month 21: diastolic BP: number analyzed (Participants) | 272 | 290 | 111
  Month 21: diastolic BP | -0.71 (8.94) | 0.65 (9.14) | -1.63 (8.06)
  Month 24: systolic BP: number analyzed (Participants) | 263 | 280 | 105
  Month 24: systolic BP | 1.30 (12.73) | 0.06 (13.55) | -1.11 (12.42)
  Month 24: diastolic BP: number analyzed (Participants) | 264 | 280 | 105
  Month 24: diastolic BP | 0.38 (8.94) | 0.28 (9.62) | -1.50 (7.75)

6. Secondary Outcome: mTSS Score at Baseline, Months 12 and 24
Description: mTSS: sum of erosion and JSN scores for 44 joints (16 per hand and 6 per foot). mTSS scores range from 0 (normal) to 448 (worst possible total score).
Time Frame: Baseline, Months 12 and 24
Population: FAS, imputation using LEP; 'n' (number of participants analyzed) signifies participants who were evaluable for this measure at a given timepoint for each group, respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 348 | 373 | 171
score on a scale
  Baseline | 19.05 (38.27) | 17.89 (38.49) | 16.11 (29.44)
  Month 12: number analyzed (Participants) | 347 | 373 | 171
  Month 12 | 19.23 (38.37) | 18.08 (38.41) | 17.32 (30.27)
  Month 24 | 19.70 (38.69) | 18.23 (38.43) | 18.26 (30.99)

7. Secondary Outcome: Change From Baseline in mTSS Score at Months 12 and 24
Description: as for outcome 2
Time Frame: Months 12 and 24
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 346 | 371 | 169
score on a scale
  Month 12: number analyzed (Participants) | 345 | 371 | 169
  Month 12 | 0.37 (0.14) | 0.17 (0.14) | 1.20 (0.20)
  Month 24 | 0.57 (0.25) | 0.28 (0.24) | 2.11 (0.35)

8. Secondary Outcome: Percentage of Participants With no Progression in mTSS at Months 6, 12, and 24
Description: mTSS: sum of erosion and JSN scores for 44 joints (16 per hand and 6 per foot). mTSS scores range from 0 (normal) to 448 (worst possible total score). A increase of less than or equal to (≤)0.5 in mTSS is considered to be no progression in the mTSS.
Time Frame: Months 6, 12, and 24
Population: FAS (LEP); 'n' (number of participants analyzed) signifies participants who were evaluable for this measure at a given timepoint for each group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 348 | 373 | 171
percentage of participants
  Month 6: number analyzed (Participants) | 348 | 372 | 167
  Month 6 | 87.07 | 89.25 | 73.65
  Month 12: number analyzed (Participants) | 347 | 373 | 171
  Month 12 | 82.42 | 87.67 | 69.01
  Month 24 | 79.89 | 83.65 | 64.91

9. Secondary Outcome: Percentage of Participants With no Worsening in Erosion Score (Increase ≤0.5) at Months 6, 12, and 24
Description: Joint erosion score: erosion severity in 44 joints (16 per hand, 6 per foot). Each joint scored according to surface area involved, from 0 (no erosion) to 5 (extensive bone loss from more than one half of articulating bone). Because each side of foot joint was graded, maximum erosion score for foot joint was 10. Thus, maximum erosion score was 280. An increase of ≤0.5 in Erosion Score is considered to be 'no worsening' in the Erosion Score.
Time Frame: Months 6, 12, and 24
Population: FAS (LEP)
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 348 | 373 | 171
percentage of participants
  Month 6: number analyzed (Participants) | 348 | 372 | 167
  Month 6 | 91.67 | 93.01 | 81.44
  Month 12: number analyzed (Participants) | 347 | 373 | 171
  Month 12 | 88.47 | 90.88 | 74.85
  Month 24 | 85.34 | 88.20 | 70.18

10. Secondary Outcome: Erosion Scores
Description: Joint erosion score: erosion severity in 44 joints (16 per hand, 6 per foot). Each joint scored according to surface area involved, from 0 (no erosion) to 5 (extensive bone loss from more than one half of articulating bone). Because each side of foot joint was graded, maximum erosion score for foot joint was 10. Thus, maximum erosion score was 280.
Time Frame: Baseline, Months 6, 12, and 24
Population: FAS, imputation using LEP
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 348 | 373 | 171
units on a scale
  Baseline | 9.05 (19.00) | 9.06 (19.50) | 8.38 (15.24)
  Month 6: number analyzed (Participants) | 348 | 372 | 167
  Month 6 | 9.18 (19.10) | 9.15 (19.50) | 8.78 (15.54)
  Month 12: number analyzed (Participants) | 347 | 373 | 171
  Month 12 | 9.05 (18.97) | 9.18 (19.42) | 8.97 (15.46)
  Month 24 | 9.21 (18.95) | 9.22 (19.36) | 9.37 (15.67)

11. Secondary Outcome: JSN Scores
Description: JSN score: severity of JSN in 42 joints (15 per hand and 6 per foot), including subluxation, scored from 0 (no/normal JSN) to 4 (complete loss of joint space, bony ankylosis, or luxation). Maximum JSN score was 168.
Time Frame: Baseline, Months 6, 12, and 24
Population: FAS, imputation using LEP
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 348 | 373 | 171
score on a scale
  Baseline | 10.01 (20.58) | 8.82 (19.80) | 7.72 (15.28)
  Month 6: number analyzed (Participants) | 348 | 372 | 167
  Month 6 | 10.09 (20.62) | 8.86 (19.79) | 8.17 (15.70)
  Month 12: number analyzed (Participants) | 347 | 373 | 171
  Month 12 | 10.18 (20.74) | 8.90 (19.77) | 8.35 (16.01)
  Month 24 | 10.50 (21.12) | 9.01 (19.87) | 8.89 (16.76)

12. Secondary Outcome: Change From Baseline in Erosion Scores
Description: Joint erosion score: erosion severity in 44 joints (16 per hand, 6 per foot). Each joint scored according to surface area involved, from 0 (no erosion) to 5 (extensive bone loss from more than one half of articulating bone). Because each side of foot joint was graded, maximum erosion score for foot joint was 10. Thus, maximum erosion score was 280. Change = score at observation minus score at Baseline. An increase in score from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Months 6, 12, and 24
Population: FAS, imputation using LEP
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 348 | 373 | 171
units on a scale
  Month 6: number analyzed (Participants) | 348 | 372 | 167
  Month 6 | 0.14 (0.04) | 0.10 (0.04) | 0.35 (0.06)
  Month 12: number analyzed (Participants) | 347 | 373 | 171
  Month 12 | 0.13 (0.07) | 0.12 (0.06) | 0.58 (0.09)
  Month 24 | 0.16 (0.11) | 0.16 (0.10) | 0.98 (0.15)

13. Secondary Outcome: Change From Baseline in JSN Scores
Description: JSN score: severity of JSN in 42 joints (15 per hand and 6 per foot), including subluxation, scored from 0 (no/normal JSN) to 4 (complete loss of joint space, bony ankylosis, or luxation). Maximum JSN score was 168. Change = scores at observation minus score at Baseline. An increase in score from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Months 6, 12, and 24
Population: FAS, imputation using LEP
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 348 | 373 | 171
units on a scale
  Month 6: number analyzed (Participants) | 348 | 372 | 167
  Month 6 | 0.06 (0.06) | 0.05 (0.06) | 0.29 (0.09)
  Month 12: number analyzed (Participants) | 347 | 373 | 171
  Month 12 | 0.23 (0.10) | 0.05 (0.10) | 0.60 (0.14)
  Month 24 | 0.39 (0.18) | 0.12 (0.17) | 1.10 (0.25)

14. Secondary Outcome: Percentage of Participants Achieving an ACR70 Response
Description: ACR70 response: ≥70% improvement in TJC or SJC and ≥70% improvement in at least 3 of 5 remaining ACR core measures: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability (disability index of HAQ), and 5) CRP.
Time Frame: Months 1, 2, 3, 9, 12, 15, 18, 21, and 24
Population: FAS (NRI)
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 366 | 391 | 182
percentage of participants
  Month 1: number analyzed (Participants) | 364 | 390 | 182
  Month 1 | 5.22 | 9.23 | 0.55
  Month 2: number analyzed (Participants) | 365 | 391 | 182
  Month 2 | 16.16 | 23.02 | 3.30
  Month 3 | 19.95 | 26.60 | 5.49
  Month 9 | 29.23 | 37.85 | 13.19
  Month 12 | 28.69 | 37.85 | 15.38
  Month 15 | 30.05 | 37.85 | 17.03
  Month 18 | 32.24 | 36.57 | 15.93
  Month 21 | 32.24 | 36.83 | 17.58
  Month 24 | 34.15 | 37.60 | 15.38

15. Secondary Outcome: Percentage of Participants Achieving an ACR20 Response
Description: ACR20 response: ≥20% improvement in TJC or SJC and ≥20% improvement in at least 3 of 5 remaining ACR core measures: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability (disability index of HAQ), and 5) CRP.
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS (NRI)
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 369 | 394 | 184
percentage of participants
  Month 1: number analyzed (Participants) | 367 | 393 | 184
  Month 1 | 49.32 | 58.27 | 21.20
  Month 2: number analyzed (Participants) | 368 | 394 | 184
  Month 2 | 63.59 | 71.57 | 42.39
  Month 3 | 69.92 | 77.92 | 51.63
  Month 6 | 71.27 | 76.14 | 50.54
  Month 9 | 72.09 | 73.60 | 55.43
  Month 12 | 67.75 | 71.57 | 51.09
  Month 15 | 68.83 | 66.24 | 47.28
  Month 18 | 64.23 | 65.99 | 46.74
  Month 21 | 65.04 | 62.18 | 45.11
  Month 24 | 64.23 | 64.21 | 42.39

16. Secondary Outcome: Percentage of Participants Achieving an ACR50 Response
Description: ACR50 response: ≥50% improvement in TJC or SJC and ≥50% improvement in at least 3 of 5 remaining ACR core measures: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability (disability index of HAQ), and 5) CRP.
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS (NRI)
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 369 | 394 | 184
percentage of participants
  Month 1: number analyzed (Participants) | 367 | 393 | 184
  Month 1 | 17.98 | 27.99 | 3.80
  Month 2: number analyzed (Participants) | 368 | 394 | 184
  Month 2 | 32.61 | 40.10 | 11.41
  Month 3 | 40.11 | 50.00 | 20.11
  Month 6 | 46.61 | 56.35 | 26.63
  Month 9 | 49.86 | 56.85 | 35.33
  Month 12 | 49.86 | 55.58 | 33.70
  Month 15 | 50.68 | 54.31 | 33.15
  Month 18 | 47.97 | 51.78 | 30.43
  Month 21 | 49.05 | 50.51 | 30.43
  Month 24 | 49.32 | 49.24 | 28.26

17. Secondary Outcome: Tender Joints Count (TJC)
Description: Sixty-eight (68) joints were assessed by a blinded joint assessor to determine the number of joints considered tender or painful. The response to pressure/motion on each joint was assessed using the following scale: Present/Absent/Not Done/Not Applicable (to be used for artificial or missing joints). Artificial joints were not assessed. 68 joints to be assessed were: upper body (temporomandibular, sternoclavicular, acromioclavicular); upper extremity: shoulder, elbow, wrist (radiocarpal, carpal and carpometacarpal considered as one unit), metacarpophalangeals (MCP I, II, III, IV, V), thumb interphalangeal (IP), proximal interphalangeals (PIP II, III, IV, V), distal interphalangeals (DIP II, III, IV, V); lower extremity: hip, knee, ankle, tarsus (includes subtalar, transverse tarsal and tarsometatarsal considered as one unit), metatarsophalangeals (MTP I, II, III, IV, V), great toe IP, proximal and distal interphalangeals combined (PIP II, III, IV, V).
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS; 'n' (number of participants analyzed) signifies participants who were evaluable for this measure at a given timepoint for each group, respectively.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
tender joints
  Baseline | 25.65 (13.81) | 25.12 (13.51) | 25.41 (15.03)
  Month 1: number analyzed (Participants) | 367 | 393 | 184
  Month 1 | 15.75 (12.98) | 13.66 (12.61) | 20.07 (14.83)
  Month 2: number analyzed (Participants) | 361 | 388 | 177
  Month 2 | 12.12 (12.31) | 10.67 (12.31) | 16.39 (14.16)
  Month 3: number analyzed (Participants) | 356 | 383 | 172
  Month 3 | 10.03 (11.52) | 8.61 (10.67) | 14.05 (14.13)
  Month 6: number analyzed (Participants) | 340 | 367 | 158
  Month 6 | 8.71 (11.04) | 6.59 (10.28) | 11.99 (13.34)
  Month 9: number analyzed (Participants) | 328 | 350 | 143
  Month 9 | 7.31 (10.45) | 6.14 (10.11) | 8.82 (11.27)
  Month 12: number analyzed (Participants) | 315 | 332 | 136
  Month 12 | 6.60 (9.78) | 5.46 (10.16) | 9.13 (12.67)
  Month 15: number analyzed (Participants) | 294 | 313 | 129
  Month 15 | 5.55 (9.15) | 5.17 (9.79) | 8.23 (10.50)
  Month 18: number analyzed (Participants) | 284 | 295 | 116
  Month 18 | 5.12 (7.15) | 4.46 (7.98) | 6.97 (8.74)
  Month 21: number analyzed (Participants) | 273 | 290 | 111
  Month 21 | 4.60 (6.87) | 4.19 (6.40) | 7.07 (9.68)
  Month 24: number analyzed (Participants) | 264 | 281 | 106
  Month 24 | 4.50 (6.75) | 4.66 (8.52) | 6.01 (6.81)

18. Secondary Outcome: Change From Baseline in TJC
Description: Sixty-eight (68) joints were assessed by a blinded joint assessor to determine the number of joints considered tender or painful. The response to pressure/motion on each joint was assessed using the following scale: Present/Absent/Not Done/Not Applicable (to be used for artificial or missing joints). Artificial joints were not assessed. 68 joints to be assessed were: upper body (temporomandibular, sternoclavicular, acromioclavicular); upper extremity: shoulder, elbow, wrist (radiocarpal, carpal and carpometacarpal considered as one unit), MCP (I, II, III, IV, V), thumb IP, PIP (II, III, IV, V), DIP (II, III, IV, V); lower extremity: hip, knee, ankle, tarsus (includes subtalar, transverse tarsal and tarsometatarsal considered as one unit), MTP (I, II, III, IV, V), great toe IP, proximal and distal interphalangeals combined (PIP II, III, IV, V).
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: tender joints
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 367 | 393 | 184
tender joints
  Month 1 | -9.43 (0.54) | -11.40 (0.52) | -5.11 (0.75)
  Month 2: number analyzed (Participants) | 361 | 388 | 177
  Month 2 | -12.95 (0.54) | -14.33 (0.52) | -8.63 (0.76)
  Month 3: number analyzed (Participants) | 356 | 383 | 172
  Month 3 | -14.95 (0.55) | -16.34 (0.52) | -10.69 (0.77)
  Month 6: number analyzed (Participants) | 340 | 367 | 158
  Month 6 | -16.00 (0.55) | -18.09 (0.53) | -12.38 (0.79)
  Month 9: number analyzed (Participants) | 328 | 350 | 143
  Month 9 | -17.16 (0.56) | -18.29 (0.54) | -15.39 (0.81)
  Month 12: number analyzed (Participants) | 315 | 332 | 136
  Month 12 | -17.85 (0.56) | -18.44 (0.54) | -14.74 (0.82)
  Month 15: number analyzed (Participants) | 294 | 313 | 129
  Month 15 | -18.86 (0.58) | -18.57 (0.55) | -15.70 (0.83)
  Month 18: number analyzed (Participants) | 284 | 295 | 116
  Month 18 | -19.08 (0.58) | -19.41 (0.56) | -16.41 (0.86)
  Month 21: number analyzed (Participants) | 273 | 290 | 111
  Month 21 | -19.54 (0.59) | -19.70 (0.57) | -16.24 (0.87)
  Month 24: number analyzed (Participants) | 264 | 281 | 106
  Month 24 | -19.64 (0.59) | -19.23 (0.57) | -17.01 (0.89)

19. Secondary Outcome: Swollen Joints Count (SJC)
Description: Sixty-six (66) joints were assessed by a blinded joint assessor for swelling using the following scale: Present/Absent/Not Done/Not Applicable (to be used for artificial or missing joints). Artificial joints were not assessed. 66 joints assessed were: upper body (temporomandibular, sternoclavicular, acromioclavicular); upper extremity: shoulder, elbow, wrist (radiocarpal, carpal and carpometacarpal considered as one unit), MCP (I, II, III, IV, V), thumb IP, PIP (II, III, IV, V), DIP (II, III, IV, V); lower extremity: knee, ankle, tarsus (includes subtalar, transverse tarsal and tarsometatarsal considered as one unit), MTP (I, II, III, IV, V), great toe IP, proximal and distal interphalangeals combined (PIP II, III, IV, V).
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
swollen joints
  Baseline | 16.27 (9.24) | 15.58 (8.37) | 16.76 (10.27)
  Month 1: number analyzed (Participants) | 367 | 393 | 184
  Month 1 | 9.90 (9.60) | 8.02 (7.03) | 12.56 (9.40)
  Month 2: number analyzed (Participants) | 361 | 388 | 177
  Month 2 | 6.84 (7.74) | 5.69 (6.29) | 9.97 (9.05)
  Month 3: number analyzed (Participants) | 356 | 383 | 172
  Month 3 | 5.81 (8.76) | 4.32 (5.53) | 7.88 (7.98)
  Month 6: number analyzed (Participants) | 340 | 367 | 158
  Month 6 | 4.70 (7.40) | 3.69 (6.05) | 6.30 (7.12)
  Month 9: number analyzed (Participants) | 328 | 350 | 143
  Month 9 | 3.83 (5.67) | 3.22 (5.93) | 4.83 (6.74)
  Month 12: number analyzed (Participants) | 315 | 332 | 136
  Month 12 | 3.30 (6.12) | 2.88 (6.77) | 5.17 (9.44)
  Month 15: number analyzed (Participants) | 294 | 313 | 129
  Month 15 | 2.63 (6.35) | 3.00 (7.95) | 4.92 (8.21)
  Month 18: number analyzed (Participants) | 284 | 295 | 116
  Month 18 | 2.44 (4.07) | 2.25 (5.28) | 3.91 (4.85)
  Month 21: number analyzed (Participants) | 273 | 290 | 111
  Month 21 | 2.28 (4.12) | 2.02 (4.00) | 3.47 (4.14)
  Month 24: number analyzed (Participants) | 264 | 281 | 106
  Month 24 | 2.00 (3.70) | 2.29 (6.44) | 3.38 (4.26)

20. Secondary Outcome: Change From Baseline in SJC
Description: as for outcome 19
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: swollen joints
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 367 | 393 | 184
swollen joints
  Month 1 | -5.99 (0.36) | -7.75 (0.35) | -3.55 (0.51)
  Month 2: number analyzed (Participants) | 361 | 388 | 177
  Month 2 | -8.95 (0.37) | -10.03 (0.35) | -5.98 (0.51)
  Month 3: number analyzed (Participants) | 356 | 383 | 172
  Month 3 | -9.97 (0.37) | -11.42 (0.35) | -7.97 (0.52)
  Month 6: number analyzed (Participants) | 340 | 367 | 158
  Month 6 | -10.89 (0.37) | -11.97 (0.36) | -9.35 (0.53)
  Month 9: number analyzed (Participants) | 328 | 350 | 143
  Month 9 | -11.47 (0.38) | -12.39 (0.36) | -11.00 (0.55)
  Month 12: number analyzed (Participants) | 315 | 332 | 136
  Month 12 | -11.97 (0.38) | -12.54 (0.37) | -10.48 (0.56)
  Month 15: number analyzed (Participants) | 294 | 313 | 129
  Month 15 | -12.55 (0.39) | -12.30 (0.38) | -10.69 (0.57)
  Month 18: number analyzed (Participants) | 284 | 295 | 116
  Month 18 | -12.63 (0.39) | -13.10 (0.38) | -11.31 (0.59)
  Month 21: number analyzed (Participants) | 273 | 290 | 111
  Month 21 | -12.74 (0.40) | -13.28 (0.38) | -11.89 (0.60)
  Month 24: number analyzed (Participants) | 264 | 281 | 106
  Month 24 | -12.99 (0.40) | -13.06 (0.39) | -11.96 (0.61)

21. Secondary Outcome: Patient Assessment of Arthritis Pain
Description: Participants rated the severity of arthritis pain on a 0 to 100 millimeter (mm) visual analogue scale (VAS), where 0 mm=no pain and 100 mm=most severe pain.
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
mm
  Baseline | 59.06 (23.87) | 61.37 (23.14) | 58.77 (23.58)
  Month 1: number analyzed (Participants) | 365 | 392 | 183
  Month 1 | 36.62 (23.72) | 32.78 (23.31) | 46.34 (24.47)
  Month 2: number analyzed (Participants) | 361 | 388 | 178
  Month 2 | 31.97 (22.94) | 30.33 (23.66) | 39.74 (23.72)
  Month 3: number analyzed (Participants) | 352 | 383 | 172
  Month 3 | 29.41 (21.53) | 27.07 (21.54) | 36.83 (21.99)
  Month 6: number analyzed (Participants) | 340 | 366 | 158
  Month 6 | 27.07 (21.21) | 24.22 (21.53) | 30.94 (22.87)
  Month 9: number analyzed (Participants) | 328 | 349 | 143
  Month 9 | 26.11 (20.35) | 23.76 (21.24) | 31.22 (22.50)
  Month 12: number analyzed (Participants) | 315 | 331 | 135
  Month 12 | 26.09 (21.29) | 22.64 (20.15) | 29.91 (20.76)
  Month 15: number analyzed (Participants) | 294 | 313 | 129
  Month 15 | 24.25 (20.39) | 23.72 (21.97) | 29.85 (22.94)
  Month 18: number analyzed (Participants) | 284 | 294 | 116
  Month 18 | 23.66 (19.29) | 22.72 (21.78) | 27.81 (20.66)
  Month 21: number analyzed (Participants) | 273 | 290 | 111
  Month 21 | 23.30 (19.86) | 22.85 (21.79) | 29.18 (21.46)
  Month 24: number analyzed (Participants) | 264 | 280 | 106
  Month 24 | 23.03 (19.80) | 21.09 (19.32) | 27.52 (20.28)

22. Secondary Outcome: Change From Baseline in Patient Assessment of Arthritis Pain
Description: Participants rated the severity of arthritis pain on a 0 to 100 mm VAS, where 0 mm=no pain and 100 mm=most severe pain.
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 365 | 392 | 183
mm
  Month 1 | -22.98 (1.17) | -27.26 (1.12) | -13.43 (1.62)
  Month 2: number analyzed (Participants) | 361 | 388 | 178
  Month 2 | -27.73 (1.17) | -29.71 (1.12) | -19.90 (1.64)
  Month 3: number analyzed (Participants) | 352 | 383 | 172
  Month 3 | -29.97 (1.18) | -32.90 (1.13) | -22.22 (1.66)
  Month 6: number analyzed (Participants) | 340 | 366 | 158
  Month 6 | -31.94 (1.19) | -35.35 (1.15) | -27.71 (1.70)
  Month 9: number analyzed (Participants) | 328 | 349 | 143
  Month 9 | -32.34 (1.21) | -35.26 (1.16) | -27.09 (1.75)
  Month 12: number analyzed (Participants) | 315 | 331 | 135
  Month 12 | -32.31 (1.22) | -35.85 (1.18) | -27.76 (1.79)
  Month 15: number analyzed (Participants) | 293 | 312 | 128
  Month 15 | -33.71 (1.25) | -34.54 (1.20) | -28.10 (1.82)
  Month 18: number analyzed (Participants) | 284 | 294 | 116
  Month 18 | -34.26 (1.26) | -35.73 (1.22) | -29.42 (1.87)
  Month 21: number analyzed (Participants) | 273 | 290 | 111
  Month 21 | -34.57 (1.27) | -35.66 (1.23) | -27.87 (1.90)
  Month 24: number analyzed (Participants) | 264 | 280 | 106
  Month 24 | -34.78 (1.28) | -37.57 (1.24) | -29.51 (1.93)

23. Secondary Outcome: Physician Global Assessment of Arthritis
Description: Physician Global Assessment of Arthritis was measured on a 0 to 100 mm VAS, where 0 mm=very good and 100 mm=very bad.
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 369 | 394 | 185
mm
  Baseline | 61.97 (16.45) | 60.50 (16.93) | 59.25 (17.70)
  Month 1: number analyzed (Participants) | 363 | 390 | 183
  Month 1 | 36.70 (19.24) | 33.05 (18.32) | 45.52 (19.73)
  Month 2: number analyzed (Participants) | 360 | 386 | 177
  Month 2 | 27.84 (18.26) | 25.80 (17.62) | 37.19 (18.61)
  Month 3: number analyzed (Participants) | 355 | 383 | 172
  Month 3 | 25.06 (17.10) | 22.80 (16.36) | 32.07 (17.28)
  Month 6: number analyzed (Participants) | 339 | 366 | 158
  Month 6 | 22.19 (17.31) | 18.32 (14.74) | 27.25 (16.80)
  Month 9: number analyzed (Participants) | 328 | 348 | 143
  Month 9 | 18.68 (15.09) | 16.61 (15.01) | 23.65 (16.55)
  Month 12: number analyzed (Participants) | 315 | 330 | 134
  Month 12 | 17.63 (15.09) | 14.19 (12.63) | 22.22 (15.30)
  Month 15: number analyzed (Participants) | 293 | 311 | 127
  Month 15 | 16.65 (14.03) | 14.97 (13.13) | 23.29 (17.36)
  Month 18: number analyzed (Participants) | 282 | 294 | 115
  Month 18 | 16.47 (12.70) | 14.02 (12.51) | 20.19 (14.74)
  Month 21: number analyzed (Participants) | 272 | 288 | 110
  Month 21 | 15.73 (12.73) | 14.61 (13.39) | 20.01 (14.02)
  Month 24: number analyzed (Participants) | 263 | 280 | 106
  Month 24 | 15.31 (14.14) | 14.42 (13.63) | 20.04 (15.54)

24. Secondary Outcome: Change From Baseline in Physician Global Assessment of Arthritis
Description: Physician Global Assessment of Arthritis was measured on a 0 to 100 mm VAS, where 0 mm=very good and 100 mm=very bad.
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 362 | 390 | 183
mm
  Month 1 | -24.89 (0.86) | -28.32 (0.82) | -15.79 (1.19)
  Month 2: number analyzed (Participants) | 357 | 385 | 177
  Month 2 | -33.92 (0.86) | -35.49 (0.82) | -24.17 (1.20)
  Month 3: number analyzed (Participants) | 351 | 380 | 171
  Month 3 | -36.41 (0.87) | -38.48 (0.83) | -28.62 (1.22)
  Month 6: number analyzed (Participants) | 336 | 363 | 157
  Month 6 | -39.04 (0.88) | -42.49 (0.84) | -33.41 (1.25)
  Month 9: number analyzed (Participants) | 324 | 345 | 142
  Month 9 | -42.09 (0.89) | -43.94 (0.85) | -36.54 (1.29)
  Month 12: number analyzed (Participants) | 312 | 328 | 133
  Month 12 | -43.07 (0.90) | -46.02 (0.87) | -37.43 (1.32)
  Month 15: number analyzed (Participants) | 291 | 309 | 126
  Month 15 | -43.91 (0.92) | -45.40 (0.88) | -36.17 (1.34)
  Month 18: number analyzed (Participants) | 281 | 292 | 114
  Month 18 | -44.00 (0.93) | -46.50 (0.90) | -38.65 (1.38)
  Month 21: number analyzed (Participants) | 270 | 288 | 109
  Month 21 | -44.76 (0.94) | -46.02 (0.90) | -38.92 (1.40)
  Month 24: number analyzed (Participants) | 261 | 279 | 105
  Month 24 | -45.07 (0.95) | -46.30 (0.91) | -38.93 (1.42)

25. Secondary Outcome: Patient Global Assessment of Arthritis
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS where 0=very well and 100=very poorly.
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
mm
  Baseline | 60.20 (24.56) | 60.88 (22.65) | 57.71 (24.30)
  Month 1: number analyzed (Participants) | 365 | 392 | 183
  Month 1 | 38.27 (24.83) | 32.63 (23.09) | 46.15 (22.82)
  Month 2: number analyzed (Participants) | 361 | 388 | 178
  Month 2 | 31.91 (22.90) | 28.94 (22.63) | 41.29 (22.73)
  Month 3: number analyzed (Participants) | 353 | 383 | 172
  Month 3 | 30.36 (21.78) | 28.60 (22.21) | 37.43 (21.20)
  Month 6: number analyzed (Participants) | 340 | 366 | 158
  Month 6 | 28.37 (21.23) | 24.84 (21.61) | 32.12 (21.92)
  Month 9: number analyzed (Participants) | 328 | 349 | 143
  Month 9 | 26.73 (20.38) | 24.98 (22.30) | 32.79 (22.42)
  Month 12: number analyzed (Participants) | 315 | 330 | 135
  Month 12 | 26.72 (20.84) | 24.38 (22.34) | 32.40 (21.69)
  Month 15: number analyzed (Participants) | 293 | 312 | 128
  Month 15 | 25.19 (20.12) | 23.79 (21.96) | 32.26 (22.79)
  Month 18: number analyzed (Participants) | 284 | 294 | 115
  Month 18 | 24.76 (19.93) | 24.38 (22.59) | 29.31 (20.91)
  Month 21: number analyzed (Participants) | 273 | 290 | 111
  Month 21 | 24.72 (20.93) | 23.86 (21.52) | 30.19 (21.15)
  Month 24: number analyzed (Participants) | 264 | 280 | 106
  Month 24 | 24.42 (21.43) | 23.61 (20.86) | 28.81 (20.54)

26. Secondary Outcome: Change From Baseline in Patient Global Assessment of Arthritis
Description: as for outcome 25
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 365 | 392 | 183
mm
  Month 1 | -22.22 (1.17) | -27.87 (1.12) | -14.12 (1.62)
  Month 2: number analyzed (Participants) | 361 | 388 | 178
  Month 2 | -28.74 (1.17) | -31.54 (1.12) | -18.86 (1.64)
  Month 3: number analyzed (Participants) | 353 | 383 | 172
  Month 3 | -30.03 (1.18) | -31.72 (1.13) | -22.18 (1.66)
  Month 6: number analyzed (Participants) | 340 | 366 | 158
  Month 6 | -31.65 (1.19) | -35.11 (1.15) | -27.00 (1.70)
  Month 9: number analyzed (Participants) | 328 | 349 | 143
  Month 9 | -32.70 (1.21) | -34.48 (1.16) | -26.15 (1.76)
  Month 12: number analyzed (Participants) | 315 | 330 | 135
  Month 12 | -32.75 (1.22) | -34.62 (1.18) | -26.07 (1.79)
  Month 15: number analyzed (Participants) | 293 | 312 | 128
  Month 15 | -33.82 (1.25) | -34.94 (1.20) | -26.70 (1.82)
  Month 18: number analyzed (Participants) | 284 | 294 | 116
  Month 18 | -34.18 (1.26) | -34.65 (1.22) | -28.64 (1.87)
  Month 21: number analyzed (Participants) | 273 | 290 | 111
  Month 21 | -34.18 (1.27) | -35.26 (1.23) | -27.56 (1.90)
  Month 24: number analyzed (Participants) | 264 | 280 | 106
  Month 24 | -34.41 (1.29) | -35.74 (1.24) | -28.81 (1.93)

27. Secondary Outcome: C-Reactive Protein
Description: CRP measured in milligrams per liter (mg/L)
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
mg/L
  Baseline | 22.68 (27.09) | 20.25 (23.92) | 25.92 (30.94)
  Month 1: number analyzed (Participants) | 366 | 390 | 184
  Month 1 | 6.62 (9.68) | 3.23 (5.35) | 17.37 (24.26)
  Month 2: number analyzed (Participants) | 360 | 386 | 176
  Month 2 | 6.47 (15.24) | 3.48 (9.38) | 16.12 (26.55)
  Month 3: number analyzed (Participants) | 353 | 384 | 172
  Month 3 | 6.75 (12.81) | 3.05 (5.60) | 11.90 (17.11)
  Month 6: number analyzed (Participants) | 339 | 366 | 158
  Month 6 | 5.22 (11.56) | 3.14 (5.51) | 12.21 (19.32)
  Month 9: number analyzed (Participants) | 327 | 349 | 143
  Month 9 | 6.01 (12.89) | 3.39 (6.32) | 8.18 (12.36)
  Month 12: number analyzed (Participants) | 314 | 330 | 135
  Month 12 | 5.26 (9.93) | 2.72 (4.46) | 9.64 (16.36)
  Month 15: number analyzed (Participants) | 290 | 311 | 128
  Month 15 | 5.57 (15.52) | 2.96 (4.40) | 8.61 (13.02)
  Month 18: number analyzed (Participants) | 280 | 291 | 116
  Month 18 | 4.57 (8.71) | 3.59 (11.42) | 8.98 (11.72)
  Month 21: number analyzed (Participants) | 272 | 288 | 111
  Month 21 | 4.89 (7.58) | 4.07 (8.12) | 9.54 (13.72)
  Month 24: number analyzed (Participants) | 262 | 279 | 103
  Month 24 | 5.57 (11.49) | 3.71 (7.00) | 10.07 (17.04)

28. Secondary Outcome: Change From Baseline in CRP
Description: Change from Baseline in CRP measured in mg/L.
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 366 | 390 | 184
mg/L
  Month 1 | -15.64 (0.68) | -18.84 (0.66) | -5.55 (0.95)
  Month 2: number analyzed (Participants) | 360 | 386 | 176
  Month 2 | -16.02 (0.69) | -18.59 (0.66) | -6.83 (0.97)
  Month 3: number analyzed (Participants) | 353 | 384 | 172
  Month 3 | -15.69 (0.69) | -19.01 (0.66) | -9.86 (0.97)
  Month 6: number analyzed (Participants) | 339 | 366 | 158
  Month 6 | -16.98 (0.70) | -18.76 (0.67) | -9.68 (1.00)
  Month 9: number analyzed (Participants) | 328 | 349 | 143
  Month 9 | -16.03 (0.71) | -18.48 (0.68) | -12.75 (1.03)
  Month 12: number analyzed (Participants) | 314 | 330 | 135
  Month 12 | -16.58 (0.72) | -19.16 (0.69) | -11.12 (1.05)
  Month 15: number analyzed (Participants) | 290 | 311 | 128
  Month 15 | -16.10 (0.73) | -18.80 (0.70) | -12.35 (1.07)
  Month 18: number analyzed (Participants) | 280 | 291 | 116
  Month 18 | -17.06 (0.74) | -18.17 (0.72) | -11.62 (1.10)
  Month 21: number analyzed (Participants) | 272 | 288 | 111
  Month 21 | -16.83 (0.75) | -17.67 (0.72) | -11.07 (1.11)
  Month 24: number analyzed (Participants) | 262 | 279 | 103
  Month 24 | -15.97 (0.75) | -17.96 (0.73) | -10.31 (1.14)

29. Secondary Outcome: Disease Activity Score Based on 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3) CRP
Description: DAS28-3(CRP) was calculated from the SJC and TJC using 28-joints count and CRP (mg/L). Total score range: 0 to approximately 10, higher score indicated more disease activity. DAS28-3(CRP) less than or equal to (≤)3.2 implied low disease activity, greater than (>)3.2 to 5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-3(CRP) less than (<)2.6 = remission.
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
units on a scale
  Baseline | 5.56 (0.91) | 5.46 (0.94) | 5.62 (0.95)
  Month 1: number analyzed (Participants) | 366 | 389 | 184
  Month 1 | 4.21 (1.08) | 3.77 (1.09) | 4.96 (1.17)
  Month 2: number analyzed (Participants) | 359 | 386 | 176
  Month 2 | 3.67 (1.21) | 3.31 (1.18) | 4.50 (1.19)
  Month 3: number analyzed (Participants) | 353 | 383 | 171
  Month 3 | 3.41 (1.21) | 3.05 (1.12) | 4.14 (1.27)
  Month 6: number analyzed (Participants) | 339 | 366 | 158
  Month 6 | 3.21 (1.25) | 2.76 (1.08) | 3.85 (1.34)
  Month 9: number analyzed (Participants) | 327 | 349 | 143
  Month 9 | 3.05 (1.22) | 2.69 (1.15) | 3.49 (1.20)
  Month 12: number analyzed (Participants) | 313 | 330 | 135
  Month 12 | 2.92 (1.18) | 2.52 (1.07) | 3.42 (1.30)
  Month 15: number analyzed (Participants) | 289 | 311 | 128
  Month 15 | 2.78 (1.10) | 2.50 (1.12) | 3.38 (1.27)
  Month 18: number analyzed (Participants) | 279 | 291 | 116
  Month 18 | 2.70 (1.06) | 2.47 (0.98) | 3.32 (1.17)
  Month 21: number analyzed (Participants) | 272 | 288 | 111
  Month 21 | 2.67 (1.10) | 2.48 (1.07) | 3.33 (1.27)
  Month 24: number analyzed (Participants) | 263 | 279 | 104
  Month 24 | 2.65 (1.08) | 2.44 (1.03) | 3.22 (1.15)

30. Secondary Outcome: Disease Activity Score Based on 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR])
Description: DAS28-4(ESR) was calculated from SJC and TJC using 28 joints count, ESR (millimeter/hour [mm/hour]) and patient's global assessment of disease activity (participant rated arthritis activity assessment). Total score range: 0 to approximately 10, higher score=more disease activity. DAS28-4(ESR) ≤3.2 implied low disease activity, >3.2 to 5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4(ESR) <2.6 = remission.
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 372 | 397 | 186
units on a scale
  Baseline | 6.62 (0.98) | 6.54 (0.96) | 6.60 (1.02)
  Month 1: number analyzed (Participants) | 338 | 369 | 167
  Month 1 | 5.18 (1.28) | 4.70 (1.32) | 5.84 (1.24)
  Month 2: number analyzed (Participants) | 333 | 366 | 163
  Month 2 | 4.54 (1.45) | 4.17 (1.39) | 5.35 (1.24)
  Month 3: number analyzed (Participants) | 329 | 360 | 159
  Month 3 | 4.21 (1.45) | 3.94 (1.31) | 4.98 (1.37)
  Month 6: number analyzed (Participants) | 319 | 345 | 146
  Month 6 | 4.05 (1.44) | 3.62 (1.31) | 4.61 (1.48)
  Month 9: number analyzed (Participants) | 305 | 329 | 132
  Month 9 | 3.84 (1.37) | 3.53 (1.36) | 4.27 (1.36)
  Month 12: number analyzed (Participants) | 292 | 309 | 123
  Month 12 | 3.69 (1.33) | 3.37 (1.29) | 4.23 (1.38)
  Month 15: number analyzed (Participants) | 276 | 293 | 116
  Month 15 | 3.59 (1.23) | 3.32 (1.31) | 4.17 (1.46)
  Month 18: number analyzed (Participants) | 264 | 272 | 106
  Month 18 | 3.51 (1.22) | 3.33 (1.18) | 4.05 (1.37)
  Month 21: number analyzed (Participants) | 254 | 269 | 100
  Month 21 | 3.49 (1.26) | 3.33 (1.29) | 4.09 (1.39)
  Month 24: number analyzed (Participants) | 238 | 254 | 92
  Month 24 | 3.43 (1.25) | 3.29 (1.29) | 3.99 (1.33)

31. Secondary Outcome: Change From Baseline in DAS28-3(CRP)
Description: DAS28-3(CRP) was calculated from the SJC and TJC using 28-joints count and CRP (mg/L). Total score range: 0 to approximately 10, higher score indicated more disease activity. DAS28-3(CRP) ≤3.2 implied low disease activity, >3.2 to 5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-3(CRP) <2.6 = remission.
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS; 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 366 | 389 | 184
units on a scale
  Month 1 | -1.30 (0.06) | -1.71 (0.06) | -0.58 (0.08)
  Month 2: number analyzed (Participants) | 359 | 386 | 176
  Month 2 | -1.85 (0.06) | -2.16 (0.06) | -1.02 (0.08)
  Month 3: number analyzed (Participants) | 353 | 383 | 171
  Month 3 | -2.09 (0.06) | -2.42 (0.06) | -1.36 (0.08)
  Month 6: number analyzed (Participants) | 339 | 366 | 158
  Month 6 | -2.27 (0.06) | -2.68 (0.06) | -1.62 (0.09)
  Month 9: number analyzed (Participants) | 327 | 349 | 143
  Month 9 | -2.40 (0.06) | -2.72 (0.06) | -1.95 (0.09)
  Month 12: number analyzed (Participants) | 313 | 330 | 135
  Month 12 | -2.52 (0.06) | -2.85 (0.06) | -1.99 (0.09)
  Month 15: number analyzed (Participants) | 289 | 311 | 128
  Month 15 | -2.65 (0.06) | -2.85 (0.06) | -2.03 (0.09)
  Month 18: number analyzed (Participants) | 279 | 291 | 116
  Month 18 | -2.72 (0.06) | -2.91 (0.06) | -2.05 (0.10)
  Month 21: number analyzed (Participants) | 272 | 288 | 111
  Month 21 | -2.75 (0.06) | -2.89 (0.06) | -2.05 (0.10)
  Month 24: number analyzed (Participants) | 263 | 279 | 104
  Month 24 | -2.76 (0.07) | -2.94 (0.06) | -2.12 (0.10)

32. Secondary Outcome: Change From Baseline in DAS28-4(ESR)
Description: DAS28-4(ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hour) and patient's global assessment of disease activity (participant rated arthritis activity assessment). Total score range: 0 to approximately 10, higher score=more disease activity. DAS28-4(ESR) ≤3.2 implied low disease activity, >3.2 to 5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4(ESR) <2.6 = remission.
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS; 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 338 | 369 | 167
units on a scale
  Month 1 | -1.40 (0.07) | -1.83 (0.07) | -0.72 (0.10)
  Month 2: number analyzed (Participants) | 333 | 366 | 163
  Month 2 | -2.03 (0.07) | -2.36 (0.07) | -1.17 (0.10)
  Month 3: number analyzed (Participants) | 329 | 360 | 159
  Month 3 | -2.34 (0.07) | -2.59 (0.07) | -1.53 (0.10)
  Month 6: number analyzed (Participants) | 319 | 345 | 146
  Month 6 | -2.47 (0.07) | -2.88 (0.07) | -1.87 (0.10)
  Month 9: number analyzed (Participants) | 305 | 329 | 132
  Month 9 | -2.64 (0.07) | -2.93 (0.07) | -2.19 (0.10)
  Month 12: number analyzed (Participants) | 292 | 309 | 123
  Month 12 | -2.78 (0.07) | -3.05 (0.07) | -2.20 (0.11)
  Month 15: number analyzed (Participants) | 276 | 293 | 116
  Month 15 | -2.87 (0.07) | -3.08 (0.07) | -2.25 (0.11)
  Month 18: number analyzed (Participants) | 264 | 272 | 106
  Month 18 | -2.92 (0.07) | -3.09 (0.07) | -2.34 (0.11)
  Month 21: number analyzed (Participants) | 254 | 269 | 100
  Month 21 | -2.96 (0.08) | -3.10 (0.07) | -2.30 (0.11)
  Month 24: number analyzed (Participants) | 238 | 254 | 92
  Month 24 | -2.99 (0.08) | -3.16 (0.07) | -2.40 (0.12)

33. Secondary Outcome: Percentage of Participants With DAS28-3(CRP) ≤3.2
Description: as for outcome 31
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS (NRI); 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 367 | 394 | 184
percentage of participants
  Month 1: number analyzed (Participants) | 366 | 389 | 184
  Month 1 | 16.67 | 33.16 | 5.98
  Month 2 | 35.42 | 47.97 | 14.13
  Month 3 | 40.33 | 56.85 | 19.57
  Month 6 | 47.68 | 62.69 | 27.72
  Month 9 | 52.04 | 60.41 | 33.15
  Month 12 | 52.59 | 64.97 | 32.61
  Month 15 | 53.41 | 58.88 | 29.89
  Month 18 | 52.59 | 56.09 | 25.00
  Month 21 | 52.59 | 55.84 | 28.26
  Month 24 | 52.32 | 56.85 | 29.35

34. Secondary Outcome: Percentage of Participants With DAS28-4(ESR) ≤3.2
Description: as for outcome 32
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS (NRI); 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 342 | 372 | 171
percentage of participants
  Month 1: number analyzed (Participants) | 338 | 369 | 167
  Month 1 | 7.40 | 14.09 | 2.99
  Month 2: number analyzed (Participants) | 342 | 372 | 170
  Month 2 | 18.42 | 25.81 | 4.71
  Month 3 | 25.15 | 30.38 | 9.94
  Month 6 | 27.78 | 38.17 | 14.04
  Month 9 | 29.24 | 39.78 | 18.13
  Month 12 | 33.33 | 41.13 | 18.71
  Month 15 | 33.04 | 40.86 | 18.13
  Month 18 | 32.16 | 35.22 | 16.37
  Month 21 | 34.21 | 38.17 | 16.37
  Month 24 | 34.80 | 36.02 | 15.79

35. Secondary Outcome: Percentage of Participants With DAS28-3(CRP) <2.6
Description: as for outcome 31
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS (NRI); 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 367 | 394 | 184
percentage of participants
  Month 1: number analyzed (Participants) | 366 | 389 | 184
  Month 1 | 7.38 | 14.14 | 2.72
  Month 2 | 20.44 | 28.68 | 5.43
  Month 3 | 25.89 | 37.82 | 9.78
  Month 6 | 31.34 | 47.21 | 15.22
  Month 9 | 36.24 | 45.69 | 17.39
  Month 12 | 36.51 | 49.49 | 20.65
  Month 15 | 37.60 | 49.24 | 19.57
  Month 18 | 38.42 | 44.67 | 19.02
  Month 21 | 37.06 | 44.67 | 17.39
  Month 24 | 38.42 | 43.91 | 18.48

36. Secondary Outcome: Percentage of Participants With DAS28-4(ESR) <2.6
Description: as for outcome 32
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS (NRI); 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 342 | 372 | 171
percentage of participants
  Month 1: number analyzed (Participants) | 338 | 369 | 167
  Month 1 | 2.07 | 5.69 | 0.00
  Month 2: number analyzed (Participants) | 342 | 372 | 170
  Month 2 | 9.06 | 12.90 | 2.35
  Month 3 | 13.74 | 17.47 | 4.68
  Month 6 | 14.62 | 21.77 | 7.60
  Month 9 | 16.37 | 23.66 | 9.94
  Month 12 | 18.71 | 23.39 | 11.70
  Month 15 | 16.37 | 24.19 | 12.87
  Month 18 | 16.96 | 19.89 | 11.11
  Month 21 | 18.42 | 21.42 | 8.77
  Month 24 | 20.76 | 22.31 | 9.94

37. Secondary Outcome: Percentage of Participants With DAS28-3(CRP) Response (Good or Moderate Improvement)
Description: DAS28-3(CRP) was calculated from the SJC and TJC using 28-joints count and CRP (mg/L). Total score range: 0 to approximately 10, higher score indicated more disease activity. DAS28 categorical responses define a good (absolute: <3.2 or >1.2 improvement from baseline [BL]), moderate (absolute: 3.2-5.1 or 0.6-1.2 change from BL), or no response (absolute: >5.1 or <0.6 change from BL).
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS (NRI); 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 367 | 394 | 184
percentage of participants
  Month 1: number analyzed (Participants) | 366 | 389 | 184
  Month 1 | 71.86 | 80.46 | 37.50
  Month 2 | 80.11 | 85.79 | 58.15
  Month 3 | 83.65 | 89.34 | 68.48
  Month 6 | 82.83 | 85.03 | 64.13
  Month 9 | 80.38 | 82.74 | 64.13
  Month 12 | 76.29 | 78.68 | 60.87
  Month 15 | 75.20 | 73.35 | 59.24
  Month 18 | 73.02 | 71.57 | 55.98
  Month 21 | 69.48 | 69.29 | 50.54
  Month 24 | 68.94 | 69.80 | 49.46

38. Secondary Outcome: Percentage of Participants With DAS28-4(ESR) Response (Good or Moderate Improvement)
Description: DAS28-4(ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hour) and patient's global assessment of disease activity (participant rated arthritis activity assessment). Total score range: 0 to approximately 10, higher score=more disease activity. DAS28 categorical responses define a good (absolute: <3.2 or >1.2 improvement from BL), moderate (absolute: 3.2-5.1 or 0.6-1.2 change from BL), or no response (absolute: >5.1 or <0.6 change from BL).
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS (NRI); 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 342 | 372 | 171
percentage of participants
  Month 1: number analyzed (Participants) | 338 | 369 | 167
  Month 1 | 62.43 | 74.25 | 33.53
  Month 2: number analyzed (Participants) | 342 | 372 | 170
  Month 2 | 74.27 | 82.26 | 50.00
  Month 3 | 80.41 | 88.17 | 66.67
  Month 6 | 78.95 | 84.14 | 60.82
  Month 9 | 78.36 | 81.72 | 61.40
  Month 12 | 76.61 | 79.57 | 59.65
  Month 15 | 74.85 | 73.12 | 56.73
  Month 18 | 70.18 | 70.97 | 52.05
  Month 21 | 69.88 | 69.89 | 48.54
  Month 24 | 68.71 | 69.62 | 49.12

39. Secondary Outcome: Percentage of Participants With an ACR70 Response Sustained at Least 6 Months
Description: as for outcome 14
Time Frame: Months 6, 9, 12, 15, 18, 21, and 24
Population: FAS, no imputation.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
percentage of participants | 28.42 | 38.54 | 13.98

40. Secondary Outcome: Percentage of Participants With Consecutive Visits of ACR20 Response by Number of Consecutive Visits
Description: as for outcome 15
Time Frame: Months 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS, no imputation.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
percentage of participants
  2 consecutive visits | 8.6 | 6.5 | 7.5
  3 consecutive visits | 8.6 | 11.1 | 14.5
  4 consecutive visits | 5.6 | 6.8 | 10.2
  5 consecutive visits | 7.0 | 4.3 | 5.4
  6 consecutive visits | 6.7 | 6.0 | 4.8
  7 consecutive visits | 6.7 | 6.8 | 5.9
  8 consecutive visits | 9.4 | 4.5 | 5.4
  9 consecutive visits | 9.7 | 11.6 | 9.7
  10 consecutive visits | 23.6 | 30.5 | 4.8

41. Secondary Outcome: Percentage of Participants With Consecutive Visits of ACR50 Response by Number of Consecutive Visits
Description: as for outcome 16
Time Frame: Months 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS, no imputation.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
percentage of participants
  2 consecutive visits | 9.9 | 9.8 | 9.1
  3 consecutive visits | 10.7 | 9.1 | 8.1
  4 consecutive visits | 6.4 | 7.3 | 5.4
  5 consecutive visits | 9.7 | 5.3 | 3.2
  6 consecutive visits | 4.6 | 4.8 | 5.4
  7 consecutive visits | 6.2 | 6.0 | 5.9
  8 consecutive visits | 5.6 | 7.1 | 2.2
  9 consecutive visits | 5.6 | 8.3 | 1.6
  10 consecutive visits | 5.9 | 11.8 | 1.1

42. Secondary Outcome: Percentage of Participants With Consecutive Visits of ACR70 Response by Number of Consecutive Visits
Description: as for outcome 14
Time Frame: Months 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS, no imputation.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
percentage of participants
  2 consecutive visits | 10.7 | 8.8 | 5.9
  3 consecutive visits | 5.9 | 7.8 | 3.8
  4 consecutive visits | 5.4 | 6.0 | 4.3
  5 consecutive visits | 4.3 | 5.8 | 1.6
  6 consecutive visits | 3.8 | 3.3 | 1.1
  7 consecutive visits | 2.9 | 4.8 | 2.7
  8 consecutive visits | 2.9 | 4.0 | NA — Values less than 1% were grouped and specific values labelled as 'not applicable'. Only 1 participant met this category
  9 consecutive visits | 3.2 | 5.8 | 1.1
  10 consecutive visits | 1.3 | 2.8 | 0

43. Secondary Outcome: Percentage of Participants With Consecutive Visits of DAS28-3(CRP) <2.6 by Number of Consecutive Visits
Description: as for outcome 31
Time Frame: Months 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS, no imputation.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
percentage of participants
  2 consecutive visits | 10.2 | 10.6 | 7.0
  3 consecutive visits | 8.6 | 8.6 | 7.0
  4 consecutive visits | 6.4 | 7.3 | 3.8
  5 consecutive visits | 5.1 | 5.5 | 4.3
  6 consecutive visits | 5.4 | 4.0 | 1.1
  7 consecutive visits | 4.0 | 7.3 | 1.6
  8 consecutive visits | 3.2 | 6.5 | 1.1
  9 consecutive visits | 4.0 | 7.6 | NA — Values less than 1% were grouped and specific values labelled as 'not applicable'. Only 1 participant met this category
  10 consecutive visits | 1.3 | 2.8 | NA — Values less than 1% were grouped and specific values labelled as 'not applicable'. Only 1 participant met this category

44. Secondary Outcome: Percentage of Participants With Consecutive Visits of DAS28-4(ESR) <2.6 by Number of Consecutive Visits
Description: as for outcome 32
Time Frame: Months 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS, no imputation.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 186
percentage of participants
  2 consecutive visits | 6.2 | 7.6 | 4.3
  3 consecutive visits | 5.4 | 5.3 | 2.7
  4 consecutive visits | 4.0 | 4.0 | 3.2
  5 consecutive visits | NA — Values less than 1% were grouped and specific values labelled as 'not applicable'. Only 2 participants met this category | 1.3 | 1.6
  6 consecutive visits | 2.4 | 2.0 | NA — Values less than 1% were grouped and specific values labelled as 'not applicable'. Only 1 participant met this category
  7 consecutive visits | 1.9 | 3.0 | NA — Values less than 1% were grouped and specific values labelled as 'not applicable'. Only 1 participant met this category
  8 consecutive visits | NA — Values less than 1% were grouped and specific values labelled as 'not applicable'. Only 2 participants met this category | 2.0 | 0
  9 consecutive visits | NA — Values less than 1% were grouped and specific values labelled as 'not applicable'. Only 2 participants met this category | 2.5 | 1.1
  10 consecutive visits | NA — Values less than 1% were grouped and specific values labelled as 'not applicable'. Only 2 participants met this category | NA — Values less than 1% were grouped and specific values labelled as 'not applicable'. Only 3 participants met this category | 0

45. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom, arise, eat, walk, hygiene, common activities over past week. Each item scored on 4-point scale from 0-3: 0=no difficulty, 1=some difficulty, 2=much difficulty, and 3=unable to do. Any activity that requires assistance from another individual or requires the use of an assistive device adjusts to a minimum score of 2 to represent a more limited functional status. Overall score was computed as sum of domain scores and divided by number of domains answered. Total possible score range 0-3: 0=least difficulty and 3=extreme difficulty.
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 396 | 186
units on a scale
  Baseline | 1.54 (0.65) | 1.50 (0.67) | 1.52 (0.65)
  Month 1: number analyzed (Participants) | 365 | 392 | 184
  Month 1 | 1.05 (0.67) | 0.89 (0.65) | 1.30 (0.67)
  Month 2: number analyzed (Participants) | 361 | 388 | 178
  Month 2 | 0.89 (0.67) | 0.74 (0.62) | 1.17 (0.66)
  Month 3: number analyzed (Participants) | 354 | 383 | 171
  Month 3 | 0.78 (0.64) | 0.67 (0.63) | 1.03 (0.63)
  Month 6: number analyzed (Participants) | 340 | 366 | 158
  Month 6 | 0.69 (0.64) | 0.57 (0.59) | 0.92 (0.62)
  Month 9: number analyzed (Participants) | 328 | 349 | 143
  Month 9 | 0.66 (0.62) | 0.56 (0.58) | 0.83 (0.57)
  Month 12: number analyzed (Participants) | 315 | 331 | 135
  Month 12 | 0.64 (0.61) | 0.51 (0.56) | 0.79 (0.58)
  Month 15: number analyzed (Participants) | 293 | 312 | 127
  Month 15 | 0.59 (0.59) | 0.51 (0.56) | 0.83 (0.64)
  Month 18: number analyzed (Participants) | 284 | 294 | 116
  Month 18 | 0.58 (0.58) | 0.48 (0.55) | 0.74 (0.60)
  Month 21: number analyzed (Participants) | 273 | 290 | 111
  Month 21 | 0.59 (0.58) | 0.49 (0.56) | 0.76 (0.64)
  Month 24: number analyzed (Participants) | 264 | 280 | 106
  Month 24 | 0.58 (0.60) | 0.48 (0.56) | 0.77 (0.64)

46. Secondary Outcome: Change From Baseline in HAQ-DI Score
Description: as for outcome 45
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS; 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 365 | 391 | 184
units on a scale
  Month 1 | -0.48 (0.03) | -0.62 (0.03) | -0.23 (0.04)
  Month 2: number analyzed (Participants) | 361 | 387 | 178
  Month 2 | -0.65 (0.03) | -0.77 (0.03) | -0.35 (0.4)
  Month 3: number analyzed (Participants) | 354 | 382 | 171
  Month 3 | -0.75 (0.03) | -0.85 (0.03) | -0.47 (0.04)
  Month 6: number analyzed (Participants) | 340 | 365 | 158
  Month 6 | -0.83 (0.03) | -0.94 (0.03) | -0.58 (0.04)
  Month 9: number analyzed (Participants) | 328 | 348 | 143
  Month 9 | -0.85 (0.03) | -0.95 (0.03) | -0.65 (0.04)
  Month 12: number analyzed (Participants) | 315 | 330 | 135
  Month 12 | -0.87 (0.03) | -0.98 (0.03) | -0.68 (0.04)
  Month 15: number analyzed (Participants) | 293 | 311 | 127
  Month 15 | -0.90 (0.03) | -0.98 (0.03) | -0.65 (0.05)
  Month 18: number analyzed (Participants) | 284 | 294 | 116
  Month 18 | -0.90 (0.03) | -1.01 (0.03) | -0.74 (0.05)
  Month 21: number analyzed (Participants) | 273 | 290 | 111
  Month 21 | -0.90 (0.03) | -1.00 (0.03) | -0.72 (0.05)
  Month 24: number analyzed (Participants) | 264 | 280 | 106
  Month 24 | -0.90 (0.03) | -1.01 (0.03) | -0.70 (0.05)

47. Secondary Outcome: Percentage of Participants With at Least 0.22 Improvement in HAQ-DI Score
Description: as for outcome 45
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS (NRI); 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 366 | 392 | 184
percentage of participants
  Month 1: number analyzed (Participants) | 365 | 391 | 184
  Month 1 | 64.38 | 73.91 | 45.65
  Month 2 | 69.13 | 79.85 | 61.41
  Month 3 | 72.95 | 80.36 | 65.22
  Month 6 | 74.32 | 77.81 | 63.04
  Month 9 | 73.50 | 73.21 | 61.41
  Month 12 | 68.03 | 71.43 | 58.70
  Month 15 | 65.30 | 67.86 | 51.63
  Month 18 | 64.21 | 64.80 | 48.91
  Month 21 | 62.30 | 65.05 | 46.74
  Month 24 | 60.11 | 65.05 | 46.74

48. Secondary Outcome: Percentage of Participants With at Least 0.3 Improvement in HAQ-DI Score
Description: as for outcome 45
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS (NRI); 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 366 | 392 | 184
percentage of participants
  Month 1: number analyzed (Participants) | 365 | 391 | 184
  Month 1 | 54.79 | 65.73 | 32.61
  Month 2 | 62.30 | 73.21 | 47.83
  Month 3 | 65.57 | 74.23 | 54.89
  Month 6 | 69.67 | 73.21 | 53.80
  Month 9 | 69.13 | 69.39 | 53.26
  Month 12 | 65.03 | 67.35 | 52.72
  Month 15 | 61.20 | 65.31 | 47.83
  Month 18 | 59.84 | 63.27 | 46.20
  Month 21 | 58.74 | 61.22 | 44.02
  Month 24 | 56.83 | 62.76 | 43.48

49. Secondary Outcome: Percentage of Participants With at Least 0.5 Improvement in HAQ-DI
Description: as for outcome 45
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS (NRI); 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Groups:
- MTX 10, 15 or 20 mg, Weekly: Participants received MTX capsules at doses of 10 to 20 mg per week and matching placebo CP-690,550 tablets, orally, BID, for up to 24 months. MTX dose was titrated to a maximum of 20 mg/week as follows: 10 mg/once weekly for 4 weeks, if tolerated the dose was titrated to 15 mg/once weekly for 4 weeks, if tolerated the dose was titrated to 20 mg/once weekly. One dose reduction was allowed for lack of tolerance.
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15 or 20 mg, Weekly
Number analyzed (Participants) | 366 | 392 | 184
percentage of participants
  Month 1: number analyzed (Participants) | 365 | 391 | 184
  Month 1 | 47.95 | 55.75 | 26.09
  Month 2 | 55.46 | 67.86 | 39.67
  Month 3 | 60.66 | 69.64 | 43.48
  Month 6 | 63.11 | 68.88 | 48.91
  Month 9 | 65.30 | 65.05 | 47.28
  Month 12 | 59.56 | 63.01 | 45.65
  Month 15 | 58.20 | 60.71 | 44.57
  Month 18 | 56.28 | 60.71 | 41.30
  Month 21 | 55.19 | 58.16 | 41.85
  Month 24 | 53.28 | 59.44 | 37.50

50. Secondary Outcome: Short Form 36 (SF-36) Mental Component Score
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning) and is reported as 2 summary scores; physical component score and mental component score. Total score range for the summary scores = 0-100, where higher score represents higher level of functioning.
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 395 | 185
units on a scale
  Baseline | 40.48 (12.00) | 40.73 (11.73) | 40.93 (11.27)
  Month 1: number analyzed (Participants) | 365 | 390 | 184
  Month 1 | 44.90 (11.40) | 46.70 (10.78) | 43.98 (10.71)
  Month 2: number analyzed (Participants) | 361 | 388 | 178
  Month 2 | 45.95 (12.10) | 46.09 (11.28) | 44.35 (10.48)
  Month 3: number analyzed (Participants) | 354 | 383 | 172
  Month 3 | 46.82 (11.21) | 46.59 (11.33) | 45.27 (10.42)
  Month 6: number analyzed (Participants) | 340 | 366 | 158
  Month 6 | 47.08 (10.97) | 47.55 (10.26) | 45.73 (12.06)
  Month 9: number analyzed (Participants) | 328 | 349 | 143
  Month 9 | 46.91 (10.74) | 48.04 (10.42) | 46.86 (10.85)
  Month 12: number analyzed (Participants) | 315 | 330 | 135
  Month 12 | 47.04 (10.67) | 48.05 (9.99) | 45.71 (11.01)
  Month 15: number analyzed (Participants) | 293 | 312 | 128
  Month 15 | 47.40 (10.31) | 48.04 (10.13) | 45.03 (11.75)
  Month 18: number analyzed (Participants) | 284 | 294 | 116
  Month 18 | 47.64 (10.32) | 48.25 (9.86) | 46.76 (11.49)
  Month 21: number analyzed (Participants) | 273 | 290 | 111
  Month 21 | 46.93 (10.85) | 48.50 (10.04) | 46.70 (11.66)
  Month 24: number analyzed (Participants) | 264 | 280 | 106
  Month 24 | 47.32 (10.23) | 48.96 (10.36) | 46.42 (10.62)

51. Secondary Outcome: SF-36 Physical Component Score
Description: as for outcome 50
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 395 | 185
units on a scale
  Baseline | 32.92 (7.36) | 33.20 (7.33) | 33.58 (7.82)
  Month 1: number analyzed (Participants) | 365 | 390 | 184
  Month 1 | 33.81 (8.47) | 40.61 (8.11) | 35.40 (8.28)
  Month 2: number analyzed (Participants) | 361 | 388 | 178
  Month 2 | 40.98 (8.44) | 42.52 (8.38) | 37.51 (8.22)
  Month 3: number analyzed (Participants) | 354 | 383 | 172
  Month 3 | 42.25 (8.57) | 43.35 (8.53) | 38.60 (8.01)
  Month 6: number analyzed (Participants) | 340 | 366 | 158
  Month 6 | 42.82 (8.42) | 44.34 (8.79) | 40.37 (8.11)
  Month 9: number analyzed (Participants) | 328 | 349 | 143
  Month 9 | 42.96 (8.69) | 44.77 (8.80) | 40.30 (7.97)
  Month 12: number analyzed (Participants) | 315 | 330 | 135
  Month 12 | 43.65 (8.68) | 45.72 (8.43) | 41.27 (8.05)
  Month 15: number analyzed (Participants) | 293 | 312 | 128
  Month 15 | 44.54 (8.83) | 45.62 (8.78) | 41.02 (8.27)
  Month 18: number analyzed (Participants) | 284 | 294 | 116
  Month 18 | 44.53 (8.42) | 45.50 (8.95) | 41.15 (8.50)
  Month 21: number analyzed (Participants) | 273 | 290 | 111
  Month 21 | 45.06 (8.36) | 45.56 (8.84) | 41.67 (8.44)
  Month 24: number analyzed (Participants) | 264 | 280 | 106
  Month 24 | 44.95 (8.76) | 45.78 (8.50) | 41.53 (8.30)

52. Secondary Outcome: Change From Baseline in SF-36 Mental Component Score
Description: as for outcome 50
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS; 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 365 | 389 | 183
units on a scale
  Month 1 | 4.37 (0.51) | 6.14 (0.49) | 3.25 (0.70)
  Month 2: number analyzed (Participants) | 361 | 386 | 177
  Month 2 | 5.39 (0.51) | 5.51 (0.49) | 3.41 (0.71)
  Month 3: number analyzed (Participants) | 354 | 381 | 171
  Month 3 | 6.12 (0.51) | 5.89 (0.49) | 4.33 (0.72)
  Month 6: number analyzed (Participants) | 340 | 365 | 157
  Month 6 | 6.36 (0.52) | 6.53 (0.50) | 4.84 (0.73)
  Month 9: number analyzed (Participants) | 328 | 349 | 142
  Month 9 | 5.99 (0.52) | 6.83 (0.50) | 6.04 (0.75)
  Month 12: number analyzed (Participants) | 315 | 330 | 134
  Month 12 | 6.21 (0.53) | 6.62 (0.51) | 4.72 (0.77)
  Month 15: number analyzed (Participants) | 293 | 312 | 127
  Month 15 | 6.38 (0.54) | 6.30 (0.52) | 4.09 (0.78)
  Month 18: number analyzed (Participants) | 284 | 294 | 115
  Month 18 | 6.51 (0.54) | 6.70 (0.52) | 5.78 (0.80)
  Month 21: number analyzed (Participants) | 273 | 290 | 110
  Month 21 | 5.80 (0.55) | 6.94 (0.53) | 5.58 (0.81)
  Month 24: number analyzed (Participants) | 264 | 280 | 106
  Month 24 | 6.23 (0.55) | 7.49 (0.53) | 5.54 (0.82)

53. Secondary Outcome: Change From Baseline in SF-36 Physical Component Score
Description: as for outcome 50
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS; 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 365 | 389 | 183
units on a scale
  Month 1 | 5.83 (0.43) | 7.54 (0.41) | 2.17 (0.59)
  Month 2: number analyzed (Participants) | 361 | 386 | 177
  Month 2 | 8.04 (0.43) | 9.45 (0.41) | 4.23 (0.60)
  Month 3: number analyzed (Participants) | 354 | 381 | 171
  Month 3 | 9.23 (0.43) | 10.32 (0.41) | 4.98 (0.60)
  Month 6: number analyzed (Participants) | 340 | 365 | 157
  Month 6 | 9.66 (0.44) | 11.24 (0.42) | 6.55 (0.62)
  Month 9: number analyzed (Participants) | 328 | 349 | 142
  Month 9 | 9.63 (0.44) | 11.53 (0.42) | 6.56 (0.63)
  Month 12: number analyzed (Participants) | 315 | 330 | 134
  Month 12 | 10.30 (0.44) | 12.35 (0.43) | 7.48 (0.65)
  Month 15: number analyzed (Participants) | 293 | 312 | 127
  Month 15 | 10.87 (0.45) | 12.06 (0.43) | 7.43 (0.65)
  Month 18: number analyzed (Participants) | 284 | 294 | 115
  Month 18 | 10.76 (0.45) | 12.04 (0.44) | 7.47 (0.67)
  Month 21: number analyzed (Participants) | 273 | 290 | 110
  Month 21 | 11.19 (0.46) | 12.19 (0.44) | 7.93 (0.68)
  Month 24: number analyzed (Participants) | 264 | 280 | 106
  Month 24 | 11.03 (0.46) | 12.46 (0.44) | 7.63 (0.68)

54. Secondary Outcome: SF-36 Domain Scores
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 396 | 186
units on a scale
  Baseline Vitality: number analyzed (Participants) | 373 | 395 | 186
  Baseline Vitality | 41.87 (9.90) | 41.63 (10.01) | 41.77 (9.56)
  Month 1 Vitality: number analyzed (Participants) | 365 | 392 | 184
  Month 1 Vitality | 47.94 (9.98) | 48.99 (9.55) | 44.83 (9.67)
  Month 2 Vitality: number analyzed (Participants) | 361 | 388 | 178
  Month 2 Vitality | 49.24 (10.90) | 49.68 (10.47) | 45.51 (9.53)
  Month 3 Vitality: number analyzed (Participants) | 354 | 383 | 172
  Month 3 Vitality | 50.10 (10.37) | 50.59 (10.00) | 47.06 (9.11)
  Month 6 Vitality: number analyzed (Participants) | 340 | 366 | 158
  Month 6 Vitality | 50.35 (10.09) | 50.69 (10.27) | 48.03 (9.87)
  Month 9 Vitality: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Vitality | 50.52 (10.05) | 51.34 (10.17) | 48.52 (9.79)
  Month 12 Vitality: number analyzed (Participants) | 315 | 331 | 135
  Month 12 Vitality | 50.43 (10.35) | 51.96 (9.50) | 48.83 (8.94)
  Month 15 Vitality: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Vitality | 51.40 (9.84) | 51.23 (9.89) | 48.21 (10.18)
  Month 18 Vitality: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Vitality | 51.18 (9.48) | 51.83 (9.62) | 48.93 (10.48)
  Month 21 Vitality: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Vitality | 51.29 (9.74) | 51.68 (9.86) | 49.26 (10.59)
  Month 24 Vitality: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Vitality | 50.81 (9.45) | 52.00 (10.12) | 49.07 (9.94)
  Baseline Social Functioning | 36.41 (11.32) | 36.66 (11.06) | 37.64 (11.32)
  Month 1 Social Functioning: number analyzed (Participants) | 365 | 392 | 184
  Month 1 Social Functioning | 41.33 (10.45) | 44.13 (9.85) | 40.12 (10.72)
  Month 2 Social Functioning: number analyzed (Participants) | 361 | 388 | 178
  Month 2 Social Functioning | 43.56 (10.89) | 43.78 (10.44) | 41.36 (10.28)
  Month 3 Social Functioning: number analyzed (Participants) | 354 | 383 | 172
  Month 3 Social Functioning | 44.75 (10.20) | 44.60 (10.49) | 42.52 (9.75)
  Month 6 Social Functioning: number analyzed (Participants) | 340 | 366 | 158
  Month 6 Social Functioning | 45.21 (9.97) | 46.18 (9.68) | 44.15 (10.42)
  Month 9 Social Functioning: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Social Functioning | 45.37 (9.47) | 46.46 (9.50) | 45.08 (9.71)
  Month 12 Social Functioning: number analyzed (Participants) | 315 | 331 | 135
  Month 12 Social Functioning | 45.43 (10.00) | 46.88 (9.45) | 43.22 (9.94)
  Month 15 Social Functioning: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Social Functioning | 46.09 (9.56) | 46.99 (9.25) | 42.96 (10.84)
  Month 18 Social Functioning: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Social Functioning | 46.39 (9.32) | 46.82 (9.34) | 44.44 (10.94)
  Month 21 Social Functioning: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Social Functioning | 46.22 (9.05) | 47.22 (9.61) | 44.49 (9.98)
  Month 24 Social Functioning: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Social Functioning | 46.52 (9.11) | 47.76 (9.27) | 43.87 (10.38)
  Basline Role Emotional | 34.01 (13.32) | 34.69 (13.06) | 34.69 (12.57)
  Month 1 Role Emotional: number analyzed (Participants) | 365 | 392 | 184
  Month 1 Role Emotional | 39.21 (12.35) | 41.31 (11.72) | 36.93 (12.10)
  Month 2 Role Emotional: number analyzed (Participants) | 361 | 388 | 178
  Month 2 Role Emotional | 40.59 (12.21) | 41.60 (11.62) | 38.30 (11.87)
  Month 3 Role Emotional: number analyzed (Participants) | 354 | 383 | 172
  Month 3 Role Emotional | 41.55 (11.59) | 42.18 (11.43) | 39.15 (11.72)
  Month 6 Role Emotional: number analyzed (Participants) | 340 | 366 | 158
  Month 6 Role Emotional | 41.95 (11.69) | 43.80 (10.75) | 40.34 (12.72)
  Month 9 Role Emotional: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Role Emotional | 41.84 (11.82) | 44.08 (10.85) | 41.12 (11.81)
  Month 12 Role Emotional: number analyzed (Participants) | 315 | 331 | 135
  Month 12 Role Emotional | 42.19 (11.43) | 44.29 (10.85) | 40.90 (11.62)
  Month 15 Role Emotional: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Role Emotional | 43.07 (10.93) | 44.72 (10.98) | 39.83 (12.09)
  Month 18 Role Emotional: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Role Emotional | 43.36 (11.02) | 44.00 (10.91) | 42.43 (11.81)
  Month 21 Role Emotional: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Role Emotional | 42.38 (11.44) | 44.53 (10.65) | 41.25 (12.14)
  Month 24 Role Emotional: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Role Emotional | 43.49 (11.12) | 45.27 (11.02) | 41.14 (11.68)
  Baseline Mental Health: number analyzed (Participants) | 373 | 395 | 186
  Baseline Mental Health | 38.87 (11.88) | 39.51 (11.76) | 39.75 (11.30)
  Month 1 Mental Health: number analyzed (Participants) | 365 | 392 | 184
  Month 1 Mental Health | 43.56 (11.28) | 45.59 (10.92) | 42.83 (10.84)
  Month 2 Mental Health: number analyzed (Participants) | 361 | 388 | 178
  Month 2 Mental Health | 44.57 (12.34) | 45.27 (11.43) | 43.35 (10.34)
  Month 3 Mental Health: number analyzed (Participants) | 354 | 383 | 172
  Month 3 Mental Health | 45.78 (11.73) | 45.71 (11.86) | 44.09 (10.55)
  Month 6 Mental Health: number analyzed (Participants) | 340 | 366 | 158
  Month 6 Mental Health | 46.21 (11.29) | 46.48 (11.07) | 44.06 (11.85)
  Month 9 Mental Health: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Mental Health | 45.85 (11.12) | 47.31 (10.93) | 45.41 (11.36)
  Month 12 Mental Health: number analyzed (Participants) | 315 | 331 | 135
  Month 12 Mental Health | 46.54 (11.33) | 47.43 (10.68) | 44.78 (11.25)
  Month 15 Mental Health: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Mental Health | 46.48 (10.87) | 47.16 (10.71) | 44.38 (11.92)
  Month 18 Mental Health: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Mental Health | 46.78 (10.82) | 48.05 (10.17) | 44.95 (12.62)
  Month 21 Mental Health: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Mental Health | 46.37 (11.64) | 48.06 (10.74) | 46.03 (12.31)
  Month 24 Mental Health: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Mental Health | 46.47 (10.53) | 48.18 (10.69) | 45.95 (10.96)
  Baseline Physical Functioning | 30.21 (9.47) | 31.57 (9.86) | 32.04 (9.57)
  Month 1 Physical Functioning: number analyzed (Participants) | 365 | 391 | 184
  Month 1 Physical Functioning | 36.41 (10.45) | 38.68 (10.31) | 32.82 (10.09)
  Month 2 Physical Functioning: number analyzed (Participants) | 361 | 388 | 178
  Month 2 Physical Functioning | 38.24 (11.05) | 40.41 (10.82) | 35.29 (10.26)
  Month 3 Physical Functioning: number analyzed (Participants) | 354 | 383 | 172
  Month 3 Physical Functioning | 39.91 (10.77) | 41.39 (10.84) | 36.12 (9.97)
  Month 6 Physical Functioning: number analyzed (Participants) | 340 | 366 | 158
  Month 6 Physical Functioning | 40.62 (10.98) | 42.79 (10.83) | 37.61 (10.17)
  Month 9 Physical Functioning: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Physical Functioning | 41.05 (11.03) | 43.45 (10.23) | 38.52 (10.34)
  Month 12 Physical Functioning: number analyzed (Participants) | 315 | 330 | 135
  Month 12 Physical Functioning | 41.72 (11.20) | 44.29 (10.17) | 39.66 (9.70)
  Month 15 Physical Functioning: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Physical Functioning | 42.67 (10.84) | 44.03 (10.58) | 38.85 (10.12)
  Month 18 Physical Functioning: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Physical Functioning | 43.06 (10.32) | 44.30 (10.64) | 39.01 (10.90)
  Month 21 Physical Functioning: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Physical Functioning | 43.01 (10.65) | 44.25 (10.31) | 39.32 (10.57)
  Month 24 Physical Functioning: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Physical Functioning | 43.45 (10.29) | 44.55 (10.40) | 39.85 (10.74)
  Baseline Role Physical | 33.54 (9.64) | 34.11 (9.35) | 33.98 (9.42)
  Month 1 Role Physical: number analyzed (Participants) | 365 | 392 | 184
  Month 1 Role Physical | 39.05 (9.74) | 41.30 (9.28) | 36.39 (9.36)
  Month 2 Role Physical: number analyzed (Participants) | 361 | 388 | 178
  Month 2 Role Physical | 41.30 (9.85) | 42.73 (9.58) | 38.43 (9.33)
  Month 3 Role Physical: number analyzed (Participants) | 354 | 383 | 172
  Month 3 Role Physical | 42.37 (9.83) | 43.51 (9.43) | 39.37 (9.67)
  Month 6 Role Physical: number analyzed (Participants) | 340 | 366 | 158
  Month 6 Role Physical | 43.27 (9.42) | 44.46 (9.82) | 40.78 (9.76)
  Month 9 Role Physical: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Role Physical | 42.78 (9.60) | 45.04 (9.47) | 40.80 (9.66)
  Month 12 Role Physical: number analyzed (Participants) | 315 | 331 | 135
  Month 12 Role Physical | 43.67 (9.36) | 45.81 (9.39) | 41.28 (9.28)
  Month 15 Role Physical: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Role Physical | 44.46 (9.41) | 45.90 (9.47) | 41.17 (9.35)
  Month 18 Role Physical: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Role Physical | 44.44 (90.4) | 45.27 (9.30) | 42.31 (10.15)
  Month 21 Role Physical: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Role Physical | 44.51 (9.18) | 45.77 (9.45) | 42.72 (9.72)
  Month 24 Role Physical: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Role Physical | 44.73 (9.34) | 46.20 (9.04) | 41.83 (10.15)
  Baseline Bodily Pain: number analyzed (Participants) | 373 | 396 | 185
  Baseline Bodily Pain | 33.29 (8.11) | 33.27 (7.25) | 33.80 (7.53)
  Month 1 Bodily Pain: number analyzed (Participants) | 365 | 391 | 184
  Month 1 Bodily Pain | 40.54 (8.47) | 42.81 (8.57) | 37.54 (7.55)
  Month 2 Bodily Pain: number analyzed (Participants) | 361 | 388 | 178
  Month 2 Bodily Pain | 42.78 (9.09) | 44.15 (9.19) | 38.93 (7.89)
  Month 3 Bodily Pain: number analyzed (Participants) | 354 | 383 | 172
  Month 3 Bodily Pain | 44.14 (8.73) | 44.79 (9.35) | 40.61 (8.19)
  Month 6 Bodily Pain: number analyzed (Participants) | 340 | 366 | 158
  Month 6 Bodily Pain | 44.44 (8.87) | 46.05 (9.47) | 42.36 (8.66)
  Month 9 Bodily Pain: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Bodily Pain | 44.37 (8.90) | 46.40 (9.58) | 42.62 (8.32)
  Month 12 Bodily Pain: number analyzed (Participants) | 315 | 331 | 135
  Month 12 Bodily Pain | 45.32 (9.32) | 47.17 (9.25) | 42.47 (8.85)
  Month 15 Bodily Pain: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Bodily Pain | 45.97 (9.38) | 47.18 (9.34) | 42.72 (9.75)
  Month 18 Bodily Pain: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Bodily Pain | 45.72 (9.26) | 47.38 (9.31) | 43.35 (9.25)
  Month 21 Bodily Pain: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Bodily Pain | 46.42 (9.30) | 47.43 (9.34) | 43.70 (9.47)
  Month 24 Bodily Pain: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Bodily Pain | 46.24 (9.46) | 47.66 (9.42) | 43.37 (9.43)
  Baseline General Health Perception | 38.02 (9.03) | 37.24 (8.55) | 37.63 (8.60)
  Month 1 General Health Perception: number analyzed (Participants) | 365 | 392 | 184
  Month 1 General Health Perception | 41.69 (9.37) | 42.40 (8.78) | 39.58 (8.69)
  Month 2 General Health Perception: number analyzed (Participants) | 361 | 388 | 178
  Month 2 General Health Perception | 43.11 (9.19) | 43.18 (9.19) | 40.68 (8.10)
  Month 3 General Health Perception: number analyzed (Participants) | 354 | 383 | 172
  Month 3 General Health Perception | 43.86 (9.43) | 43.72 (8.99) | 41.35 (8.07)
  Month 6 General Health Perception: number analyzed (Participants) | 340 | 366 | 158
  Month 6 General Health Perception | 44.00 (9.48) | 44.32 (9.24) | 42.53 (8.11)
  Month 9 General Health Perception: number analyzed (Participants) | 328 | 349 | 143
  Month 9 General Health Perception | 44.17 (9.32) | 44.53 (9.73) | 42.09 (8.51)
  Month 12 General Health Perception: number analyzed (Participants) | 315 | 331 | 135
  Month 12 General Health Perception | 44.24 (9.18) | 45.06 (9.35) | 42.74 (8.30)
  Month 15 General Health Perception: number analyzed (Participants) | 293 | 312 | 128
  Month 15 General Health Perception | 44.78 (9.23) | 45.14 (9.40) | 41.85 (8.40)
  Month 18 General Health Perception: number analyzed (Participants) | 284 | 294 | 116
  Month 18 General Health Perception | 44.92 (8.93) | 45.00 (9.60) | 42.15 (9.92)
  Month 21 General Health Perception: number analyzed (Participants) | 273 | 290 | 111
  Month 21 General Health Perception | 45.03 (9.08) | 45.02 (9.73) | 42.69 (9.06)
  Month 24 General Health Perception: number analyzed (Participants) | 264 | 280 | 106
  Month 24 General Health Perception | 44.75 (8.78) | 45.14 (9.41) | 42.75 (8.65)

55. Secondary Outcome: Change From Baseline in SF-36 Domain Scores
Description: as for outcome 54
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: FAS; 'n' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 365 | 391 | 184
units on a scale
  Month 1 Vitality: number analyzed (Participants) | 365 | 390 | 184
  Month 1 Vitality | 6.04 (0.49) | 7.27 (0.47) | 3.03 (0.68)
  Month 2 Vitality: number analyzed (Participants) | 361 | 386 | 178
  Month 2 Vitality | 7.36 (0.49) | 7.94 (0.47) | 3.68 (0.69)
  Month 3 Vitality: number analyzed (Participants) | 354 | 381 | 172
  Month 3 Vitality | 8.13 (0.49) | 8.79 (0.47) | 4.99 (0.69)
  Month 6 Vitality: number analyzed (Participants) | 340 | 365 | 158
  Month 6 Vitality | 8.36 (0.50) | 8.58 (0.48) | 5.89 (0.71)
  Month 9 Vitality: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Vitality | 8.32 (0.50) | 9.06 (0.49) | 6.33 (0.73)
  Month 12 Vitality: number analyzed (Participants) | 315 | 331 | 135
  Month 12 Vitality | 8.30 (0.51) | 9.31 (0.49) | 6.44 (0.74)
  Month 15 Vitality: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Vitality | 9.00 (0.52) | 8.33 (0.50) | 5.79 (0.75)
  Month 18 Vitality: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Vitality | 8.65 (0.52) | 9.09 (0.51) | 6.46 (0.77)
  Month 21 Vitality: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Vitality | 8.66 (0.53) | 8.94 (0.51) | 6.73 (0.78)
  Month 24 Vitality: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Vitality | 8.19 (0.53) | 9.29 (0.51) | 6.47 (0.79)
  Month 1 Social Functioning | 4.69 (0.50) | 7.46 (0.48) | 3.10 (0.69)
  Month 2 Social Functioning: number analyzed (Participants) | 361 | 387 | 178
  Month 2 Social Functioning | 6.97 (0.50) | 7.15 (0.48) | 4.18 (0.70)
  Month 3 Social Functioning: number analyzed (Participants) | 354 | 382 | 172
  Month 3 Social Functioning | 8.06 (0.50) | 7.90 (0.48) | 5.18 (0.71)
  Month 6 Social Functioning: number analyzed (Participants) | 340 | 366 | 158
  Month 6 Social Functioning | 8.35 (0.51) | 9.23 (0.49) | 6.82 (0.72)
  Month 9 Social Functioning: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Social Functioning | 8.39 (0.51) | 9.37 (0.49) | 7.78 (0.75)
  Month 12 Social Functioning: number analyzed (Participants) | 315 | 331 | 135
  Month 12 Social Functioning | 8.46 (0.52) | 9.60 (0.50) | 5.83 (0.76)
  Month 15 Social Functioning: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Social Functioning | 8.85 (0.53) | 9.49 (0.51) | 5.85 (0.77)
  Month 18 Social Functioning: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Social Functioning | 8.99 (0.54) | 9.44 (0.52) | 7.33 (0.79)
  Month 21 Social Functioning: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Social Functioning | 8.76 (0.54) | 9.87 (0.52) | 7.37 (0.80)
  Month 24 Social Functioning: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Social Functioning | 9.05 (0.55) | 10.43 (0.53) | 6.85 (0.82)
  Month 1 Role Emotional | 5.06 (0.56) | 6.88 (0.54) | 2.58 (0.77)
  Month 2 Role Emotional: number analyzed (Participants) | 361 | 387 | 178
  Month 2 Role Emotional | 6.39 (0.56) | 7.26 (0.54) | 3.62 (0.78)
  Month 3 Role Emotional: number analyzed (Participants) | 354 | 382 | 172
  Month 3 Role Emotional | 7.20 (0.56) | 7.73 (0.54) | 4.38 (0.79)
  Month 6 Role Emotional: number analyzed (Participants) | 340 | 366 | 158
  Month 6 Role Emotional | 7.49 (0.57) | 9.17 (0.55) | 5.58 (0.81)
  Month 9 Role Emotional: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Role Emotional | 7.21 (0.58) | 9.35 (0.55) | 6.37 (0.83)
  Month 12 Role Emotional: number analyzed (Participants) | 315 | 331 | 135
  Month 12 Role Emotional | 7.63 (0.58) | 9.38 (0.56) | 5.94 (0.85)
  Month 15 Role Emotional: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Role Emotional | 8.21 (0.59) | 9.61 (0.57) | 4.97 (0.86)
  Month 18 Role Emotional: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Role Emotional | 8.43 (0.60) | 9.16 (0.58) | 7.53 (0.89)
  Month 21 Role Emotional: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Role Emotional | 7.48 (0.60) | 9.70 (0.58) | 6.32 (0.90)
  Month 24 Role Emotional: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Role Emotional | 8.61 (0.61) | 10.51 (0.59) | 6.59 (0.91)
  Month 1 Mental Health: number analyzed (Participants) | 365 | 390 | 184
  Month 1 Mental Health | 4.57 (0.52) | 6.37 (0.50) | 3.50 (0.72)
  Month 2 Mental Health: number analyzed (Participants) | 361 | 386 | 178
  Month 2 Mental Health | 5.53 (0.52) | 6.05 (0.50) | 3.94 (0.72)
  Month 3 Mental Health: number analyzed (Participants) | 354 | 381 | 172
  Month 3 Mental Health | 6.59 (0.52) | 6.35 (0.50) | 4.67 (0.73)
  Month 6 Mental Health: number analyzed (Participants) | 340 | 365 | 158
  Month 6 Mental Health | 7.05 (0.53) | 6.81 (0.51) | 4.65 (0.75)
  Month 9 Mental Health: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Mental Health | 6.46 (0.53) | 7.39 (0.51) | 6.10 (0.77)
  Month 12 Mental Health: number analyzed (Participants) | 315 | 331 | 135
  Month 12 Mental Health | 7.27 (0.54) | 7.31 (0.52) | 5.38 (0.78)
  Month 15 Mental Health: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Mental Health | 7.01 (0.55) | 6.73 (0.53) | 5.02 (0.79)
  Month 18 Mental Health: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Mental Health | 7.21 (0.55) | 7.74 (0.54) | 5.41 (0.82)
  Month 21 Mental Health: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Mental Health | 6.78 (0.56) | 7.75 (0.54) | 6.39 (0.83)
  Month 24 Mental Health: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Mental Health | 6.88 (0.56) | 8.05 (0.54) | 6.40 (0.84)
  Month 1 Physical Functioning: number analyzed (Participants) | 365 | 390 | 184
  Month 1 Physical Functioning | 5.74 (0.52) | 7.41 (0.49) | 1.34 (0.71)
  Month 2 Physical Functioning: number analyzed (Participants) | 361 | 387 | 178
  Month 2 Physical Functioning | 7.59 (0.52) | 9.19 (0.50) | 3.66 (0.72)
  Month 3 Physical Functioning: number analyzed (Participants) | 354 | 382 | 172
  Month 3 Physical Functioning | 9.18 (0.52) | 10.16 (0.50) | 4.30 (0.73)
  Month 6 Physical Functioning: number analyzed (Participants) | 340 | 366 | 158
  Month 6 Physical Functioning | 9.70 (0.53) | 11.39 (0.50) | 5.69 (0.74)
  Month 9 Physical Functioning: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Physical Functioning | 9.98 (0.53) | 12.00 (0.51) | 6.32 (0.76)
  Month 12 Physical Functioning: number analyzed (Participants) | 315 | 330 | 135
  Month 12 Physical Functioning | 10.68 (0.54) | 12.76 (0.52) | 7.41 (0.77)
  Month 15 Physical Functioning: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Physical Functioning | 11.18 (0.55) | 12.29 (0.52) | 6.89 (0.79)
  Month 18 Physical Functioning: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Physical Functioning | 11.50 (0.55) | 12.66 (0.53) | 7.05 (0.81)
  Month 21 Physical Functioning: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Physical Functioning | 11.33 (0.55) | 12.71 (0.53) | 7.35 (0.82)
  Month 24 Physical Functioning: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Physical Functioning | 11.66 (0.56) | 13.04 (0.54) | 7.93 (0.83)
  Month 1 Role Physical | 5.52 (0.48) | 7.57 (0.46) | 2.75 (0.66)
  Month 2 Role Physical: number analyzed (Participants) | 361 | 387 | 178
  Month 2 Role Physical | 7.81 (0.48) | 9.05 (0.46) | 4.57 (0.67)
  Month 3 Role Physical: number analyzed (Participants) | 354 | 382 | 172
  Month 3 Role Physical | 8.77 (0.48) | 9.81 (0.46) | 5.24 (0.67)
  Month 6 Role Physical: number analyzed (Participants) | 340 | 366 | 158
  Month 6 Role Physical | 9.55 (0.49) | 10.63 (0.47) | 6.60 (0.69)
  Month 9 Role Physical: number analyzed (Participants) | 328 | 349 | 143
  Month 9 Role Physical | 8.88 (0.49) | 11.13 (0.47) | 6.57 (0.71)
  Month 12 Role Physical: number analyzed (Participants) | 315 | 331 | 135
  Month 12 Role Physical | 9.79 (0.50) | 11.72 (0.48) | 7.03 (0.72)
  Month 15 Role Physical: number analyzed (Participants) | 293 | 312 | 128
  Month 15 Role Physical | 10.27 (0.50) | 11.64 (0.49) | 7.06 (0.73)
  Month 18 Role Physical: number analyzed (Participants) | 284 | 294 | 116
  Month 18 Role Physical | 10.10 (0.51) | 11.23 (0.49) | 8.20 (0.75)
  Month 21 Role Physical: number analyzed (Participants) | 273 | 290 | 111
  Month 21 Role Physical | 10.11 (0.51) | 11.78 (0.49) | 8.65 (0.76)
  Month 24 Role Physical: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Role Physical | 10.31 (0.52) | 12.26 (0.50) | 7.78 (0.77)
  Month 1 Bodily Pain: number analyzed (Participants) | 365 | 390 | 183
  Month 1 Bodily Pain | 7.21 (0.48) | 9.54 (0.46) | 4.10 (0.66)
  Month 2 Bodily Pain: number analyzed (Participants) | 361 | 387 | 177
  Month 2 Bodily Pain | 9.45 (0.48) | 10.88 (0.46) | 5.40 (0.67)
  Month 3 Bodily Pain: number analyzed (Participants) | 354 | 382 | 171
  Month 3 Bodily Pain | 10.69 (0.48) | 11.49 (0.46) | 6.81 (0.68)
  Month 6 Bodily Pain: number analyzed (Participants) | 340 | 366 | 157
  Month 6 Bodily Pain | 10.90 (0.49) | 12.58 (0.47) | 8.32 (0.69)
  Month 9 Bodily Pain: number analyzed (Participants) | 328 | 349 | 142
  Month 9 Bodily Pain | 10.66 (0.49) | 12.74 (0.47) | 8.77 (0.71)
  Month 12 Bodily Pain: number analyzed (Participants) | 315 | 331 | 134
  Month 12 Bodily Pain | 11.64 (0.50) | 13.32 (0.48) | 8.43 (0.73)
  Month 15 Bodily Pain: number analyzed (Participants) | 293 | 312 | 127
  Month 15 Bodily Pain | 12.09 (0.51) | 13.10 (0.49) | 8.72 (0.74)
  Month 18 Bodily Pain: number analyzed (Participants) | 284 | 294 | 115
  Month 18 Bodily Pain | 11.75 (0.51) | 13.43 (0.50) | 9.11 (0.76)
  Month 21 Bodily Pain: number analyzed (Participants) | 273 | 290 | 110
  Month 21 Bodily Pain | 12.35 (0.52) | 13.52 (0.50) | 9.39 (0.77)
  Month 24 Bodily Pain: number analyzed (Participants) | 264 | 280 | 106
  Month 24 Bodily Pain | 12.16 (0.52) | 13.80 (0.50) | 9.06 (0.78)
  Month 1 General Health Perception | 3.94 (0.41) | 5.19 (0.39) | 2.15 (0.57)
  Month 2 General Health Perception: number analyzed (Participants) | 361 | 387 | 178
  Month 2 General Health Perception | 5.37 (0.41) | 5.97 (0.39) | 3.27 (0.57)
  Month 3 General Health Perception: number analyzed (Participants) | 354 | 382 | 172
  Month 3 General Health Perception | 6.04 (0.41) | 6.44 (0.39) | 3.86 (0.58)
  Month 6 General Health Perception: number analyzed (Participants) | 340 | 366 | 158
  Month 6 General Health Perception | 6.14 (0.42) | 6.84 (0.40) | 4.87 (0.59)
  Month 9 General Health Perception: number analyzed (Participants) | 328 | 349 | 143
  Month 9 General Health Perception | 6.08 (0.42) | 6.89 (0.40) | 4.71 (0.60)
  Month 12 General Health Perception: number analyzed (Participants) | 315 | 331 | 135
  Month 12 General Health Perception | 6.08 (0.42) | 7.20 (0.41) | 5.33 (0.61)
  Month 15 General Health Perception: number analyzed (Participants) | 293 | 312 | 128
  Month 15 General Health Perception | 6.41 (0.43) | 7.04 (0.41) | 4.57 (0.62)
  Month 18 General Health Perception: number analyzed (Participants) | 284 | 294 | 116
  Month 18 General Health Perception | 6.50 (0.43) | 6.95 (0.42) | 4.61 (0.64)
  Month 21 General Health Perception: number analyzed (Participants) | 273 | 290 | 111
  Month 21 General Health Perception | 6.62 (0.44) | 7.06 (0.42) | 4.96 (0.64)
  Month 24 General Health Perception: number analyzed (Participants) | 264 | 280 | 106
  Month 24 General Health Perception | 6.39 (0.44) | 7.37 (0.42) | 4.75 (0.65)

56. Secondary Outcome: Work Limitation Questionnaire (WLQ) Score
Description: WLQ: participant-reported 25-item scale to evaluate degree to which health problems interfere with an ability to perform job roles along 4 dimensions: Time Management scale (5-items); Physical Demands scale (6-item); Mental-Interpersonal Demands Scale (9-items); Output Demands scale (5-items). All the scales ranged from 0 (limited none of the time) to 100 (limited all of the time).
Time Frame: Baseline and Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 194 | 212 | 99
units on a scale
  Baseline: Time Management: number analyzed (Participants) | 187 | 209 | 97
  Baseline: Time Management | 46.41 (25.59) | 47.79 (28.29) | 47.26 (28.19)
  Baseline: Physical Demands: number analyzed (Participants) | 190 | 206 | 97
  Baseline: Physical Demands | 51.18 (23.02) | 50.99 (25.47) | 50.15 (25.54)
  Baseline: Mental Demands | 31.29 (24.72) | 33.84 (26.72) | 28.57 (26.35)
  Baseline: Output Demands: number analyzed (Participants) | 189 | 201 | 93
  Baseline: Output Demands | 40.77 (27.36) | 40.50 (28.07) | 38.34 (28.09)
  Month 1: Time Management: number analyzed (Participants) | 1 | 2 | 1
  Month 1: Time Management | 40.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 37.50 (53.03) | 40.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 2: Time Management: number analyzed (Participants) | 2 | 1 | 3
  Month 2: Time Management | 25.00 (35.36) | 15.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 95.00 (8.66)
  Month 3: Time Management: number analyzed (Participants) | 192 | 192 | 87
  Month 3: Time Management | 31.47 (27.99) | 29.02 (29.19) | 34.76 (27.70)
  Month 3: Physical Demands: number analyzed (Participants) | 190 | 195 | 85
  Month 3: Physical Demands | 48.11 (31.33) | 45.77 (32.86) | 54.47 (28.36)
  Month 3: Mental Demands: number analyzed (Participants) | 194 | 195 | 86
  Month 3: Mental Demands | 23.84 (26.67) | 22.50 (27.28) | 22.66 (24.71)
  Month 3: Output Demands: number analyzed (Participants) | 192 | 196 | 82
  Month 3: Output Demands | 26.46 (26.26) | 25.63 (28.30) | 27.77 (26.38)
  Month 6: Physical Demands: number analyzed (Participants) | 178 | 181 | 78
  Month 6: Physical Demands | 50.13 (31.81) | 45.76 (35.45) | 46.46 (30.78)
  Month 6: Time Management: number analyzed (Participants) | 175 | 180 | 76
  Month 6: Time Management | 29.18 (28.16) | 25.11 (28.08) | 27.87 (25.18)
  Month 6: Mental Demands: number analyzed (Participants) | 181 | 182 | 77
  Month 6: Mental Demands | 22.01 (24.05) | 18.00 (24.11) | 20.29 (23.90)
  Month 6: Output Demands: number analyzed (Participants) | 175 | 178 | 74
  Month 6: Output Demands | 24.55 (24.47) | 20.31 (23.33) | 24.66 (25.38)
  Month 9: Time Management: number analyzed (Participants) | 1 | 5 | 3
  Month 9: Time Management | 70.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 35.00 (33.91) | 62.92 (32.12)
  Month 12: Time Management: number analyzed (Participants) | 161 | 166 | 67
  Month 12: Time Management | 30.82 (29.76) | 24.43 (28.49) | 25.86 (25.57)
  Month 12: Physical Demands: number analyzed (Participants) | 164 | 166 | 68
  Month 12: Physical Demands | 47.87 (33.29) | 46.42 (37.18) | 39.98 (32.42)
  Month 12: Mental Demands: number analyzed (Participants) | 168 | 167 | 67
  Month 12: Mental Demands | 22.99 (25.59) | 15.11 (21.94) | 17.21 (21.88)
  Month 12: Output Demands: number analyzed (Participants) | 162 | 164 | 65
  Month 12: Output Demands | 25.65 (25.74) | 17.36 (22.98) | 21.49 (26.87)
  Month 15: Time Management: number analyzed (Participants) | 1 | 3 | 1
  Month 15: Time Management | 5.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 8.33 (14.43) | 75.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 15: Physical Demands: number analyzed (Participants) | 1 | 3 | 3
  Month 15: Physical Demands | 8.33 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 33.33 (57.74) | 54.17 (25.34)
  Month 15: Mental Demands: number analyzed (Participants) | 1 | 3 | 2
  Month 15: Mental Demands | 5.56 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 0.00 (0.00) | 37.50 (53.03)
  Month 15: Output Demands: number analyzed (Participants) | 1 | 3 | 2
  Month 15: Output Demands | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 6.67 (11.55) | 48.33 (44.78)
  Month 18: Time Management: number analyzed (Participants) | 149 | 147 | 57
  Month 18: Time Management | 23.19 (25.28) | 22.16 (26.77) | 25.09 (28.46)
  Month 18: Physical Demands: number analyzed (Participants) | 153 | 143 | 57
  Month 18: Physical Demands | 50.79 (34.51) | 43.14 (37.06) | 43.93 (33.15)
  Month 18: Mental Demands: number analyzed (Participants) | 153 | 147 | 58
  Month 18: Mental Demands | 19.24 (23.15) | 17.51 (23.83) | 17.78 (22.99)
  Month 18: Output Demands: number analyzed (Participants) | 158 | 144 | 57
  Month 18: Output Demands | 22.85 (24.60) | 19.83 (25.37) | 22.63 (26.31)
  Month 21: Time Management: number analyzed (Participants) | 2 | 2 | 1
  Month 21: Time Management | 67.50 (17.68) | 60.00 (35.36) | 80.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 21: Physical Demands: number analyzed (Participants) | 3 | 2 | 1
  Month 21: Physical Demands | 62.50 (29.17) | 27.08 (20.62) | 62.50 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 21: Mental Demands: number analyzed (Participants) | 3 | 2 | 1
  Month 21: Mental Demands | 29.63 (26.98) | 87.50 (17.68) | 25.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 21: Output Demands: number analyzed (Participants) | 3 | 2 | 1
  Month 21: Output Demands | 31.67 (27.54) | 82.50 (24.75) | 45.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 24: Time Management: number analyzed (Participants) | 138 | 140 | 52
  Month 24: Time Management | 28.17 (29.38) | 21.06 (25.37) | 25.11 (25.07)
  Month 24: Physical Demands: number analyzed (Participants) | 134 | 137 | 52
  Month 24: Physical Demands | 51.10 (35.26) | 45.94 (36.65) | 43.75 (33.06)
  Month 24: Mental Demands: number analyzed (Participants) | 143 | 141 | 55
  Month 24: Mental Demands | 19.44 (22.70) | 17.25 (23.29) | 17.50 (24.04)
  Month 24: Output Demands: number analyzed (Participants) | 141 | 141 | 55
  Month 24: Output Demands | 22.98 (25.23) | 19.39 (24.03) | 20.02 (23.85)

57. Secondary Outcome: Change From Baseline in WLQ Scores
Description: WLQ: participant-reported 25-item scale to evaluate degree to which health problems interfere with an ability to perform job roles along 4 dimensions: Time Management scale (5 items); Physical Demands scale (6 items); Mental-Interpersonal Demands Scale (9 items); Output Demands scale (5 items). All the scales ranged from 0 (limited none of the time) to 100 (limited all of the time).
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15 or 20 mg, Weekly
Number analyzed (Participants) | 170 | 177 | 81
units on a scale
  Month 3 Time Management Scale: number analyzed (Participants) | 165 | 174 | 81
  Month 3 Time Management Scale | -14.28 (2.11) | -16.87 (2.04) | -10.46 (2.98)
  Month 6 Time Management Scale: number analyzed (Participants) | 155 | 162 | 72
  Month 6 Time Management Scale | -16.99 (2.16) | -20.12 (2.10) | -15.78 (3.10)
  Month 12 Time Management Scale: number analyzed (Participants) | 141 | 143 | 62
  Month 12 Time Management Scale | -16.22 (2.23) | -20.72 (2.20) | -18.32 (3.29)
  Month 15 Time Management Scale: number analyzed (Participants) | 1 | 2 | 1
  Month 15 Time Management Scale | -32.18 (21.24) | -14.92 (15.04) | 29.59 (21.29)
  Month 18 Time Management Scale: number analyzed (Participants) | 124 | 125 | 53
  Month 18 Time Management Scale | -21.55 (2.33) | -22.60 (2.30) | -18.68 (3.47)
  Month 21 Time Management Scale: number analyzed (Participants) | 2 | 1 | 1
  Month 21 Time Management Scale | 5.99 (14.90) | -16.26 (20.82) | -7.27 (20.89)
  Month 24 Time Management Scale: number analyzed (Participants) | 117 | 118 | 46
  Month 24 Time Management Scale | -15.44 (2.37) | -22.25 (2.35) | -18.54 (3.64)
  Month 3 Physical Demand: number analyzed (Participants) | 164 | 172 | 78
  Month 3 Physical Demand | -6.44 (2.62) | -8.36 (2.55) | 0.13 (3.74)
  Month 6 Physical Demand: number analyzed (Participants) | 156 | 160 | 71
  Month 6 Physical Demand | -1.25 (2.68) | -9.48 (2.64) | -6.45 (3.88)
  Month 12 Physical Demand: number analyzed (Participants) | 142 | 142 | 62
  Month 12 Physical Demand | -5.36 (2.77) | -6.66 (2.76) | -14.62 (4.11)
  Month 15 Physical Demand: number analyzed (Participants) | 1 | 3 | 3
  Month 15 Physical Demand | -28.94 (28.32) | -12.26 (16.51) | -13.80 (16.68)
  Month 18 Physical Demand: number analyzed (Participants) | 130 | 119 | 53
  Month 18 Physical Demand | -2.35 (2.86) | -11.77 (2.95) | -7.77 (4.38)
  Month 21 Physical Demand: number analyzed (Participants) | 3 | 1 | 1
  Month 21 Physical Demand | 3.65 (16.22) | -18.17 (27.87) | 4.80 (27.94)
  Month 24 Physical Demand: number analyzed (Participants) | 113 | 112 | 46
  Month 24 Physical Demand | -2.71 (3.02) | -9.56 (3.03) | -8.03 (4.62)
  Month 3 Mental/Interpersonal Demands | -6.81 (1.68) | -8.56 (1.64) | -5.99 (2.39)
  Month 6 Mental/Interpersonal Demands: number analyzed (Participants) | 160 | 164 | 73
  Month 6 Mental/Interpersonal Demands | -10.03 (1.72) | -12.35 (1.69) | -9.36 (2.49)
  Month 12 Mental/Interpersonal Demands: number analyzed (Participants) | 146 | 145 | 63
  Month 12 Mental/Interpersonal Demands | -9.35 (1.77) | -15.21 (11.76) | -11.64 (2.63)
  Month 15 Mental/Interpersonal Demands: number analyzed (Participants) | 1 | 3 | 2
  Month 15 Mental/Interpersonal Demands | -17.52 (17.41) | -21.78 (10.18) | 15.00 (12.54)
  Month 18 Mental/Interpersonal Demands: number analyzed (Participants) | 132 | 125 | 55
  Month 18 Mental/Interpersonal Demands | -11.09 (1.83) | -13.08 (1.86) | -11.33 (2.76)
  Month 21 Mental/Interpersonal Demands: number analyzed (Participants) | 3 | 1 | 1
  Month 21 Mental/Interpersonal Demands | -4.00 (9.96) | 23.24 (17.09) | -29.23 (17.14)
  Month 24 Mental/Interpersonal Demands: number analyzed (Participants) | 121 | 117 | 49
  Month 24 Mental/Interpersonal Demands | -9.34 (1.89) | -13.58 (1.90) | -13.14 (2.87)
  Month 3 Output Demand: number analyzed (Participants) | 167 | 170 | 74
  Month 3 Output Demand | -12.69 (1.84) | -13.43 (1.82) | -8.73 (2.72)
  Month 6 Output Demand: number analyzed (Participants) | 155 | 154 | 68
  Month 6 Output Demand | -14.78 (1.89) | -19.16 (1.89) | -14.02 (2.80)
  Month 12 Output Demand: number analyzed (Participants) | 145 | 137 | 59
  Month 12 Output Demand | -14.83 (1.93) | -21.15 (1.96) | -15.84 (2.95)
  Month 15 Output Demand: number analyzed (Participants) | 1 | 3 | 2
  Month 15 Output Demand | -29.63 (18.09) | -18.43 (10.61) | 17.17 (13.10)
  Month 18 Output Demand: number analyzed (Participants) | 134 | 118 | 51
  Month 18 Output Demand | -14.17 (1.98) | -18.82 (2.06) | -14.15 (3.09)
  Month 21 Output Demand: number analyzed (Participants) | 2 | 1 | 1
  Month 21 Output Demand | 0.32 (12.69) | 16.85 (17.72) | -20.75 (17.79)
  Month 24 Output Demand: number analyzed (Participants) | 120 | 116 | 47
  Month 24 Output Demand | -13.60 (2.05) | -20.77 (2.08) | -16.40 (3.17)

58. Secondary Outcome: WLQ Work Loss Index Score
Description: WLQ: participant-reported 25-item scale to evaluate degree to which health problems interfere with an ability to perform job roles along 4 dimensions: Time Management scale (5-items); Physical Demands scale (6-item); Mental-Interpersonal Demands Scale (9-items); Output Demands scale (5-items). All the scales ranged from 0 (limited none of the time) to 100 (limited all of the time). Work Loss Index, which represented percentage of lost work over time period relative to a normative population, was derived (total score:0 [no loss] to 100 [complete loss of work]).
Time Frame: Baseline and Months 3, 6, and 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 199 | 215 | 99
units on a scale
  Baseline: number analyzed (Participants) | 197 | 215 | 99
  Baseline | 11.00 (5.93) | 11.21 (6.08) | 10.55 (6.24)
  Month 3: number analyzed (Participants) | 199 | 203 | 89
  Month 3 | 8.05 (6.25) | 7.60 (6.43) | 8.32 (5.78)
  Month 6: number analyzed (Participants) | 182 | 187 | 79
  Month 6 | 7.72 (5.74) | 6.49 (5.62) | 7.29 (5.69)
  Month 12: number analyzed (Participants) | 169 | 173 | 68
  Month 12 | 7.89 (6.07) | 5.88 (5.31) | 6.47 (5.90)

59. Secondary Outcome: Change From Baseline in WLQ Work Loss Index Score
Description: as for outcome 58
Time Frame: Months 3, 6, 12, 15, 18, 21, and 24
Population: FAS; 'n' (number of participants analyzed) signifies participants who were evaluable for this measure at a specific timepoint for each treatment group, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15 or 20 mg, Weekly
Number analyzed (Participants) | 176 | 185 | 83
units on a scale
  Month 3 | -2.82 (0.41) | -3.21 (0.40) | -2.03 (0.59)
  Month 6: number analyzed (Participants) | 163 | 168 | 74
  Month 6 | -3.24 (0.42) | -4.23 (0.41) | -3.18 (0.61)
  Month 12: number analyzed (Participants) | 149 | 151 | 64
  Month 12 | -3.35 (0.44) | -4.99 (0.43) | -3.84 (0.65)
  Month 15: number analyzed (Participants) | 1 | 3 | 3
  Month 15 | -7.10 (4.07) | -4.99 (2.39) | -0.19 (2.43)
  Month 18: number analyzed (Participants) | 137 | 129 | 55
  Month 18 | -3.61 (0.45) | -4.90 (0.45) | -3.48 (0.68)
  Month 21: number analyzed (Participants) | 3 | 1 | 1
  Month 21 | -1.14 (2.33) | 2.24 (3.99) | -4.92 (4.00)
  Month 24: number analyzed (Participants) | 125 | 121 | 50
  Month 24 | -3.18 (0.46) | -4.96 (0.46) | -4.11 (0.70)

60. Secondary Outcome: European Quality of Life (EuroQol) Five Dimensions (EQ-5D) Health State Profile Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline and Months 3, 6, 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 397 | 185
units on a scale
  Baseline | 0.39 (0.33) | 0.42 (0.31) | 0.46 (0.30)
  Month 3: number analyzed (Participants) | 352 | 381 | 171
  Month 3 | 0.67 (0.25) | 0.69 (0.23) | 0.63 (0.23)
  Month 6: number analyzed (Participants) | 338 | 364 | 158
  Month 6 | 0.68 (0.23) | 0.72 (0.22) | 0.63 (0.26)
  Month 12: number analyzed (Participants) | 315 | 330 | 135
  Month 12 | 0.70 (0.25) | 0.74 (0.22) | 0.66 (0.21)
  Month 18: number analyzed (Participants) | 284 | 293 | 116
  Month 18 | 0.73 (0.22) | 0.75 (0.23) | 0.66 (0.24)
  Month 24: number analyzed (Participants) | 262 | 279 | 105
  Month 24 | 0.72 (0.24) | 0.76 (0.22) | 0.71 (0.19)

61. Secondary Outcome: Change From Baseline in EQ-5D Health State Profile Utility Score
Description: as for outcome 60
Time Frame: Months 3, 6, 12, 18, and 24
Population: FAS; 'n' (number of participants analyzed) signifies participants who were evaluable for this measure at a given timepoints for each group, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 352 | 381 | 170
units on a scale
  Month 3 | 0.26 (0.01) | 0.28 (0.01) | 0.21 (0.02)
  Month 6: number analyzed (Participants) | 338 | 364 | 158
  Month 6 | 0.27 (0.01) | 0.30 (0.01) | 0.20 (0.02)
  Month 12: number analyzed (Participants) | 315 | 330 | 135
  Month 12 | 0.28 (0.01) | 0.31 (0.01) | 0.23 (0.02)
  Month 18: number analyzed (Participants) | 284 | 293 | 116
  Month 18 | 0.31 (0.01) | 0.33 (0.01) | 0.23 (0.02)
  Month 24: number analyzed (Participants) | 262 | 279 | 105
  Month 24 | 0.30 (0.01) | 0.33 (0.01) | 0.28 (0.02)

62. Secondary Outcome: Work Productivity and Healthcare Resource Utilization (HCRU) at Baseline and Months 3 and 6
Description: Rheumatoid Arthritis (RA)-HCRU assessed healthcare usage during last 3 months for direct, indirect medical cost domains. Direct cost: visit to doctor, non-medical practitioner, nursing home, hospital, surgery, emergency room (ER) treatment, diagnostic tests, overnight stay, home healthcare services, aids/devices used. Indirect costs associated with functional disability: employment status, willingness to work, work disability due to RA, sick leave, part time work, ability to perform chores, chores done by family/friends/housekeeper. Assessment was based on 0 to 2-point scale; higher score=higher medical cost.
Time Frame: Baseline and Months 3 and 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 372 | 396 | 186
units on a scale
  BL: seen any doctor: number analyzed (Participants) | 370 | 395 | 186
  BL: seen any doctor | 1.12 (0.33) | 1.13 (0.33) | 1.12 (0.32)
  BL: treated in ER: number analyzed (Participants) | 371 | 396 | 186
  BL: treated in ER | 1.95 (0.21) | 1.91 (0.28) | 1.91 (0.28)
  BL:admitted for overnight stay: number analyzed (Participants) | 17 | 35 | 16
  BL:admitted for overnight stay | 0.24 (0.56) | 0.31 (0.83) | 0.25 (0.58)
  BL: hospitalized | 1.89 (0.31) | 1.93 (0.26) | 1.88 (0.33)
  BL: any outpatient surgery | 1.98 (0.15) | 1.96 (0.19) | 1.98 (0.15)
  BL: non-study diagnostic tests | 1.74 (0.44) | 1.74 (0.44) | 1.69 (0.46)
  BL: in a nursing home: number analyzed (Participants) | 371 | 396 | 186
  BL: in a nursing home | 2.00 (0.00) | 1.99 (0.11) | 1.98 (0.13)
  BL: home healthcare services: number analyzed (Participants) | 371 | 396 | 186
  BL: home healthcare services | 1.99 (0.10) | 1.99 (0.11) | 1.98 (0.13)
  BL: used aids/devices | 1.90 (0.30) | 1.91 (0.29) | 1.91 (0.29)
  BL: non-medical practitioner | 1.97 (0.17) | 1.96 (0.20) | 1.96 (0.19)
  BL: currently employed: number analyzed (Participants) | 371 | 396 | 186
  BL: currently employed | 1.55 (0.50) | 1.53 (0.50) | 1.54 (0.50)
  BL: feel well enough to work: number analyzed (Participants) | 194 | 196 | 98
  BL: feel well enough to work | 1.78 (0.42) | 1.78 (0.42) | 1.78 (0.42)
  BL: unable to work due to RA: number analyzed (Participants) | 196 | 197 | 99
  BL: unable to work due to RA | 1.45 (0.50) | 1.49 (0.50) | 1.42 (0.50)
  BL: Lost job/retired early: number analyzed (Participants) | 194 | 195 | 98
  BL: Lost job/retired early | 1.75 (0.44) | 1.81 (0.40) | 1.77 (0.43)
  BL: work disabled due to RA: number analyzed (Participants) | 193 | 194 | 99
  BL: work disabled due to RA | 1.55 (0.50) | 1.58 (0.50) | 1.59 (0.50)
  BL: retired: number analyzed (Participants) | 194 | 201 | 101
  BL: retired | 1.60 (0.49) | 1.61 (0.49) | 1.53 (0.50)
  BL: sick leave due to RA: number analyzed (Participants) | 328 | 347 | 166
  BL: sick leave due to RA | 1.74 (0.44) | 1.73 (0.45) | 1.74 (0.44)
  BL: performed part time work: number analyzed (Participants) | 331 | 344 | 164
  BL: performed part time work | 1.90 (0.30) | 1.88 (0.33) | 1.83 (0.38)
  BL: performed paid work: number analyzed (Participants) | 330 | 349 | 163
  BL: performed paid work | 1.61 (0.49) | 1.57 (0.50) | 1.57 (0.50)
  BL: unable to do chores: number analyzed (Participants) | 369 | 394 | 186
  BL: unable to do chores | 1.41 (0.49) | 1.40 (0.49) | 1.44 (0.50)
  BL: chores by housekeeper: number analyzed (Participants) | 370 | 394 | 185
  BL: chores by housekeeper | 1.91 (0.29) | 1.87 (0.33) | 1.93 (0.26)
  BL: chores by family/friends: number analyzed (Participants) | 372 | 395 | 185
  BL: chores by family/friends | 1.48 (0.50) | 1.50 (0.50) | 1.49 (0.50)
  Month 3: seen any doctor: number analyzed (Participants) | 349 | 382 | 171
  Month 3: seen any doctor | 1.36 (0.48) | 1.30 (0.46) | 1.30 (0.46)
  Month 3: treated in ER: number analyzed (Participants) | 351 | 382 | 171
  Month 3: treated in ER | 1.97 (0.18) | 1.96 (0.20) | 1.98 (0.13)
  Month 3:admitted for overnight stay: number analyzed (Participants) | 12 | 16 | 3
  Month 3:admitted for overnight stay | 0.08 (0.29) | 0.06 (0.25) | 0.33 (0.58)
  Month 3:hospitalization: number analyzed (Participants) | 351 | 382 | 171
  Month 3:hospitalization | 1.99 (0.11) | 1.99 (0.09) | 1.99 (0.11)
  Month 3: outpatient surgery: number analyzed (Participants) | 351 | 382 | 171
  Month 3: outpatient surgery | 1.99 (0.12) | 1.98 (0.13) | 1.99 (0.11)
  Month 3: non-study diagnostic tests: number analyzed (Participants) | 351 | 382 | 171
  Month 3: non-study diagnostic tests | 1.90 (0.30) | 1.90 (0.31) | 1.92 (0.27)
  Month 3: in nursing home: number analyzed (Participants) | 351 | 382 | 171
  Month 3: in nursing home | 2.00 (0.05) | 1.99 (0.09) | 2.00 (0.00)
  Month 3: home healthcare services: number analyzed (Participants) | 351 | 382 | 171
  Month 3: home healthcare services | 2.00 (0.05) | 1.99 (0.10) | 2.00 (0.00)
  Month 3: required aids/devices: number analyzed (Participants) | 351 | 381 | 171
  Month 3: required aids/devices | 1.94 (0.23) | 1.95 (0.22) | 1.92 (0.27)
  Month 3: non-medical practitioner: number analyzed (Participants) | 351 | 382 | 171
  Month 3: non-medical practitioner | 1.98 (0.14) | 1.98 (0.12) | 1.99 (0.11)
  Month 3: currently employed: number analyzed (Participants) | 351 | 382 | 171
  Month 3: currently employed | 1.51 (0.50) | 1.53 (0.50) | 1.53 (0.50)
  Month 3: feel well enough to work: number analyzed (Participants) | 170 | 187 | 90
  Month 3: feel well enough to work | 1.62 (0.49) | 1.58 (0.50) | 1.67 (0.47)
  Month 3: unable to work due to RA: number analyzed (Participants) | 172 | 188 | 90
  Month 3: unable to work due to RA | 1.56 (0.50) | 1.64 (0.48) | 1.50 (0.50)
  Month 3: lost job/retired early: number analyzed (Participants) | 169 | 187 | 89
  Month 3: lost job/retired early | 1.70 (0.46) | 1.79 (0.41) | 1.83 (0.38)
  Month 3: work disabled due to RA: number analyzed (Participants) | 170 | 188 | 89
  Month 3: work disabled due to RA | 1.64 (0.48) | 1.68 (0.47) | 1.67 (0.47)
  Month 3: retired: number analyzed (Participants) | 171 | 190 | 91
  Month 3: retired | 1.56 (0.50) | 1.59 (0.49) | 1.54 (0.50)
  Month 3: sick leave due to RA: number analyzed (Participants) | 302 | 328 | 149
  Month 3: sick leave due to RA | 1.87 (0.33) | 1.90 (0.31) | 1.85 (0.36)
  Month 3: performed part-time work: number analyzed (Participants) | 301 | 326 | 147
  Month 3: performed part-time work | 1.93 (0.25) | 1.95 (0.21) | 1.92 (0.27)
  Month 3: performed paid work: number analyzed (Participants) | 304 | 331 | 146
  Month 3: performed paid work | 1.69 (0.46) | 1.72 (0.45) | 1.66 (0.47)
  Month 3: unable to do chores: number analyzed (Participants) | 350 | 381 | 171
  Month 3: unable to do chores | 1.69 (0.46) | 1.71 (0.45) | 1.54 (0.50)
  Month 3: chores by housekeeper: number analyzed (Participants) | 351 | 382 | 171
  Month 3: chores by housekeeper | 1.95 (0.22) | 1.92 (0.27) | 1.89 (0.31)
  Month 3: chores by family/friends: number analyzed (Participants) | 351 | 381 | 171
  Month 3: chores by family/friends | 1.70 (0.46) | 1.71 (0.45) | 1.58 (0.50)
  Month 6: seen any doctor: number analyzed (Participants) | 338 | 362 | 158
  Month 6: seen any doctor | 1.40 (0.49) | 1.39 (0.49) | 1.35 (0.48)
  Month 6: treated in ER: number analyzed (Participants) | 338 | 364 | 158
  Month 6: treated in ER | 1.96 (0.20) | 1.95 (0.22) | 1.98 (0.14)
  Month 6:admitted for overnight stay: number analyzed (Participants) | 14 | 19 | 3
  Month 6:admitted for overnight stay | 0.36 (0.74) | 0.21 (0.54) | 1.33 (1.15)
  Month 6: Hospitalization: number analyzed (Participants) | 338 | 364 | 158
  Month 6: Hospitalization | 1.99 (0.09) | 1.98 (0.14) | 1.97 (0.16)
  Month 6: outpatient surgery: number analyzed (Participants) | 338 | 364 | 158
  Month 6: outpatient surgery | 1.98 (0.13) | 1.98 (0.14) | 1.97 (0.16)
  Month 6: non-study diagnostic test: number analyzed (Participants) | 337 | 364 | 158
  Month 6: non-study diagnostic test | 1.91 (0.29) | 1.88 (0.32) | 1.89 (0.31)
  Month 6: in nursing home: number analyzed (Participants) | 338 | 364 | 158
  Month 6: in nursing home | 2.00 (0.05) | 2.00 (0.05) | 1.99 (0.08)
  Month 6: home healthcare services: number analyzed (Participants) | 338 | 364 | 158
  Month 6: home healthcare services | 1.99 (0.09) | 1.99 (0.07) | 2.00 (0.00)
  Month 6: required aids/devices: number analyzed (Participants) | 338 | 364 | 158
  Month 6: required aids/devices | 1.94 (0.24) | 1.96 (0.19) | 1.95 (0.22)
  Month 6: non-medical practitioner: number analyzed (Participants) | 338 | 364 | 158
  Month 6: non-medical practitioner | 1.99 (0.12) | 1.99 (0.07) | 1.97 (0.16)
  Month 6: currently employed: number analyzed (Participants) | 337 | 365 | 158
  Month 6: currently employed | 1.50 (0.50) | 1.53 (0.50) | 1.55 (0.50)
  Month 6: feel well enough to work: number analyzed (Participants) | 169 | 182 | 83
  Month 6: feel well enough to work | 1.55 (0.50) | 1.57 (0.50) | 1.65 (0.48)
  Month 6: unable to work due to RA: number analyzed (Participants) | 167 | 181 | 83
  Month 6: unable to work due to RA | 1.64 (0.48) | 1.66 (0.47) | 1.52 (0.50)
  Month 6: lost job/retired early: number analyzed (Participants) | 167 | 182 | 82
  Month 6: lost job/retired early | 1.74 (0.44) | 1.81 (0.40) | 1.78 (0.42)
  Month 6: work disabled due to RA: number analyzed (Participants) | 167 | 181 | 82
  Month 6: work disabled due to RA | 1.68 (0.47) | 1.70 (0.46) | 1.68 (0.47)
  Month 6: retired: number analyzed (Participants) | 167 | 190 | 85
  Month 6: retired | 1.55 (0.50) | 1.57 (0.50) | 1.52 (0.50)
  Month 6: sick leave due to RA: number analyzed (Participants) | 289 | 306 | 133
  Month 6: sick leave due to RA | 1.94 (0.24) | 1.94 (0.23) | 1.89 (0.31)
  Month 6: performed part-time work: number analyzed (Participants) | 289 | 303 | 132
  Month 6: performed part-time work | 1.97 (0.16) | 1.97 (0.17) | 1.95 (0.22)
  Month 6: performed paid work: number analyzed (Participants) | 289 | 306 | 132
  Month 6: performed paid work | 1.77 (0.42) | 1.82 (0.38) | 1.69 (0.46)
  Month 6: unable to do chores: number analyzed (Participants) | 335 | 360 | 158
  Month 6: unable to do chores | 1.79 (0.41) | 1.81 (0.40) | 1.70 (0.46)
  Month 6: chores by housekeeper: number analyzed (Participants) | 337 | 362 | 158
  Month 6: chores by housekeeper | 1.96 (0.20) | 1.94 (0.24) | 1.94 (0.24)
  Month 6: chores by family/friends: number analyzed (Participants) | 337 | 362 | 158
  Month 6: chores by family/friends | 1.78 (0.41) | 1.83 (0.37) | 1.71 (0.46)

63. Secondary Outcome: Work Productivity and Healthcare Resource Utilization (HCRU) at Months 12, 18, and 24
Description: RA-HCRU assessed healthcare usage during last 3 months for direct, indirect medical cost domains. Direct cost: visit to doctor, non-medical practitioner, nursing home, hospital, surgery, ER treatment, diagnostic tests, overnight stay, home healthcare services, aids/devices used. Indirect costs associated with functional disability: employment status, willingness to work, work disability due to RA, sick leave, part time work, ability to perform chores, chores done by family/friends/housekeeper. Assessment was based on 0 to 2-point scale; higher score=higher medical cost.
Time Frame: Months 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 314 | 328 | 135
units on a scale
  Month 12: seen any doctor: number analyzed (Participants) | 314 | 327 | 135
  Month 12: seen any doctor | 1.45 (0.50) | 1.44 (0.50) | 1.41 (0.49)
  Month 12: treated in ER | 1.95 (0.21) | 1.98 (0.15) | 1.96 (0.19)
  Month12:admitted for overnight stay: number analyzed (Participants) | 16 | 8 | 5
  Month12:admitted for overnight stay | 0.19 (0.54) | 0.25 (0.46) | 0.20 (0.45)
  Month 12: hospitalized | 1.98 (0.15) | 1.99 (0.11) | 1.99 (0.12)
  Month 12:any outpatient surgery | 1.97 (0.17) | 1.98 (0.15) | 1.98 (0.15)
  Month 12:non-study diagnostic tests | 1.90 (0.30) | 1.88 (0.33) | 1.92 (0.27)
  Month 12: in a nursing home | 2.00 (0.00) | 1.99 (0.08) | 1.99 (0.09)
  Month 12: home healthcare services: number analyzed (Participants) | 314 | 327 | 135
  Month 12: home healthcare services | 1.99 (0.08) | 1.99 (0.08) | 2.00 (0.00)
  Month 12: used aids/devices | 1.94 (0.24) | 1.97 (0.16) | 1.97 (0.17)
  Month 12: non-medical practitioner | 1.99 (0.08) | 1.99 (0.11) | 2.00 (0.00)
  Month 12: currently employed | 1.51 (0.50) | 1.53 (0.50) | 1.53 (0.50)
  Month 12: feel well enough to work: number analyzed (Participants) | 153 | 170 | 69
  Month 12: feel well enough to work | 1.61 (0.49) | 1.56 (0.50) | 1.61 (0.49)
  Month 12: unable to work due to RA: number analyzed (Participants) | 154 | 169 | 71
  Month 12: unable to work due to RA | 1.64 (0.48) | 1.73 (0.44) | 1.61 (0.49)
  Month 12: Lost job/retired early: number analyzed (Participants) | 154 | 168 | 70
  Month 12: Lost job/retired early | 1.75 (0.44) | 1.81 (0.39) | 1.80 (0.40)
  Month 12: work disabled due to RA: number analyzed (Participants) | 155 | 169 | 70
  Month 12: work disabled due to RA | 1.66 (0.48) | 1.73 (0.44) | 1.73 (0.45)
  Month 12: retired: number analyzed (Participants) | 156 | 170 | 72
  Month 12: retired | 1.51 (0.50) | 1.52 (0.50) | 1.42 (0.50)
  Month 12: sick leave due to RA: number analyzed (Participants) | 271 | 281 | 111
  Month 12: sick leave due to RA | 1.94 (0.24) | 1.98 (0.14) | 1.93 (0.26)
  Month 12: performed part time work: number analyzed (Participants) | 270 | 276 | 111
  Month 12: performed part time work | 1.97 (0.18) | 1.97 (0.16) | 1.97 (0.16)
  Month 12: performed paid work: number analyzed (Participants) | 269 | 275 | 111
  Month 12: performed paid work | 1.80 (0.40) | 1.84 (0.36) | 1.72 (0.45)
  Month 12: unable to do chores: number analyzed (Participants) | 312 | 327 | 135
  Month 12: unable to do chores | 1.79 (0.41) | 1.83 (0.37) | 1.79 (0.41)
  Month 12: chores by housekeeper | 1.96 (0.18) | 1.95 (0.21) | 1.96 (0.19)
  Month 12: chores by family/friends | 1.83 (0.38) | 1.86 (0.35) | 1.79 (0.41)
  Month 18: seen any doctor: number analyzed (Participants) | 283 | 292 | 116
  Month 18: seen any doctor | 1.43 (0.50) | 1.49 (0.50) | 1.41 (0.49)
  Month 18: treated in ER: number analyzed (Participants) | 283 | 292 | 116
  Month 18: treated in ER | 1.96 (0.18) | 1.97 (0.17) | 1.96 (0.20)
  Month18:admitted for overnight stay: number analyzed (Participants) | 10 | 9 | 5
  Month18:admitted for overnight stay | 0.60 (0.97) | 0.33 (0.71) | 0.40 (0.89)
  Month 18:hospitalization: number analyzed (Participants) | 283 | 292 | 116
  Month 18:hospitalization | 1.99 (0.10) | 1.98 (0.14) | 1.97 (0.16)
  Month 18: outpatient surgery: number analyzed (Participants) | 283 | 292 | 116
  Month 18: outpatient surgery | 1.98 (0.14) | 1.98 (0.15) | 1.97 (0.16)
  Month 18:non-study diagnostic tests: number analyzed (Participants) | 283 | 292 | 116
  Month 18:non-study diagnostic tests | 1.91 (0.29) | 1.91 (0.29) | 1.90 (0.31)
  Month 18: in nursing home: number analyzed (Participants) | 283 | 292 | 116
  Month 18: in nursing home | 2.00 (0.06) | 2.00 (0.00) | 2.00 (0.00)
  Month 18: home healthcare services: number analyzed (Participants) | 281 | 292 | 116
  Month 18: home healthcare services | 2.00 (0.06) | 2.00 (0.00) | 2.00 (0.00)
  Month 18: required aids/devices: number analyzed (Participants) | 283 | 292 | 116
  Month 18: required aids/devices | 1.96 (0.20) | 1.97 (0.16) | 1.97 (0.18)
  Month 18: non-medical practitioner: number analyzed (Participants) | 283 | 292 | 116
  Month 18: non-medical practitioner | 1.99 (0.08) | 1.99 (0.12) | 1.99 (0.09)
  Month 18: currently employed: number analyzed (Participants) | 283 | 292 | 116
  Month 18: currently employed | 1.50 (0.50) | 1.51 (0.50) | 1.55 (0.50)
  Month 18: feel well enough to work: number analyzed (Participants) | 136 | 145 | 60
  Month 18: feel well enough to work | 1.53 (0.50) | 1.57 (0.50) | 1.67 (0.48)
  Month 18: unable to work due to RA: number analyzed (Participants) | 137 | 145 | 61
  Month 18: unable to work due to RA | 1.73 (0.45) | 1.72 (0.45) | 1.59 (0.50)
  Month 18: lost job/retired early: number analyzed (Participants) | 135 | 143 | 61
  Month 18: lost job/retired early | 1.80 (0.40) | 1.83 (0.38) | 1.80 (0.40)
  Month 18: work disabled due to RA: number analyzed (Participants) | 135 | 145 | 61
  Month 18: work disabled due to RA | 1.76 (0.43) | 1.78 (0.42) | 1.66 (0.48)
  Month 18: retired: number analyzed (Participants) | 137 | 145 | 62
  Month 18: retired | 1.49 (0.50) | 1.53 (0.50) | 1.48 (0.50)
  Month 18: sick leave due to RA: number analyzed (Participants) | 252 | 253 | 96
  Month 18: sick leave due to RA | 1.94 (0.23) | 1.96 (0.20) | 1.95 (0.22)
  Month 18: performed part-time work: number analyzed (Participants) | 252 | 249 | 97
  Month 18: performed part-time work | 1.98 (0.15) | 1.98 (0.14) | 1.98 (0.14)
  Month 18: performed paid work: number analyzed (Participants) | 252 | 254 | 97
  Month 18: performed paid work | 1.78 (0.41) | 1.83 (0.38) | 1.79 (0.41)
  Month 18: unable to do chores: number analyzed (Participants) | 283 | 292 | 116
  Month 18: unable to do chores | 1.84 (0.36) | 1.84 (0.36) | 1.78 (0.42)
  Month 18: chores by housekeeper: number analyzed (Participants) | 283 | 292 | 116
  Month 18: chores by housekeeper | 1.98 (0.14) | 1.96 (0.20) | 1.95 (0.22)
  Month 18: chores by family/friends: number analyzed (Participants) | 283 | 292 | 116
  Month 18: chores by family/friends | 1.86 (0.35) | 1.89 (0.32) | 1.84 (0.37)
  Month 24: seen any doctor: number analyzed (Participants) | 262 | 278 | 105
  Month 24: seen any doctor | 1.46 (0.50) | 1.50 (0.50) | 1.47 (0.50)
  Month 24: treated in ER: number analyzed (Participants) | 263 | 279 | 106
  Month 24: treated in ER | 1.96 (0.19) | 1.96 (0.20) | 1.97 (0.17)
  Month24:admitted for overnight stay: number analyzed (Participants) | 10 | 12 | 3
  Month24:admitted for overnight stay | 0.20 (0.63) | 0.67 (0.98) | 0.00 (0.00)
  Month 24: Hospitalization: number analyzed (Participants) | 263 | 279 | 106
  Month 24: Hospitalization | 1.99 (0.11) | 1.99 (0.12) | 1.98 (0.14)
  Month 24: outpatient surgery: number analyzed (Participants) | 263 | 279 | 106
  Month 24: outpatient surgery | 1.98 (0.12) | 1.98 (0.13) | 1.99 (0.10)
  Month 24:non-study diagnostic test: number analyzed (Participants) | 263 | 278 | 106
  Month 24:non-study diagnostic test | 1.92 (0.27) | 1.89 (0.32) | 1.86 (0.35)
  Month 24: in nursing home: number analyzed (Participants) | 263 | 279 | 106
  Month 24: in nursing home | 2.00 (0.06) | 1.99 (0.08) | 1.98 (0.14)
  Month 24: home healthcare services: number analyzed (Participants) | 262 | 278 | 106
  Month 24: home healthcare services | 2.00 (0.00) | 1.99 (0.10) | 1.99 (0.10)
  Month 24: required aids/devices: number analyzed (Participants) | 263 | 279 | 106
  Month 24: required aids/devices | 1.95 (0.22) | 1.96 (0.20) | 1.96 (0.19)
  Month 24: non-medical practitioner: number analyzed (Participants) | 263 | 279 | 106
  Month 24: non-medical practitioner | 1.99 (0.11) | 1.98 (0.13) | 2.00 (0.00)
  Month 24: currently employed: number analyzed (Participants) | 263 | 279 | 106
  Month 24: currently employed | 1.49 (0.50) | 1.54 (0.50) | 1.55 (0.50)
  Month 24: feel well enough to work: number analyzed (Participants) | 119 | 138 | 54
  Month 24: feel well enough to work | 1.55 (0.50) | 1.57 (0.50) | 1.65 (0.48)
  Month 24: unable to work due to RA: number analyzed (Participants) | 118 | 138 | 54
  Month 24: unable to work due to RA | 1.70 (0.46) | 1.75 (0.43) | 1.52 (0.50)
  Month 24: lost job/retired early: number analyzed (Participants) | 116 | 137 | 54
  Month 24: lost job/retired early | 1.76 (0.43) | 1.83 (0.38) | 1.81 (0.39)
  Month 24: work disabled due to RA: number analyzed (Participants) | 117 | 137 | 54
  Month 24: work disabled due to RA | 1.75 (0.43) | 1.77 (0.42) | 1.70 (0.46)
  Month 24: retired: number analyzed (Participants) | 119 | 141 | 56
  Month 24: retired | 1.47 (0.50) | 1.49 (0.50) | 1.52 (0.50)
  Month 24: sick leave due to RA: number analyzed (Participants) | 224 | 240 | 87
  Month 24: sick leave due to RA | 1.96 (0.20) | 1.98 (0.13) | 1.90 (0.31)
  Month 24: performed part-time work: number analyzed (Participants) | 223 | 236 | 87
  Month 24: performed part-time work | 1.98 (0.15) | 1.99 (0.09) | 1.95 (0.21)
  Month 24: performed paid work: number analyzed (Participants) | 223 | 238 | 88
  Month 24: performed paid work | 1.82 (0.39) | 1.82 (0.39) | 1.75 (0.44)
  Month 24: unable to do chores: number analyzed (Participants) | 262 | 279 | 106
  Month 24: unable to do chores | 1.83 (0.37) | 1.86 (0.35) | 1.80 (0.40)
  Month 24: chores by housekeeper: number analyzed (Participants) | 263 | 279 | 106
  Month 24: chores by housekeeper | 1.96 (0.19) | 1.96 (0.20) | 1.97 (0.17)
  Month 24: chores by family/friends: number analyzed (Participants) | 263 | 279 | 106
  Month 24: chores by family/friends | 1.87 (0.34) | 1.88 (0.33) | 1.81 (0.39)

64. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Baseline and Months 3 and 6
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA/non-RA related number of events including visits to doctor, non-medical practitioner, hospital ER treatment, hospitalizations, number of surgeries, diagnostic tests, and devices/aids used were reported.
Time Frame: Baseline and Months 3 and 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 326 | 345 | 165
events
  BL: doctor visits: number analyzed (Participants) | 324 | 345 | 164
  BL: doctor visits | 4.81 (5.57) | 4.37 (3.86) | 4.82 (5.31)
  BL: RA-related doctor visits | 1.55 (1.07) | 1.46 (0.95) | 1.56 (0.96)
  BL: hospital ER visit: number analyzed (Participants) | 16 | 35 | 13
  BL: hospital ER visit | 2.13 (2.73) | 1.49 (0.98) | 1.38 (0.65)
  BL: RA-related ER visits: number analyzed (Participants) | 17 | 36 | 16
  BL: RA-related ER visits | 1.12 (0.86) | 1.00 (0.83) | 1.13 (1.02)
  BL: hospitalization: number analyzed (Participants) | 39 | 29 | 22
  BL: hospitalization | 1.03 (0.16) | 1.00 (0.00) | 1.05 (0.21)
  BL: RA-related hospitalization: number analyzed (Participants) | 41 | 29 | 23
  BL: RA-related hospitalization | 1.27 (0.55) | 1.24 (0.69) | 1.13 (0.55)
  BL: outpatient surgery: number analyzed (Participants) | 9 | 15 | 4
  BL: outpatient surgery | 2.56 (3.24) | 2.13 (2.61) | 1.25 (0.50)
  BL: RA-related outpatient surgery: number analyzed (Participants) | 9 | 15 | 4
  BL: RA-related outpatient surgery | 0.33 (0.50) | 0.80 (0.86) | 0.00 (0.00)
  BL:non-study diagnostic tests: number analyzed (Participants) | 91 | 103 | 56
  BL:non-study diagnostic tests | 2.25 (1.60) | 2.05 (1.27) | 1.75 (1.18)
  BL: RA-related diagnostic tests: number analyzed (Participants) | 94 | 103 | 57
  BL: RA-related diagnostic tests | 1.20 (1.22) | 1.21 (1.21) | 1.09 (0.91)
  BL: non-medical practitioner visits: number analyzed (Participants) | 11 | 15 | 7
  BL: non-medical practitioner visits | 23.82 (56.10) | 10.07 (19.72) | 8.57 (11.13)
  BL: RA-related non-medical visits: number analyzed (Participants) | 10 | 16 | 7
  BL: RA-related non-medical visits | 1.00 (0.82) | 1.13 (0.81) | 1.14 (0.69)
  Month 3: doctor visits: number analyzed (Participants) | 225 | 266 | 121
  Month 3: doctor visits | 3.45 (2.99) | 3.44 (3.12) | 3.57 (2.94)
  Month 3: RA-related doctor visits: number analyzed (Participants) | 226 | 267 | 121
  Month 3: RA-related doctor visits | 0.99 (0.77) | 0.96 (0.62) | 1.03 (0.72)
  Month 3: hospital ER visits: number analyzed (Participants) | 12 | 16 | 3
  Month 3: hospital ER visits | 1.83 (1.34) | 1.94 (2.08) | 1.00 (0.00)
  Month 3: RA-related ER visits: number analyzed (Participants) | 12 | 16 | 3
  Month 3: RA-related ER visits | 0.33 (0.65) | 0.13 (0.34) | 0.00 (0.00)
  Month 3: hospitalization: number analyzed (Participants) | 4 | 3 | 2
  Month 3: hospitalization | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00)
  Month 3: RA-related hospitalization: number analyzed (Participants) | 4 | 3 | 2
  Month 3: RA-related hospitalization | 0.25 (0.50) | 0.33 (0.58) | 0.50 (0.71)
  Month 3: outpatient surgery: number analyzed (Participants) | 4 | 7 | 2
  Month 3: outpatient surgery | 1.25 (0.50) | 1.00 (0.00) | 1.00 (0.00)
  Month 3:RA-related outpatient surgery: number analyzed (Participants) | 5 | 7 | 2
  Month 3:RA-related outpatient surgery | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Month 3: non-study diagnostic tests: number analyzed (Participants) | 34 | 40 | 14
  Month 3: non-study diagnostic tests | 1.32 (0.64) | 1.33 (0.73) | 1.57 (1.02)
  Month 3: RA-related diagnostic tests: number analyzed (Participants) | 34 | 41 | 14
  Month 3: RA-related diagnostic tests | 0.18 (0.39) | 0.27 (0.50) | 0.21 (0.80)
  Month 3:non-medical practitioner visits: number analyzed (Participants) | 6 | 6 | 2
  Month 3:non-medical practitioner visits | 10.33 (15.13) | 4.50 (2.43) | 9.00 (7.07)
  Month 3:RA-related non-medical visits: number analyzed (Participants) | 6 | 6 | 2
  Month 3:RA-related non-medical visits | 0.67 (0.82) | 1.00 (0.63) | 2.00 (0.00)
  Month 6: doctor visits: number analyzed (Participants) | 201 | 223 | 103
  Month 6: doctor visits | 2.57 (3.64) | 2.48 (2.82) | 2.12 (1.72)
  Month 6: RA-related doctor visits: number analyzed (Participants) | 204 | 224 | 103
  Month 6: RA-related doctor visits | 0.82 (0.72) | 0.74 (0.64) | 0.74 (0.54)
  Month 6: hospital ER visits: number analyzed (Participants) | 14 | 18 | 3
  Month 6: hospital ER visits | 1.36 (0.84) | 1.22 (0.73) | 5.33 (5.86)
  Month 6: RA-related ER visits: number analyzed (Participants) | 15 | 19 | 3
  Month 6: RA-related ER visits | 0.07 (0.26) | 0.26 (0.65) | 1.00 (1.00)
  Month 6: hospitalization: number analyzed (Participants) | 3 | 7 | 4
  Month 6: hospitalization | 1.00 (0.00) | 2.29 (3.40) | 1.00 (0.00)
  Month 6: RA-related hospitalization: number analyzed (Participants) | 3 | 7 | 4
  Month 6: RA-related hospitalization | 0.00 (0.00) | 0.14 (0.38) | 0.75 (0.96)
  Month 6: outpatient surgery: number analyzed (Participants) | 6 | 7 | 4
  Month 6: outpatient surgery | 1.50 (1.22) | 1.43 (0.79) | 1.25 (0.50)
  Month 6:RA-related outpatient surgery: number analyzed (Participants) | 6 | 7 | 4
  Month 6:RA-related outpatient surgery | 0.00 (0.00) | 0.14 (0.38) | 0.25 (0.50)
  Month 6: non-study diagnostic tests: number analyzed (Participants) | 30 | 41 | 17
  Month 6: non-study diagnostic tests | 1.73 (1.39) | 1.54 (1.00) | 1.47 (0.94)
  Month 6: RA related diagnostic tests: number analyzed (Participants) | 31 | 41 | 17
  Month 6: RA related diagnostic tests | 0.26 (0.63) | 0.12 (0.40) | 0.35 (0.79)
  Month 6:non-medical practitioner visits: number analyzed (Participants) | 5 | 2 | 4
  Month 6:non-medical practitioner visits | 10.40 (14.05) | 5.50 (6.36) | 4.75 (1.26)
  Month 6:RA-related non-medical visits: number analyzed (Participants) | 5 | 2 | 4
  Month 6:RA-related non-medical visits | 1.20 (1.30) | 1.50 (0.71) | 1.25 (1.26)

65. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Months 12, 18, and 24
Description: as for outcome 64
Time Frame: Months 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 173 | 185 | 79
events
  Month 12: doctor visit | 2.19 (1.81) | 2.19 (1.72) | 2.22 (1.62)
  Month 12: RA-related doctor visit | 0.77 (0.61) | 0.74 (0.70) | 0.89 (0.77)
  Month 12: hospital ER visit: number analyzed (Participants) | 16 | 8 | 5
  Month 12: hospital ER visit | 1.06 (0.25) | 1.13 (0.35) | 1.00 (0.00)
  Month 12: RA-related ER visit: number analyzed (Participants) | 16 | 8 | 5
  Month 12: RA-related ER visit | 0.13 (0.50) | 0.00 (0.00) | 0.20 (0.45)
  Month 12: hospitalization: number analyzed (Participants) | 7 | 3 | 2
  Month 12: hospitalization | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00)
  Month 12: RA-related hospitalization: number analyzed (Participants) | 7 | 4 | 2
  Month 12: RA-related hospitalization | 0.29 (0.49) | 0.00 (0.00) | 0.50 (0.71)
  Month 12: outpatient surgery: number analyzed (Participants) | 9 | 8 | 3
  Month 12: outpatient surgery | 1.00 (0.00) | 1.50 (1.07) | 1.33 (0.58)
  Month 12: RA-related outpatient surgery: number analyzed (Participants) | 9 | 8 | 3
  Month 12: RA-related outpatient surgery | 0.11 (0.33) | 0.13 (0.35) | 0.00 (0.00)
  Month 12:non-study diagnostic tests: number analyzed (Participants) | 31 | 41 | 11
  Month 12:non-study diagnostic tests | 1.61 (1.05) | 1.34 (0.57) | 1.18 (0.40)
  Month 12: RA-related diagnostic tests: number analyzed (Participants) | 31 | 41 | 11
  Month 12: RA-related diagnostic tests | 0.13 (0.50) | 0.22 (0.57) | 0.36 (0.67)
  Month 12:non-medical practitioner visits: number analyzed (Participants) | 2 | 3 | 0
  Month 12:non-medical practitioner visits | 17.00 (18.38) | 13.33 (6.43) |
  Month 12:RA-related non-medical visits: number analyzed (Participants) | 2 | 3 | 0
  Month 12:RA-related non-medical visits | 1.00 (1.41) | 1.33 (1.15) |
  Month 18: doctor visits: number analyzed (Participants) | 160 | 149 | 69
  Month 18: doctor visits | 2.17 (1.91) | 2.21 (1.83) | 2.93 (3.02)
  Month 18: RA-related doctor visit: number analyzed (Participants) | 162 | 149 | 69
  Month 18: RA-related doctor visit | 0.78 (0.74) | 0.82 (0.66) | 0.80 (0.65)
  Month 18: hospital ER visit: number analyzed (Participants) | 10 | 9 | 5
  Month 18: hospital ER visit | 1.60 (1.35) | 1.89 (1.36) | 1.40 (0.89)
  Month 18: RA-related ER visit: number analyzed (Participants) | 10 | 9 | 5
  Month 18: RA-related ER visit | 0.20 (0.63) | 0.00 (0.00) | 0.00 (0.00)
  Month 18: hospitalization: number analyzed (Participants) | 3 | 6 | 3
  Month 18: hospitalization | 2.33 (2.31) | 1.00 (0.00) | 1.00 (0.00)
  Month 18:RA-related hospitalization: number analyzed (Participants) | 3 | 6 | 3
  Month 18:RA-related hospitalization | 0.00 (0.00) | 0.67 (1.03) | 0.67 (1.15)
  Month 18: outpatient surgery: number analyzed (Participants) | 6 | 7 | 3
  Month 18: outpatient surgery | 1.00 (0.00) | 2.14 (1.68) | 3.00 (2.65)
  Month 18:RA-related outpatient surgery: number analyzed (Participants) | 6 | 7 | 3
  Month 18:RA-related outpatient surgery | 0.33 (0.82) | 0.14 (0.38) | 0.00 (0.00)
  Month 18:non-study diagnostic tests: number analyzed (Participants) | 25 | 26 | 12
  Month 18:non-study diagnostic tests | 1.48 (0.77) | 1.85 (1.43) | 1.50 (0.80)
  Month 18:RA-related diagnostic tests: number analyzed (Participants) | 26 | 26 | 12
  Month 18:RA-related diagnostic tests | 0.08 (0.39) | 0.19 (0.49) | 0.08 (0.29)
  Month 18:non-medical practitioner visits: number analyzed (Participants) | 2 | 4 | 1
  Month 18:non-medical practitioner visits | 16.00 (19.80) | 18.00 (16.25) | 4.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 18:RA-related non-medical visits: number analyzed (Participants) | 2 | 4 | 1
  Month 18:RA-related non-medical visits | 2.00 (0.00) | 1.50 (1.91) | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 24: doctor visits: number analyzed (Participants) | 142 | 140 | 57
  Month 24: doctor visits | 2.27 (2.17) | 2.78 (3.80) | 2.75 (2.03)
  Month 24: RA-related doctor visits: number analyzed (Participants) | 142 | 139 | 57
  Month 24: RA-related doctor visits | 0.83 (0.60) | 0.76 (0.71) | 0.93 (0.80)
  Month 24 hospital ER visits: number analyzed (Participants) | 10 | 12 | 3
  Month 24 hospital ER visits | 1.40 (0.70) | 1.33 (0.65) | 1.00 (0.00)
  Month 24: RA-related ER visits: number analyzed (Participants) | 10 | 12 | 3
  Month 24: RA-related ER visits | 0.00 (0.00) | 0.00 (0.00) | 1.33 (1.15)
  Month 24: hospitalization: number analyzed (Participants) | 3 | 4 | 2
  Month 24: hospitalization | 1.00 (0.00) | 1.25 (0.50) | 1.50 (0.71)
  Month 24:RA-related hospitalization: number analyzed (Participants) | 3 | 4 | 2
  Month 24:RA-related hospitalization | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Month 24: outpatient surgery: number analyzed (Participants) | 4 | 5 | 1
  Month 24: outpatient surgery | 3.25 (4.50) | 2.00 (2.24) | 3.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 24:RA-related outpatient surgery: number analyzed (Participants) | 4 | 5 | 1
  Month 24:RA-related outpatient surgery | 0.00 (0.00) | 0.00 (0.00) | 2.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 24:non-study diagnostic tests: number analyzed (Participants) | 20 | 31 | 15
  Month 24:non-study diagnostic tests | 1.50 (0.83) | 1.29 (0.53) | 1.40 (0.51)
  Month 24:RA related diagnostic tests: number analyzed (Participants) | 19 | 31 | 15
  Month 24:RA related diagnostic tests | 0.11 (0.32) | 0.03 (0.18) | 0.27 (0.59)
  Month 24:non-medical practitioner visits: number analyzed (Participants) | 3 | 4 | 0
  Month 24:non-medical practitioner visits | 20.67 (3.06) | 3.50 (1.91) |
  Month 24:RA-related non-medical visits: number analyzed (Participants) | 3 | 4 | 0
  Month 24:RA-related non-medical visits | 0.67 (1.15) | 1.00 (1.15) |

66. Secondary Outcome: Number of Days as Assessed Using RA-HCRU at Baseline and Months 3 and 6
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA or non-RA related number of days spent in hospital, nursing home, aids/devices used, on sick leave, work per week, performed part time work, performed paid work, chores done by housekeeper and chores done by family/friends.
Time Frame: Baseline and Months 3 and 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 190 | 196 | 94
days
  BL: hospital length of stay: number analyzed (Participants) | 41 | 29 | 22
  BL: hospital length of stay | 19.07 (10.86) | 23.76 (18.95) | 15.45 (11.61)
  BL: days in nursing home: number analyzed (Participants) | 0 | 5 | 3
  BL: days in nursing home |  | 30.60 (33.62) | 41.67 (42.00)
  BL: days aids/devices used: number analyzed (Participants) | 36 | 36 | 17
  BL: days aids/devices used | 99.94 (107.83) | 93.06 (130.53) | 162.88 (140.39)
  BL: RA-related aids used: number analyzed (Participants) | 36 | 36 | 17
  BL: RA-related aids used | 1.61 (1.15) | 1.75 (1.36) | 2.24 (1.95)
  BL: days of work per week: number analyzed (Participants) | 167 | 183 | 85
  BL: days of work per week | 5.11 (0.98) | 4.96 (0.97) | 5.12 (0.91)
  BL: days on sick leave due to RA: number analyzed (Participants) | 85 | 93 | 43
  BL: days on sick leave due to RA | 23.52 (25.55) | 16.59 (22.38) | 27.67 (30.63)
  BL: days of part-time work: number analyzed (Participants) | 33 | 42 | 28
  BL: days of part-time work | 11.94 (20.56) | 12.12 (18.10) | 11.39 (14.06)
  BL: paid work, bothered by RA: number analyzed (Participants) | 131 | 150 | 69
  BL: paid work, bothered by RA | 35.69 (30.24) | 38.54 (47.28) | 31.68 (30.31)
  BL: chores by housekeeper: number analyzed (Participants) | 34 | 48 | 12
  BL: chores by housekeeper | 19.56 (27.62) | 25.46 (33.29) | 21.25 (32.37)
  BL: chores by family | 32.35 (34.46) | 34.13 (34.19) | 34.35 (33.04)
  Month 3: hospital length of stay: number analyzed (Participants) | 4 | 3 | 2
  Month 3: hospital length of stay | 14.25 (17.19) | 7.00 (7.21) | 20.00 (1.41)
  Month 3: days in nursing home: number analyzed (Participants) | 1 | 3 | 0
  Month 3: days in nursing home | 28.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 43.33 (40.43) |
  Month 3: days aids/devices used: number analyzed (Participants) | 20 | 20 | 14
  Month 3: days aids/devices used | 109.00 (116.27) | 123.85 (76.69) | 105.86 (77.06)
  Month 3: RA-related aids used: number analyzed (Participants) | 20 | 20 | 14
  Month 3: RA-related aids used | 1.45 (1.23) | 1.75 (0.55) | 1.71 (0.91)
  Month 3: days of work per week: number analyzed (Participants) | 171 | 180 | 79
  Month 3: days of work per week | 5.16 (1.06) | 4.99 (1.02) | 5.08 (0.80)
  Month 3:days on sick leave due to RA: number analyzed (Participants) | 38 | 33 | 23
  Month 3:days on sick leave due to RA | 20.76 (30.15) | 26.97 (34.53) | 36.61 (37.92)
  Month 3: days of part time work: number analyzed (Participants) | 20 | 15 | 12
  Month 3: days of part time work | 14.85 (25.99) | 29.67 (38.10) | 16.17 (25.29)
  Month 3: paid work, bothered by RA: number analyzed (Participants) | 93 | 92 | 47
  Month 3: paid work, bothered by RA | 21.04 (26.24) | 19.48 (25.23) | 22.13 (28.03)
  Month 3: chores by housekeeper: number analyzed (Participants) | 17 | 30 | 18
  Month 3: chores by housekeeper | 22.53 (30.49) | 21.43 (28.45) | 17.33 (28.24)
  Month 3: chores by family: number analyzed (Participants) | 104 | 109 | 70
  Month 3: chores by family | 23.13 (29.61) | 21.06 (27.81) | 24.80 (28.39)
  Month 6: hospital length of stay: number analyzed (Participants) | 3 | 6 | 4
  Month 6: hospital length of stay | 9.33 (5.03) | 9.00 (13.62) | 10.75 (9.00)
  Month 6: days in nursing home: number analyzed (Participants) | 1 | 1 | 1
  Month 6: days in nursing home | 14.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 90.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 61.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 6: days aids/devices used: number analyzed (Participants) | 20 | 12 | 8
  Month 6: days aids/devices used | 74.15 (65.25) | 159.08 (138.46) | 190.25 (93.12)
  Month 6: RA-related aids used: number analyzed (Participants) | 20 | 14 | 8
  Month 6: RA-related aids used | 1.25 (0.55) | 2.00 (1.36) | 2.38 (0.74)
  Month 6: days of work per week: number analyzed (Participants) | 168 | 170 | 71
  Month 6: days of work per week | 5.11 (0.95) | 4.93 (1.05) | 5.10 (0.99)
  Month 6:days on sick leave due to RA: number analyzed (Participants) | 17 | 17 | 14
  Month 6:days on sick leave due to RA | 18.00 (19.68) | 21.94 (33.32) | 40.07 (41.32)
  Month 6: days of part time work: number analyzed (Participants) | 8 | 9 | 7
  Month 6: days of part time work | 14.13 (14.71) | 7.11 (5.49) | 11.71 (21.31)
  Month 6: paid work, bothered by RA: number analyzed (Participants) | 66 | 56 | 39
  Month 6: paid work, bothered by RA | 26.23 (30.00) | 16.41 (23.15) | 24.49 (28.36)
  Month 6: chores by housekeeper: number analyzed (Participants) | 14 | 23 | 10
  Month 6: chores by housekeeper | 21.57 (29.10) | 20.57 (28.22) | 13.80 (27.20)
  Month 6: chores by family: number analyzed (Participants) | 73 | 60 | 46
  Month 6: chores by family | 23.62 (29.77) | 20.05 (26.35) | 22.09 (28.50)

67. Secondary Outcome: Number of Days as Assessed Using RA-HCRU at Months 12, 18, and 24
Description: as for outcome 66
Time Frame: Months 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 154 | 153 | 64
days
  Month 12: hospital length of stay: number analyzed (Participants) | 7 | 4 | 2
  Month 12: hospital length of stay | 10.43 (8.62) | 9.25 (3.59) | 9.00 (8.49)
  Month 12: days in nursing home: number analyzed (Participants) | 0 | 2 | 1
  Month 12: days in nursing home |  | 54.00 (50.91) | 20.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 12: days aids/devices used: number analyzed (Participants) | 20 | 8 | 4
  Month 12: days aids/devices used | 118.05 (99.31) | 231.00 (190.27) | 65.75 (16.50)
  Month 12: RA-related aids used: number analyzed (Participants) | 20 | 9 | 4
  Month 12: RA-related aids used | 1.50 (0.83) | 1.89 (1.96) | 1.50 (0.58)
  Month 12: days of work per week | 5.14 (0.98) | 4.95 (1.01) | 5.05 (0.93)
  Month 12:days on sick leave due to RA: number analyzed (Participants) | 17 | 7 | 8
  Month 12:days on sick leave due to RA | 17.47 (28.41) | 10.14 (9.94) | 2.75 (1.49)
  Month 12: days of part-time work: number analyzed (Participants) | 9 | 6 | 2
  Month 12: days of part-time work | 5.56 (6.82) | 12.17 (10.11) | 16.00 (15.56)
  Month 12:paid work, bothered by RA: number analyzed (Participants) | 52 | 43 | 30
  Month 12:paid work, bothered by RA | 19.31 (21.34) | 16.23 (22.36) | 21.10 (26.11)
  Month 12: chores by housekeeper: number analyzed (Participants) | 11 | 14 | 5
  Month 12: chores by housekeeper | 13.09 (25.89) | 24.36 (35.96) | 7.40 (3.58)
  Month 12: chores by family: number analyzed (Participants) | 54 | 45 | 27
  Month 12: chores by family | 22.04 (30.72) | 20.11 (27.19) | 17.74 (25.33)
  Month 18: hospital length of stay: number analyzed (Participants) | 3 | 6 | 3
  Month 18: hospital length of stay | 6.67 (3.06) | 13.67 (9.42) | 33.33 (11.55)
  Month 18: days in nursing home: number analyzed (Participants) | 1 | 0 | 0
  Month 18: days in nursing home | 15.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |  |
  Month 18: days aids/devices used: number analyzed (Participants) | 12 | 8 | 4
  Month 18: days aids/devices used | 126.67 (125.26) | 169.50 (157.29) | 159.50 (41.00)
  Month 18: RA-related aids used: number analyzed (Participants) | 12 | 8 | 4
  Month 18: RA-related aids used | 2.25 (1.06) | 2.25 (1.67) | 2.50 (1.00)
  Month 18: days of work per week: number analyzed (Participants) | 142 | 142 | 52
  Month 18: days of work per week | 5.13 (1.00) | 5.01 (0.99) | 5.00 (0.69)
  Month 18:days on sick leave due to RA: number analyzed (Participants) | 14 | 11 | 5
  Month 18:days on sick leave due to RA | 16.93 (23.97) | 6.09 (5.87) | 4.20 (1.64)
  Month 18: days of part time work: number analyzed (Participants) | 6 | 5 | 2
  Month 18: days of part time work | 4.33 (3.01) | 6.80 (4.66) | 31.00 (41.01)
  Month 18:paid work, bothered by RA: number analyzed (Participants) | 55 | 43 | 20
  Month 18:paid work, bothered by RA | 16.82 (22.67) | 16.30 (22.60) | 19.35 (25.33)
  Month 18: chores by housekeeper: number analyzed (Participants) | 5 | 12 | 6
  Month 18: chores by housekeeper | 9.40 (6.99) | 21.75 (33.15) | 3.83 (2.48)
  Month 18: chores by family: number analyzed (Participants) | 39 | 33 | 19
  Month 18: chores by family | 20.49 (29.77) | 21.30 (30.38) | 27.37 (35.36)
  Month 24: hospital length of stay: number analyzed (Participants) | 3 | 4 | 2
  Month 24: hospital length of stay | 5.33 (5.77) | 21.00 (10.65) | 6.00 (2.83)
  Month 24: days in nursing home: number analyzed (Participants) | 1 | 1 | 2
  Month 24: days in nursing home | 2.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 21.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 15.50 (7.78)
  Month 24: days aids/devices used: number analyzed (Participants) | 13 | 10 | 4
  Month 24: days aids/devices used | 137.85 (150.03) | 178.20 (178.98) | 136.50 (87.00)
  Month 24: RA-related aids used: number analyzed (Participants) | 13 | 11 | 4
  Month 24: RA-related aids used | 2.15 (1.52) | 1.82 (2.09) | 1.50 (1.00)
  Month 24: days of work per week: number analyzed (Participants) | 134 | 128 | 48
  Month 24: days of work per week | 5.10 (1.02) | 5.03 (1.01) | 5.15 (0.80)
  Month 24:days on sick leave due to RA: number analyzed (Participants) | 9 | 4 | 8
  Month 24:days on sick leave due to RA | 19.33 (27.95) | 3.25 (2.50) | 7.25 (12.46)
  Month 24: days of part time work: number analyzed (Participants) | 5 | 2 | 4
  Month 24: days of part time work | 6.60 (4.10) | 3.00 (2.83) | 19.00 (30.69)
  Month 24: paid work, bothered by RA: number analyzed (Participants) | 40 | 42 | 22
  Month 24: paid work, bothered by RA | 21.95 (27.30) | 9.17 (9.50) | 16.95 (17.31)
  Month 24: chores by housekeeper: number analyzed (Participants) | 10 | 12 | 3
  Month 24: chores by housekeeper | 6.90 (8.28) | 4.75 (2.99) | 4.00 (2.00)
  Month 24: chores by family: number analyzed (Participants) | 34 | 33 | 19
  Month 24: chores by family | 16.65 (23.82) | 12.18 (21.46) | 17.21 (26.87)

68. Secondary Outcome: Number of Hours Per Day as Assessed Using RA-HCRU at Baseline and Months 3 and 6
Description: RA-HCRU assessed healthcare (HC) usage during previous 3 months for direct or indirect medical cost domains. Any RA or non-RA related number of hours spent per day for home healthcare services, chores done by housekeeper, chores done by family or friends, work done, and work missed were reported.
Time Frame: Baseline and Months 3 and 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 191 | 195 | 92
hours per day
  BL: home healthcare services: number analyzed (Participants) | 4 | 5 | 3
  BL: home healthcare services | 1.50 (0.58) | 2.20 (1.64) | 1.00 (1.00)
  BL: RA-related home HC services: number analyzed (Participants) | 4 | 6 | 3
  BL: RA-related home HC services | 1.00 (0.82) | 0.83 (0.75) | 1.33 (0.58)
  BL: work done: number analyzed (Participants) | 167 | 184 | 85
  BL: work done | 8.53 (5.33) | 8.25 (4.02) | 7.68 (1.81)
  BL: missed work due to RA: number analyzed (Participants) | 33 | 42 | 28
  BL: missed work due to RA | 4.36 (4.98) | 5.62 (13.58) | 6.21 (8.96)
  BL: chores by housekeeper: number analyzed (Participants) | 34 | 48 | 12
  BL: chores by housekeeper | 4.85 (2.31) | 6.46 (9.83) | 4.75 (2.45)
  BL: chores by family | 4.26 (4.56) | 3.92 (4.23) | 4.08 (4.01)
  Month 3: home healthcare services: number analyzed (Participants) | 1 | 4 | 0
  Month 3: home healthcare services | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 1.25 (0.50) |
  Month 3:RA-related home HC services: number analyzed (Participants) | 1 | 4 | 0
  Month 3:RA-related home HC services | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 0.25 (0.50) |
  Month 3: work done: number analyzed (Participants) | 171 | 180 | 79
  Month 3: work done | 8.53 (4.70) | 8.55 (5.23) | 8.33 (3.71)
  Month 3: missed work due to RA: number analyzed (Participants) | 19 | 14 | 12
  Month 3: missed work due to RA | 4.11 (2.51) | 8.86 (15.72) | 5.58 (7.95)
  Month 3: chores by housekeeper: number analyzed (Participants) | 18 | 30 | 17
  Month 3: chores by housekeeper | 4.50 (2.43) | 5.40 (4.61) | 4.00 (2.55)
  Month 3: chores by family: number analyzed (Participants) | 104 | 109 | 70
  Month 3: chores by family | 3.44 (3.77) | 3.35 (3.50) | 3.61 (4.19)
  Month 6: home healthcare services: number analyzed (Participants) | 3 | 2 | 0
  Month 6: home healthcare services | 5.00 (6.08) | 4.50 (0.71) |
  Month 6: RA-related home HC services: number analyzed (Participants) | 3 | 2 | 0
  Month 6: RA-related home HC services | 0.67 (0.58) | 2.00 (2.83) |
  Month 6: work done: number analyzed (Participants) | 168 | 171 | 71
  Month 6: work done | 7.97 (2.84) | 8.29 (4.40) | 7.85 (1.47)
  Month 6: missed work due to RA: number analyzed (Participants) | 7 | 9 | 6
  Month 6: missed work due to RA | 4.14 (2.67) | 4.11 (3.44) | 6.33 (5.75)
  Month 6: chores by housekeeper: number analyzed (Participants) | 14 | 23 | 10
  Month 6: chores by housekeeper | 4.93 (2.70) | 5.17 (2.92) | 4.80 (2.20)
  Month 6: chores by family: number analyzed (Participants) | 72 | 60 | 46
  Month 6: chores by family | 3.86 (2.84) | 3.28 (2.29) | 4.22 (6.14)

69. Secondary Outcome: Number of Hours Per Day as Assessed Using RA-HCRU at Months 12, 18, and 24
Description: RA-HCRU assessed HC usage during previous 3 months for direct or indirect medical cost domains. Any RA or non-RA related number of hours spent per day for home healthcare services, chores done by housekeeper, chores done by family or friends, work done, and work missed were reported.
Time Frame: Months 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 154 | 153 | 64
hours per day
  Month 12: home healthcare services: number analyzed (Participants) | 2 | 2 | 0
  Month 12: home healthcare services | 2.00 (0.00) | 25.00 (32.53) |
  Month 12:RA-related home HC services: number analyzed (Participants) | 2 | 2 | 0
  Month 12:RA-related home HC services | 0.00 (0.00) | 0.00 (0.00) |
  Month 12: work done | 8.38 (3.90) | 7.99 (3.59) | 8.34 (4.32)
  Month 12: missed work due to RA: number analyzed (Participants) | 8 | 6 | 2
  Month 12: missed work due to RA | 2.25 (1.28) | 4.83 (5.34) | 3.50 (0.71)
  Month 12: chores by housekeeper: number analyzed (Participants) | 11 | 15 | 5
  Month 12: chores by housekeeper | 6.64 (4.67) | 4.60 (2.29) | 3.80 (1.92)
  Month 12: chores by family: number analyzed (Participants) | 54 | 45 | 27
  Month 12: chores by family | 3.44 (3.66) | 3.29 (2.40) | 3.19 (2.25)
  Month 18: home healthcare services: number analyzed (Participants) | 1 | 0 | 0
  Month 18: home healthcare services | 2.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |  |
  Month 18:RA-related home HC services: number analyzed (Participants) | 1 | 0 | 0
  Month 18:RA-related home HC services | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |  |
  Month 18: work done: number analyzed (Participants) | 142 | 142 | 52
  Month 18: work done | 8.18 (3.73) | 8.32 (4.16) | 8.02 (1.45)
  Month 18: missed work due to RA: number analyzed (Participants) | 6 | 5 | 2
  Month 18: missed work due to RA | 3.00 (2.53) | 1.80 (1.64) | 2.50 (0.71)
  Month 18: chores by housekeeper: number analyzed (Participants) | 5 | 12 | 6
  Month 18: chores by housekeeper | 5.60 (1.34) | 4.92 (2.94) | 4.33 (3.01)
  Month 18: chores by family: number analyzed (Participants) | 39 | 33 | 18
  Month 18: chores by family | 3.74 (4.42) | 3.70 (3.28) | 3.44 (2.57)
  Month 24:home healthcare services: number analyzed (Participants) | 0 | 3 | 1
  Month 24:home healthcare services |  | 2.67 (1.15) | 2.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 24: RA-related home HC services: number analyzed (Participants) | 0 | 3 | 1
  Month 24: RA-related home HC services |  | 0.00 (0.00) | 2.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 24: work done: number analyzed (Participants) | 134 | 128 | 48
  Month 24: work done | 8.63 (4.69) | 7.84 (2.36) | 8.02 (1.48)
  Month 24: missed work due to RA: number analyzed (Participants) | 4 | 2 | 4
  Month 24: missed work due to RA | 6.50 (6.61) | 2.00 (0.00) | 4.50 (7.72)
  Month 24: chores by housekeeper: number analyzed (Participants) | 10 | 12 | 3
  Month 24: chores by housekeeper | 8.50 (8.63) | 5.25 (2.93) | 4.33 (0.58)
  Month 24: chores by family: number analyzed (Participants) | 34 | 32 | 20
  Month 24: chores by family | 2.97 (2.14) | 2.81 (2.22) | 3.75 (3.19)

70. Secondary Outcome: Work Performance in Past 3 Months on Days Bothered as Assessed Using RA-HCRU
Description: Work performance of participants on number of days bothered was based on a 0 to 10-point scale, where higher score indicated lower work performance.
Time Frame: Baseline, Months 3, 6, 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 276 | 292 | 138
units on a scale
  Baseline | 4.94 (3.26) | 4.71 (3.07) | 4.57 (3.15)
  Month 3: number analyzed (Participants) | 256 | 277 | 118
  Month 3 | 3.59 (2.92) | 3.25 (3.78) | 3.57 (2.80)
  Month 6: number analyzed (Participants) | 250 | 266 | 109
  Month 6 | 2.97 (3.58) | 2.27 (2.58) | 3.04 (2.75)
  Month 12: number analyzed (Participants) | 236 | 235 | 95
  Month 12 | 2.69 (2.75) | 2.08 (2.38) | 2.94 (3.85)
  Month 18: number analyzed (Participants) | 233 | 223 | 82
  Month 18 | 2.33 (2.63) | 2.11 (2.47) | 2.11 (2.38)
  Month 24: number analyzed (Participants) | 200 | 206 | 73
  Month 24 | 2.47 (2.63) | 2.35 (2.75) | 2.52 (2.68)

71. Secondary Outcome: Change From Baseline in Work Productivity and HCRU at Months 3 and 6
Description: RA-HCRU assessed HC usage during last 3 months for direct, indirect medical cost domains. Direct cost: visit to doctor, non-medical practitioner, nursing home, hospital, surgery, ER treatment, diagnostic tests, overnight stay, home healthcare services, aids/devices used. Indirect costs associated with functional disability: employment status, willingness to work, work disability due to RA, sick leave, part time work, ability to perform chores, chores done by family/friends/housekeeper. Assessment was based on 0 to 2-point scale; higher score=higher medical cost.
Time Frame: Months 3 and 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 351 | 381 | 171
units on a scale
  Month 3: seen any doctor: number analyzed (Participants) | 349 | 380 | 171
  Month 3: seen any doctor | 0.24 (0.49) | 0.18 (0.48) | 0.18 (0.46)
  Month 3: treated in ER: number analyzed (Participants) | 350 | 381 | 171
  Month 3: treated in ER | 0.01 (0.25) | 0.04 (0.32) | 0.06 (0.31)
  Month 3:admitted for overnight stay: number analyzed (Participants) | 3 | 5 | 0
  Month 3:admitted for overnight stay | 0.00 (0.00) | -0.60 (0.89) |
  Month 3:hospitalization | 0.10 (0.33) | 0.07 (0.26) | 0.12 (0.36)
  Month 3: outpatient surgery | 0.01 (0.19) | 0.02 (0.24) | 0.01 (0.17)
  Month 3: non-study diagnostic test | 0.16 (0.51) | 0.17 (0.47) | 0.23 (0.50)
  Month 3: in nursing home | -0.00 (0.05) | 0.00 (0.11) | 0.02 (0.13)
  Month 3: home healthcare services: number analyzed (Participants) | 350 | 381 | 171
  Month 3: home healthcare services | 0.01 (0.12) | 0.00 (0.11) | 0.02 (0.13)
  Month 3: required aids/devices: number analyzed (Participants) | 351 | 380 | 171
  Month 3: required aids/devices | 0.05 (0.29) | 0.04 (0.27) | -0.01 (0.25)
  Month 3: non-medical practitioner | 0.01 (0.18) | 0.03 (0.20) | 0.03 (0.20)
  Month 3: currently employed | -0.03 (0.26) | -0.00 (0.27) | 0.00 (0.27)
  Month 3: feel well enough to work: number analyzed (Participants) | 160 | 163 | 81
  Month 3: feel well enough to work | -0.16 (0.46) | -0.17 (0.45) | -0.11 (0.45)
  Month 3: unable to work due to RA: number analyzed (Participants) | 162 | 165 | 81
  Month 3: unable to work due to RA | 0.12 (0.44) | 0.13 (0.52) | 0.05 (0.55)
  Month 3: lost job/retired early: number analyzed (Participants) | 159 | 162 | 79
  Month 3: lost job/retired early | -0.07 (0.47) | -0.02 (0.38) | 0.05 (0.45)
  Month 3: work disabled due to RA: number analyzed (Participants) | 159 | 162 | 81
  Month 3: work disabled due to RA | 0.10 (0.42) | 0.11 (0.49) | 0.06 (0.43)
  Month 3: retired: number analyzed (Participants) | 160 | 168 | 83
  Month 3: retired | -0.01 (0.24) | -0.02 (0.28) | 0.01 (0.33)
  Month 3: sick leave due to RA: number analyzed (Participants) | 290 | 312 | 144
  Month 3: sick leave due to RA | 0.14 (0.42) | 0.18 (0.45) | 0.13 (0.44)
  Month 3: performed part-time work: number analyzed (Participants) | 292 | 308 | 140
  Month 3: performed part-time work | 0.04 (0.31) | 0.08 (0.36) | 0.09 (0.41)
  Month 3: performed paid work: number analyzed (Participants) | 294 | 315 | 138
  Month 3: performed paid work | 0.09 (0.48) | 0.16 (0.51) | 0.12 (0.46)
  Month 3: unable to do chores: number analyzed (Participants) | 348 | 379 | 171
  Month 3: unable to do chores | 0.28 (0.57) | 0.32 (0.54) | 0.09 (0.53)
  Month 3: chores by housekeeper: number analyzed (Participants) | 349 | 379 | 170
  Month 3: chores by housekeeper | 0.04 (0.29) | 0.05 (0.29) | -0.04 (0.29)
  Month 3: chores by family/friends: number analyzed (Participants) | 351 | 379 | 170
  Month 3: chores by family/friends | 0.21 (0.53) | 0.21 (0.49) | 0.09 (0.53)
  Month 6: seen any doctor: number analyzed (Participants) | 338 | 362 | 158
  Month 6: seen any doctor | 0.28 (0.53) | 0.26 (0.50) | 0.22 (0.47)
  Month 6: treated in ER: number analyzed (Participants) | 337 | 364 | 158
  Month 6: treated in ER | 0.00 (0.29) | 0.03 (0.33) | 0.05 (0.29)
  Month 6:admitted for overnight stay: number analyzed (Participants) | 0 | 5 | 0
  Month 6:admitted for overnight stay |  | -0.20 (0.45) |
  Month 6: Hospitalization: number analyzed (Participants) | 338 | 364 | 158
  Month 6: Hospitalization | 0.10 (0.33) | 0.06 (0.29) | 0.09 (0.35)
  Month 6: outpatient surgery: number analyzed (Participants) | 338 | 364 | 158
  Month 6: outpatient surgery | 0.01 (0.21) | 0.02 (0.24) | -0.01 (0.21)
  Month 6: non-study diagnostic test: number analyzed (Participants) | 337 | 364 | 158
  Month 6: non-study diagnostic test | 0.17 (0.54) | 0.15 (0.52) | 0.18 (0.54)
  Month 6: in nursing home: number analyzed (Participants) | 338 | 364 | 158
  Month 6: in nursing home | -0.00 (0.05) | 0.01 (0.09) | 0.01 (0.14)
  Month 6: home healthcare services: number analyzed (Participants) | 338 | 364 | 158
  Month 6: home healthcare services | 0.00 (0.14) | 0.01 (0.14) | 0.01 (0.11)
  Month 6: required aids/devices: number analyzed (Participants) | 338 | 364 | 158
  Month 6: required aids/devices | 0.04 (0.28) | 0.05 (0.29) | 0.04 (0.27)
  Month 6: non-medical practitioner: number analyzed (Participants) | 338 | 364 | 158
  Month 6: non-medical practitioner | 0.01 (0.18) | 0.04 (0.20) | 0.00 (0.20)
  Month 6: currently employed: number analyzed (Participants) | 337 | 365 | 158
  Month 6: currently employed | -0.04 (0.28) | -0.01 (0.27) | 0.00 (0.28)
  Month 6: feel well enough to work: number analyzed (Participants) | 152 | 158 | 73
  Month 6: feel well enough to work | -0.24 (0.55) | -0.19 (0.45) | -0.10 (0.53)
  Month 6: unable to work due to RA: number analyzed (Participants) | 153 | 158 | 74
  Month 6: unable to work due to RA | 0.18 (0.54) | 0.15 (0.50) | 0.05 (0.55)
  Month 6: lost job/retired early: number analyzed (Participants) | 152 | 156 | 71
  Month 6: lost job/retired early | 0.00 (0.47) | 0.01 (0.35) | 0.04 (0.46)
  Month 6: work disabled due to RA: number analyzed (Participants) | 151 | 156 | 73
  Month 6: work disabled due to RA | 0.14 (0.49) | 0.13 (0.44) | 0.07 (0.42)
  Month 6: retired: number analyzed (Participants) | 153 | 168 | 76
  Month 6: retired | -0.01 (0.30) | -0.03 (0.30) | 0.03 (0.36)
  Month 6: sick leave due to RA: number analyzed (Participants) | 276 | 286 | 129
  Month 6: sick leave due to RA | 0.21 (0.46) | 0.23 (0.43) | 0.17 (0.44)
  Month 6: performed part-time work: number analyzed (Participants) | 279 | 281 | 126
  Month 6: performed part-time work | 0.09 (0.34) | 0.09 (0.33) | 0.12 (0.45)
  Month 6: performed paid work: number analyzed (Participants) | 279 | 288 | 125
  Month 6: performed paid work | 0.18 (0.51) | 0.26 (0.52) | 0.14 (0.48)
  Month 6: unable to do chores: number analyzed (Participants) | 333 | 358 | 158
  Month 6: unable to do chores | 0.37 (0.54) | 0.41 (0.54) | 0.24 (0.56)
  Month 6: chores by housekeeper: number analyzed (Participants) | 335 | 360 | 157
  Month 6: chores by housekeeper | 0.04 (0.25) | 0.08 (0.32) | 0.01 (0.24)
  Month 6: chores by family/friends: number analyzed (Participants) | 337 | 361 | 157
  Month 6: chores by family/friends | 0.30 (0.52) | 0.34 (0.50) | 0.22 (0.56)

72. Secondary Outcome: Change From Baseline in Work Productivity and HCRU at Months 12, 18, and 24
Description: as for outcome 71
Time Frame: Months 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 314 | 327 | 135
units on a scale
  Month 12: seen any doctor: number analyzed (Participants) | 314 | 326 | 135
  Month 12: seen any doctor | 0.34 (0.51) | 0.31 (0.52) | 0.26 (0.46)
  Month 12: treated in ER | 0.00 (0.27) | 0.05 (0.29) | 0.04 (0.31)
  Month12:admitted for overnight stay: number analyzed (Participants) | 4 | 2 | 1
  Month12:admitted for overnight stay | 0.00 (0.00) | 0.50 (0.71) | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 12: hospitalized | 0.08 (0.33) | 0.06 (0.29) | 0.09 (0.33)
  Month 12:any outpatient surgery | -0.00 (0.23) | 0.01 (0.23) | -0.01 (0.19)
  Month 12:non-study diagnostic tests | 0.15 (0.51) | 0.13 (0.51) | 0.21 (0.51)
  Month 12: in a nursing home | 0.00 (0.00) | 0.01 (0.08) | 0.01 (0.15)
  Month 12: home healthcare services: number analyzed (Participants) | 314 | 326 | 135
  Month 12: home healthcare services | 0.01 (0.14) | 0.01 (0.14) | 0.01 (0.12)
  Month 12: used aids/devices | 0.04 (0.28) | 0.06 (0.29) | 0.06 (0.29)
  Month 12: non-medical practitioner | 0.03 (0.18) | 0.03 (0.18) | 0.02 (0.15)
  Month 12: currently employed | -0.03 (0.34) | -0.01 (0.34) | -0.02 (0.26)
  Month 12: feel well enough to work: number analyzed (Participants) | 133 | 140 | 63
  Month 12: feel well enough to work | -0.17 (0.52) | -0.18 (0.47) | -0.19 (0.50)
  Month 12: unable to work due to RA: number analyzed (Participants) | 135 | 141 | 65
  Month 12: unable to work due to RA | 0.18 (0.52) | 0.23 (0.53) | 0.18 (0.58)
  Month 12: Lost job/retired early: number analyzed (Participants) | 134 | 138 | 64
  Month 12: Lost job/retired early | 0.02 (0.43) | -0.01 (0.44) | 0.02 (0.49)
  Month 12: work disabled due to RA: number analyzed (Participants) | 134 | 138 | 64
  Month 12: work disabled due to RA | 0.10 (0.55) | 0.13 (0.48) | 0.11 (0.48)
  Month 12: retired: number analyzed (Participants) | 137 | 144 | 67
  Month 12: retired | -0.02 (0.35) | -0.07 (0.35) | -0.03 (0.43)
  Month 12: sick leave due to RA: number analyzed (Participants) | 257 | 259 | 104
  Month 12: sick leave due to RA | 0.21 (0.45) | 0.27 (0.46) | 0.20 (0.45)
  Month 12: performed part time work: number analyzed (Participants) | 258 | 254 | 103
  Month 12: performed part time work | 0.09 (0.32) | 0.09 (0.33) | 0.17 (0.42)
  Month 12: performed paid work: number analyzed (Participants) | 255 | 257 | 103
  Month 12: performed paid work | 0.22 (0.50) | 0.28 (0.54) | 0.18 (0.52)
  Month 12: unable to do chores: number analyzed (Participants) | 309 | 324 | 135
  Month 12: unable to do chores | 0.36 (0.56) | 0.44 (0.56) | 0.30 (0.55)
  Month 12: chores by housekeeper: number analyzed (Participants) | 312 | 325 | 134
  Month 12: chores by housekeeper | 0.04 (0.26) | 0.09 (0.30) | 0.01 (0.21)
  Month 12: chores by family/friends: number analyzed (Participants) | 314 | 326 | 134
  Month 12: chores by family/friends | 0.35 (0.53) | 0.36 (0.51) | 0.28 (0.54)
  Month 18: seen any doctor: number analyzed (Participants) | 283 | 292 | 116
  Month 18: seen any doctor | 0.32 (0.54) | 0.36 (0.55) | 0.28 (0.54)
  Month 18: treated in ER: number analyzed (Participants) | 283 | 292 | 116
  Month 18: treated in ER | 0.01 (0.27) | 0.04 (0.31) | 0.03 (0.28)
  Month18:admitted for overnight stay: number analyzed (Participants) | 1 | 1 | 2
  Month18:admitted for overnight stay | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 2.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 0.00 (0.00)
  Month 18:hospitalization: number analyzed (Participants) | 283 | 292 | 116
  Month 18:hospitalization | 0.10 (0.33) | 0.05 (0.30) | 0.08 (0.33)
  Month 18: outpatient surgery: number analyzed (Participants) | 283 | 292 | 116
  Month 18: outpatient surgery | 0.01 (0.21) | 0.01 (0.24) | -0.01 (0.21)
  Month 18:non-study diagnostic tests: number analyzed (Participants) | 283 | 292 | 116
  Month 18:non-study diagnostic tests | 0.16 (0.49) | 0.17 (0.54) | 0.19 (0.57)
  Month 18: in nursing home: number analyzed (Participants) | 283 | 292 | 116
  Month 18: in nursing home | -0.00 (0.06) | 0.01 (0.12) | 0.02 (0.13)
  Month 18: home healthcare services: number analyzed (Participants) | 281 | 292 | 116
  Month 18: home healthcare services | 0.01 (0.13) | 0.01 (0.10) | 0.02 (0.13)
  Month 18: required aids/devices: number analyzed (Participants) | 283 | 292 | 116
  Month 18: required aids/devices | 0.06 (0.25) | 0.06 (0.29) | 0.07 (0.29)
  Month 18: non-medical practitioner: number analyzed (Participants) | 283 | 292 | 116
  Month 18: non-medical practitioner | 0.02 (0.18) | 0.03 (0.18) | 0.02 (0.19)
  Month 18: currently employed: number analyzed (Participants) | 283 | 292 | 116
  Month 18: currently employed | -0.03 (0.36) | -0.03 (0.39) | 0.01 (0.28)
  Month 18: feel well enough to work: number analyzed (Participants) | 114 | 113 | 53
  Month 18: feel well enough to work | -0.27 (0.54) | -0.17 (0.44) | -0.08 (0.55)
  Month 18: unable to work due to RA: number analyzed (Participants) | 116 | 115 | 55
  Month 18: unable to work due to RA | 0.28 (0.57) | 0.21 (0.58) | 0.15 (0.56)
  Month 18: lost job/retired early: number analyzed (Participants) | 113 | 111 | 54
  Month 18: lost job/retired early | 0.05 (0.46) | 0.03 (0.48) | 0.00 (0.51)
  Month 18: work disabled due to RA: number analyzed (Participants) | 112 | 113 | 55
  Month 18: work disabled due to RA | 0.21 (0.56) | 0.17 (0.48) | 0.02 (0.49)
  Month 18: retired: number analyzed (Participants) | 116 | 118 | 55
  Month 18: retired | -0.04 (0.38) | -0.05 (0.39) | 0.02 (0.49)
  Month 18: sick leave due to RA: number analyzed (Participants) | 235 | 229 | 87
  Month 18: sick leave due to RA | 0.20 (0.49) | 0.26 (0.46) | 0.22 (0.47)
  Month 18: performed part-time work: number analyzed (Participants) | 237 | 224 | 88
  Month 18: performed part-time work | 0.09 (0.31) | 0.11 (0.36) | 0.19 (0.43)
  Month 18: performed paid work: number analyzed (Participants) | 236 | 231 | 88
  Month 18: performed paid work | 0.18 (0.55) | 0.27 (0.52) | 0.27 (0.54)
  Month 18: unable to do chores: number analyzed (Participants) | 280 | 290 | 116
  Month 18: unable to do chores | 0.41 (0.53) | 0.47 (0.56) | 0.29 (0.58)
  Month 18: chores by housekeeper: number analyzed (Participants) | 281 | 290 | 115
  Month 18: chores by housekeeper | 0.06 (0.27) | 0.10 (0.33) | 0.00 (0.26)
  Month 18: chores by family/friends: number analyzed (Participants) | 283 | 291 | 115
  Month 18: chores by family/friends | 0.37 (0.53) | 0.41 (0.51) | 0.34 (0.54)
  Month 24: seen any doctor: number analyzed (Participants) | 262 | 278 | 105
  Month 24: seen any doctor | 0.34 (0.53) | 0.36 (0.55) | 0.34 (0.50)
  Month 24: treated in ER: number analyzed (Participants) | 263 | 278 | 106
  Month 24: treated in ER | 0.01 (0.25) | 0.03 (0.33) | 0.03 (0.29)
  Month24:admitted for overnight stay: number analyzed (Participants) | 3 | 1 | 0
  Month24:admitted for overnight stay | 0.00 (0.00) | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |
  Month 24: Hospitalization: number analyzed (Participants) | 263 | 278 | 106
  Month 24: Hospitalization | 0.09 (0.32) | 0.06 (0.29) | 0.07 (0.32)
  Month 24: outpatient surgery: number analyzed (Participants) | 263 | 278 | 106
  Month 24: outpatient surgery | 0.01 (0.17) | 0.02 (0.23) | 0.01 (0.17)
  Month 24:non-study diagnostic test: number analyzed (Participants) | 263 | 278 | 106
  Month 24:non-study diagnostic test | 0.18 (0.52) | 0.16 (0.53) | 0.13 (0.60)
  Month 24: in nursing home: number analyzed (Participants) | 263 | 278 | 106
  Month 24: in nursing home | -0.00 (0.06) | 0.01 (0.13) | 0.00 (0.20)
  Month 24: home healthcare services: number analyzed (Participants) | 262 | 278 | 106
  Month 24: home healthcare services | 0.02 (0.12) | 0.00 (0.15) | -0.01 (0.10)
  Month 24: required aids/devices: number analyzed (Participants) | 263 | 278 | 106
  Month 24: required aids/devices | 0.05 (0.27) | 0.04 (0.30) | 0.08 (0.27)
  Month 24: non-medical practitioner: number analyzed (Participants) | 263 | 278 | 106
  Month 24: non-medical practitioner | 0.02 (0.19) | 0.02 (0.17) | 0.03 (0.17)
  Month 24: currently employed: number analyzed (Participants) | 263 | 278 | 106
  Month 24: currently employed | -0.04 (0.37) | 0.00 (0.40) | 0.01 (0.32)
  Month 24: feel well enough to work: number analyzed (Participants) | 101 | 108 | 47
  Month 24: feel well enough to work | -0.26 (0.58) | -0.19 (0.51) | -0.13 (0.54)
  Month 24: unable to work due to RA: number analyzed (Participants) | 101 | 108 | 48
  Month 24: unable to work due to RA | 0.30 (0.58) | 0.27 (0.61) | 0.08 (0.50)
  Month 24: lost job/retired early: number analyzed (Participants) | 98 | 106 | 47
  Month 24: lost job/retired early | 0.00 (0.50) | 0.04 (0.46) | 0.04 (0.41)
  Month 24: work disabled due to RA: number analyzed (Participants) | 98 | 105 | 48
  Month 24: work disabled due to RA | 0.18 (0.52) | 0.19 (0.57) | 0.13 (0.53)
  Month 24: retired: number analyzed (Participants) | 102 | 114 | 50
  Month 24: retired | -0.05 (0.38) | -0.05 (0.44) | 0.08 (0.49)
  Month 24: sick leave due to RA: number analyzed (Participants) | 209 | 213 | 79
  Month 24: sick leave due to RA | 0.22 (0.44) | 0.29 (0.46) | 0.16 (0.56)
  Month 24: performed part-time work: number analyzed (Participants) | 210 | 208 | 79
  Month 24: performed part-time work | 0.10 (0.33) | 0.12 (0.34) | 0.15 (0.46)
  Month 24: performed paid work: number analyzed (Participants) | 208 | 213 | 80
  Month 24: performed paid work | 0.24 (0.56) | 0.28 (0.53) | 0.20 (0.56)
  Month 24: unable to do chores: number analyzed (Participants) | 259 | 276 | 106
  Month 24: unable to do chores | 0.41 (0.52) | 0.47 (0.56) | 0.32 (0.58)
  Month 24: chores by housekeeper: number analyzed (Participants) | 261 | 276 | 105
  Month 24: chores by housekeeper | 0.04 (0.27) | 0.08 (0.33) | 0.03 (0.22)
  Month 24: chores by family/friends: number analyzed (Participants) | 263 | 277 | 105
  Month 24: chores by family/friends | 0.40 (0.52) | 0.40 (0.53) | 0.31 (0.54)

73. Secondary Outcome: Change From Baseline in Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Months 3 and 6
Description: as for outcome 64
Time Frame: Months 3 and 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 215 | 250 | 115
events
  Month 3: doctor visits: number analyzed (Participants) | 213 | 249 | 115
  Month 3: doctor visits | -1.83 (5.24) | -1.12 (4.13) | -1.52 (5.46)
  Month 3: RA-related doctor visit | -0.55 (1.30) | -0.50 (1.14) | -0.48 (0.99)
  Month 3: hospital ER visit: number analyzed (Participants) | 3 | 5 | 0
  Month 3: hospital ER visit | -4.33 (5.86) | 1.60 (3.78) |
  Month 3: RA-related ER visit: number analyzed (Participants) | 3 | 5 | 0
  Month 3: RA-related ER visit | -0.67 (1.15) | -1.00 (1.58) |
  Month 3: hospitalization: number analyzed (Participants) | 0 | 2 | 0
  Month 3: hospitalization |  | 0.00 (0.00) |
  Month 3: RA-related hospitalization: number analyzed (Participants) | 0 | 2 | 0
  Month 3: RA-related hospitalization |  | -0.50 (0.71) |
  Month 3: non-study diagnostic test: number analyzed (Participants) | 11 | 23 | 8
  Month 3: non-study diagnostic test | -0.73 (2.24) | -0.61 (1.50) | 0.38 (1.19)
  Month 3: RA-related diagnostic test: number analyzed (Participants) | 11 | 24 | 8
  Month 3: RA-related diagnostic test | -0.73 (1.01) | -0.67 (1.20) | -0.50 (0.93)
  Month 3:non-medical practitioner visit: number analyzed (Participants) | 3 | 3 | 1
  Month 3:non-medical practitioner visit | -62.33 (102.11) | -2.33 (2.52) | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 3:RA-related non-medical visit: number analyzed (Participants) | 3 | 3 | 1
  Month 3:RA-related non-medical visit | -0.67 (0.58) | -0.33 (0.58) | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 6: doctor visit: number analyzed (Participants) | 186 | 213 | 99
  Month 6: doctor visit | -2.44 (4.87) | -1.98 (4.65) | -2.72 (5.43)
  Month 6: RA-related doctor visit: number analyzed (Participants) | 190 | 214 | 99
  Month 6: RA-related doctor visit | -0.69 (1.27) | -0.66 (1.23) | -0.77 (1.10)
  Month 6: hospital ER visit: number analyzed (Participants) | 0 | 5 | 0
  Month 6: hospital ER visit |  | 0.60 (1.34) |
  Month 6: RA-related ER visit: number analyzed (Participants) | 0 | 5 | 0
  Month 6: RA-related ER visit |  | -0.40 (1.14) |
  Month 6: hospitalization: number analyzed (Participants) | 0 | 2 | 1
  Month 6: hospitalization |  | 0.00 (0.00) | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 6: RA-related hospitalization: number analyzed (Participants) | 0 | 2 | 1
  Month 6: RA-related hospitalization |  | -1.50 (0.71) | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 6: non-study diagnostic test: number analyzed (Participants) | 5 | 15 | 6
  Month 6: non-study diagnostic test | -0.60 (1.52) | -0.40 (1.30) | -0.67 (2.16)
  Month 6: RA related diagnostic test: number analyzed (Participants) | 5 | 16 | 6
  Month 6: RA related diagnostic test | -0.80 (1.64) | -0.88 (1.09) | -0.67 (0.82)
  Month 6:non-medical practitioner visit: number analyzed (Participants) | 2 | 1 | 1
  Month 6:non-medical practitioner visit | -8.00 (2.83) | -5.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 1.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 6:RA-related non-medical visit: number analyzed (Participants) | 2 | 1 | 1
  Month 6:RA-related non-medical visit | 0.00 (0.00) | -1.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 1.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.

74. Secondary Outcome: Change From Baseline in Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Months 12, 18, and 24
Description: RA-HCRU assessed HC usage during previous 3 months for direct or indirect medical cost domains. Any RA/non-RA related number of events including visits to doctor, non-medical practitioner, hospital ER treatment, hospitalizations, number of surgeries, diagnostic tests, and devices/aids used were reported.
Time Frame: Months 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 167 | 174 | 78
events
  Month 12: doctor visit: number analyzed (Participants) | 166 | 174 | 78
  Month 12: doctor visit | -2.57 (5.87) | -2.32 (4.33) | -3.17 (5.86)
  Month 12: RA-related doctor visit | -0.72 (1.30) | -0.68 (1.12) | -0.72 (1.14)
  Month 12: hospital ER visit: number analyzed (Participants) | 4 | 2 | 0
  Month 12: hospital ER visit | -3.50 (5.07) | 0.00 (0.00) |
  Month 12: RA-related ER visit: number analyzed (Participants) | 4 | 2 | 1
  Month 12: RA-related ER visit | -1.25 (0.96) | -1.00 (1.41) | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 12: hospitalization: number analyzed (Participants) | 2 | 0 | 0
  Month 12: hospitalization | 0.00 (0.00) |  |
  Month 12: RA-related hospitalization: number analyzed (Participants) | 2 | 0 | 0
  Month 12: RA-related hospitalization | -0.50 (0.71) |  |
  Month 12:non-study diagnostic tests: number analyzed (Participants) | 11 | 17 | 5
  Month 12:non-study diagnostic tests | -0.09 (2.88) | -0.71 (1.69) | -1.00 (1.00)
  Month 12: RA-related diagnostic tests: number analyzed (Participants) | 11 | 17 | 5
  Month 12: RA-related diagnostic tests | -0.82 (1.25) | -0.88 (1.69) | -0.60 (0.89)
  Month 12:non-medical practitioner visit: number analyzed (Participants) | 1 | 2 | 0
  Month 12:non-medical practitioner visit | -8.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 8.00 (11.31) |
  Month 12:RA-related non-medical visit: number analyzed (Participants) | 1 | 2 | 0
  Month 12:RA-related non-medical visit | -2.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 0.00 (0.00) |
  Month 18: doctor visits: number analyzed (Participants) | 148 | 138 | 64
  Month 18: doctor visits | -2.58 (4.37) | -1.98 (3.67) | -2.20 (6.97)
  Month 18: RA-related doctor visit: number analyzed (Participants) | 150 | 138 | 64
  Month 18: RA-related doctor visit | -0.69 (1.17) | -0.51 (1.03) | -0.69 (1.21)
  Month 18: hospital ER visit: number analyzed (Participants) | 1 | 1 | 0
  Month 18: hospital ER visit | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | -1.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |
  Month 18: RA-related ER visit: number analyzed (Participants) | 1 | 1 | 2
  Month 18: RA-related ER visit | 1.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | -1.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | -0.50 (0.71)
  Month 18: hospitalization: number analyzed (Participants) | 0 | 0 | 1
  Month 18: hospitalization |  |  | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint
  Month 18:RA-related hospitalization: number analyzed (Participants) | 0 | 0 | 1
  Month 18:RA-related hospitalization |  |  | -1.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 18: outpatient surgery: number analyzed (Participants) | 1 | 0 | 0
  Month 18: outpatient surgery | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |  |
  Month 18:RA-related outpatient surgery: number analyzed (Participants) | 1 | 0 | 0
  Month 18:RA-related outpatient surgery | 2.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |  |
  Month 18:non-study diagnostic test: number analyzed (Participants) | 11 | 5 | 2
  Month 18:non-study diagnostic test | -1.55 (2.73) | 0.00 (2.24) | -0.50 (2.12)
  Month 24:RA-related diagnostic test: number analyzed (Participants) | 3 | 11 | 2
  Month 24:RA-related diagnostic test | -0.33 (0.58) | -0.64 (0.67) | -0.50 (0.71)
  Month 18:non-medical practitioner visit: number analyzed (Participants) | 1 | 3 | 0
  Month 18:non-medical practitioner visit | -10.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | -15.67 (28.01) |
  Month 18:RA-related non-medical visit: number analyzed (Participants) | 1 | 3 | 0
  Month 18:RA-related non-medical visit | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | 0.33 (1.53) |
  Month 24: doctor visit: number analyzed (Participants) | 134 | 130 | 56
  Month 24: doctor visit | -2.78 (6.00) | -1.65 (5.42) | -2.41 (6.48)
  Month 24: RA-related doctor visit: number analyzed (Participants) | 134 | 128 | 56
  Month 24: RA-related doctor visit | -0.71 (1.37) | -0.63 (1.15) | -0.63 (1.10)
  Month 24: hospital ER visit: number analyzed (Participants) | 3 | 1 | 0
  Month 24: hospital ER visit | 0.00 (0.00) | -1.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |
  Month 24: RA-related ER visit: number analyzed (Participants) | 3 | 1 | 0
  Month 24: RA-related ER visit | -0.67 (1.15) | -2.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |
  Month 24: outpatient surgery: number analyzed (Participants) | 1 | 0 | 0
  Month 24: outpatient surgery | 4.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |  |
  Month 24:RA-relate outpatient surgery: number analyzed (Participants) | 1 | 0 | 0
  Month 24:RA-relate outpatient surgery | -1.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |  |
  Month 24:non-study diagnostic test: number analyzed (Participants) | 4 | 11 | 2
  Month 24:non-study diagnostic test | -1.50 (4.20) | -0.18 (1.08) | -0.50 (0.71)
  Month 24:RA related diagnostic test: number analyzed (Participants) | 3 | 11 | 2
  Month 24:RA related diagnostic test | -0.33 (0.58) | -0.64 (0.67) | -0.50 (0.71)
  Month 24:non-medical practitioner visit: number analyzed (Participants) | 1 | 2 | 0
  Month 24:non-medical practitioner visit | -168.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | -1.00 (1.41) |
  Month 24:RA-related non-medical visit: number analyzed (Participants) | 1 | 3 | 0
  Month 24:RA-related non-medical visit | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. | -0.33 (0.58) |

75. Secondary Outcome: Change From Baseline in Number of Days as Assessed Using RA-HCRU at Months 3 and 6
Description: RA-HCRU assessed HC usage during previous 3 months for direct or indirect medical cost domains. Any RA or non-RA related number of days spent in hospital, nursing home, aids/devices used, on sick leave, work per week, performed part time work, performed paid work, chores done by housekeeper and chores done by family/friends.
Time Frame: Months 3 and 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 154 | 164 | 74
days
  Month 3: hospital length of stay: number analyzed (Participants) | 0 | 2 | 0
  Month 3: hospital length of stay |  | -10.00 (7.07) |
  Month 3: days in nursing home: number analyzed (Participants) | 0 | 1 | 0
  Month 3: days in nursing home |  | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |
  Month 3: days aids/devices used: number analyzed (Participants) | 12 | 14 | 8
  Month 3: days aids/devices used | -45.92 (91.00) | -12.36 (173.11) | -65.50 (200.00)
  Month 3: RA-related aids used: number analyzed (Participants) | 13 | 14 | 8
  Month 3: RA-related aids used | -0.31 (1.11) | -0.43 (1.91) | -0.25 (2.05)
  Month 3: days of work per week | 0.13 (0.69) | 0.06 (0.74) | -0.01 (0.54)
  Month 3:days on sick leave due to RA: number analyzed (Participants) | 30 | 24 | 17
  Month 3:days on sick leave due to RA | 0.40 (32.44) | 7.58 (26.57) | 10.94 (33.96)
  Month 3: days of part time work: number analyzed (Participants) | 12 | 7 | 6
  Month 3: days of part time work | 1.92 (32.76) | 15.14 (34.60) | -0.17 (26.90)
  Month 3: paid work, bothered by RA: number analyzed (Participants) | 71 | 70 | 40
  Month 3: paid work, bothered by RA | -15.31 (39.58) | -15.16 (34.88) | -9.30 (31.97)
  Month 3: chores by housekeeper: number analyzed (Participants) | 10 | 23 | 7
  Month 3: chores by housekeeper | -20.70 (35.90) | -11.61 (31.25) | -9.29 (36.09)
  Month 3: chores by family: number analyzed (Participants) | 85 | 97 | 51
  Month 3: chores by family | -19.14 (40.06) | -17.71 (36.57) | -12.18 (35.70)
  Month 6: hospital length of stay: number analyzed (Participants) | 0 | 2 | 1
  Month 6: hospital length of stay |  | -22.00 (2.83) | 8.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 6: days in nursing home: number analyzed (Participants) | 0 | 1 | 0
  Month 6: days in nursing home |  | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |
  Month 6: days aids/devices used: number analyzed (Participants) | 14 | 7 | 5
  Month 6: days aids/devices used | -46.93 (127.42) | 58.00 (126.45) | -93.20 (211.52)
  Month 6: RA-related aids used: number analyzed (Participants) | 14 | 8 | 5
  Month 6: RA-related aids used | -0.64 (1.50) | 0.13 (0.99) | -1.60 (2.70)
  Month 6: days of work per week: number analyzed (Participants) | 148 | 153 | 65
  Month 6: days of work per week | 0.07 (0.67) | 0.03 (0.73) | 0.00 (0.50)
  Month 6:days on sick leave due to RA: number analyzed (Participants) | 11 | 16 | 11
  Month 6:days on sick leave due to RA | -18.27 (17.19) | 13.56 (27.92) | 13.82 (46.97)
  Month 6: days of part time work: number analyzed (Participants) | 4 | 5 | 1
  Month 6: days of part time work | 11.50 (14.34) | -2.60 (18.57) | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 6: paid work, bothered by RA: number analyzed (Participants) | 51 | 44 | 32
  Month 6: paid work, bothered by RA | -15.90 (36.80) | -16.43 (30.15) | -7.81 (38.47)
  Month 6: chores by housekeeper: number analyzed (Participants) | 10 | 16 | 5
  Month 6: chores by housekeeper | -13.80 (19.66) | -11.94 (33.28) | -2.40 (7.70)
  Month 6: chores by family: number analyzed (Participants) | 64 | 57 | 34
  Month 6: chores by family | -14.94 (39.94) | -20.54 (37.40) | -20.94 (40.56)

76. Secondary Outcome: Change From Baseline in Number of Days as Assessed Using RA-HCRU at Months 12, 18, and 24
Description: as for outcome 75
Time Frame: Months 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: days
Groups:
- MTX 10,15, or 20 mg, Weekly: Participants received MTX capsules at doses of 10 to 20 mg per week and matching placebo CP-690,550 tablets, orally, BID, for up to 24 months. MTX dose was titrated to a maximum of 20 mg/week as follows: 10 mg/once weekly for 4 weeks, if tolerated the dose was titrated to 15 mg/once weekly for 4 weeks, if tolerated the dose was titrated to 20 mg/once weekly. One dose reduction was allowed for lack of tolerance.
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10,15, or 20 mg, Weekly
Number analyzed (Participants) | 131 | 130 | 57
days
  Month 12: hospital length of stay: number analyzed (Participants) | 2 | 0 | 0
  Month 12: hospital length of stay | -2.00 (2.83) |  |
  Month 12: days in nursing home: number analyzed (Participants) | 0 | 2 | 0
  Month 12: days in nursing home |  | 3.50 (4.95) |
  Month 12: days aids/devices used: number analyzed (Participants) | 14 | 4 | 2
  Month 12: days aids/devices used | -27.07 (159.25) | -5.00 (81.85) | -75.00 (63.64)
  Month 12: RA-related aids used: number analyzed (Participants) | 13 | 4 | 2
  Month 12: RA-related aids used | -0.46 (1.71) | 0.00 (0.82) | 0.00 (0.00)
  Month 12: days of work per week | 0.11 (0.86) | -0.01 (0.66) | 0.04 (0.42)
  Month 12:days on sick leave due to RA: number analyzed (Participants) | 12 | 5 | 5
  Month 12:days on sick leave due to RA | 5.25 (28.21) | -2.80 (16.41) | -2.20 (2.49)
  Month 12: days of part-time work: number analyzed (Participants) | 5 | 3 | 0
  Month 12: days of part-time work | 2.20 (6.83) | -15.00 (17.00) |
  Month 12:paid work, bothered by RA: number analyzed (Participants) | 41 | 32 | 23
  Month 12:paid work, bothered by RA | -18.49 (28.09) | -12.63 (34.77) | -12.35 (37.16)
  Month 12: chores by housekeeper: number analyzed (Participants) | 7 | 12 | 3
  Month 12: chores by housekeeper | -8.43 (14.55) | -1.92 (6.19) | 4.67 (5.03)
  Month 12: chores by family: number analyzed (Participants) | 45 | 40 | 21
  Month 12: chores by family | -13.11 (34.25) | -20.05 (44.57) | -15.24 (29.17)
  Month 18: hospital length of stay: number analyzed (Participants) | 0 | 0 | 1
  Month 18: hospital length of stay |  |  | 21.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 18: days aids/devices used: number analyzed (Participants) | 11 | 4 | 3
  Month 18: days aids/devices used | 65.09 (81.85) | 96.00 (53.39) | -77.33 (289.83)
  Month 18: RA-related aids used: number analyzed (Participants) | 11 | 4 | 3
  Month 18: RA-related aids used | 0.82 (0.87) | 1.00 (0.82) | 0.00 (1.73)
  Month 18: days of work per week: number analyzed (Participants) | 120 | 115 | 47
  Month 18: days of work per week | 0.13 (0.85) | -0.04 (0.85) | -0.06 (0.60)
  Month 18:days on sick leave due to RA: number analyzed (Participants) | 5 | 9 | 3
  Month 18:days on sick leave due to RA | -4.80 (13.18) | -6.78 (8.94) | -31.67 (47.93)
  Month 18: days of part time work: number analyzed (Participants) | 5 | 1 | 0
  Month 18: days of part time work | -1.00 (4.85) | -35.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |
  Month 18:paid work, bothered by RA: number analyzed (Participants) | 36 | 34 | 15
  Month 18:paid work, bothered by RA | -15.19 (39.72) | -20.12 (33.90) | -15.07 (43.23)
  Month 18: chores by housekeeper: number analyzed (Participants) | 4 | 9 | 2
  Month 18: chores by housekeeper | -24.50 (32.54) | -19.22 (28.80) | -5.50 (7.78)
  Month 18: chores by family: number analyzed (Participants) | 33 | 30 | 14
  Month 18: chores by family | -9.15 (34.94) | -14.17 (35.55) | 3.36 (30.47)
  Month 24: days aids/devices used: number analyzed (Participants) | 10 | 4 | 4
  Month 24: days aids/devices used | 79.90 (127.89) | -38.50 (50.79) | -45.00 (198.24)
  Month 24: RA-related aids used: number analyzed (Participants) | 10 | 4 | 4
  Month 24: RA-related aids used | 1.10 (1.20) | -0.50 (1.00) | -0.75 (2.36)
  Month 24: days of work per week: number analyzed (Participants) | 111 | 105 | 42
  Month 24: days of work per week | 0.06 (0.87) | 0.05 (0.78) | 0.05 (0.79)
  Month 24:days on sick leave due to RA: number analyzed (Participants) | 7 | 2 | 1
  Month 24:days on sick leave due to RA | -3.86 (7.06) | -3.00 (5.66) | -5.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 24: days of part time work: number analyzed (Participants) | 3 | 1 | 0
  Month 24: days of part time work | 1.67 (6.03) | -45.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |
  Month 24: paid work, bothered by RA: number analyzed (Participants) | 26 | 30 | 15
  Month 24: paid work, bothered by RA | -12.54 (37.97) | -23.63 (26.77) | -22.47 (25.29)
  Month 24: chores by housekeeper: number analyzed (Participants) | 6 | 8 | 2
  Month 24: chores by housekeeper | -15.33 (24.10) | -12.00 (29.28) | 0.00 (5.66)
  Month 24: chores by family: number analyzed (Participants) | 30 | 28 | 14
  Month 24: chores by family | -7.30 (31.83) | -27.54 (37.94) | -13.86 (37.70)

77. Secondary Outcome: Change From Baseline in Number of Hours Per Day as Assessed Using RA-HCRU at Months 3 and 6
Description: RA-HCRU assessed HC usage during previous 3 months for direct or indirect medical cost domains. Any RA or non-RA related number of hours spent per day for home HC services, chores done by housekeeper, chores done by family or friends, work done and work missed were reported.
Time Frame: Months 3 and 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 154 | 165 | 74
hours per day
  Month 3: home healthcare services: number analyzed (Participants) | 0 | 2 | 0
  Month 3: home healthcare services |  | -1.00 (1.41) |
  Month 3:RA-related home HC services: number analyzed (Participants) | 0 | 2 | 0
  Month 3:RA-related home HC services |  | 0.00 (0.00) |
  Month 3: work done | 0.23 (4.19) | 0.34 (6.12) | 0.80 (3.82)
  Month 3: missed work due to RA: number analyzed (Participants) | 11 | 7 | 6
  Month 3: missed work due to RA | -1.00 (8.94) | 1.29 (5.06) | 3.00 (9.36)
  Month 3: chores by housekeeper: number analyzed (Participants) | 10 | 23 | 7
  Month 3: chores by housekeeper | -0.80 (1.62) | -0.61 (2.37) | -1.14 (1.86)
  Month 3: chores by family: number analyzed (Participants) | 86 | 96 | 51
  Month 3: chores by family | -1.98 (4.92) | -0.39 (3.90) | -1.63 (5.14)
  Month 6: work done: number analyzed (Participants) | 148 | 155 | 65
  Month 6: work done | -0.34 (4.32) | 0.03 (4.79) | 0.23 (1.48)
  Month 6: missed work due to RA: number analyzed (Participants) | 3 | 5 | 1
  Month 6: missed work due to RA | -1.67 (5.13) | -0.40 (1.14) | -4.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 6: chores by housekeeper: number analyzed (Participants) | 10 | 16 | 5
  Month 6: chores by housekeeper | -1.10 (2.38) | -0.25 (3.19) | -0.20 (1.30)
  Month 6: chores by family: number analyzed (Participants) | 63 | 57 | 33
  Month 6: chores by family | -0.68 (4.15) | -0.51 (3.02) | -0.45 (6.24)

78. Secondary Outcome: Change From Baseline in Number of Hours Per Day as Assessed Using RA-HCRU at Months 12, 18, and 24
Description: as for outcome 77
Time Frame: Months 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 131 | 131 | 57
hours per day
  Month 12: work done | 0.34 (4.30) | -0.21 (4.37) | 0.75 (4.43)
  Month 12: missed work due to RA: number analyzed (Participants) | 5 | 3 | 0
  Month 12: missed work due to RA | -1.60 (4.93) | 0.00 (1.00) |
  Month 12: chores by housekeeper: number analyzed (Participants) | 7 | 13 | 2
  Month 12: chores by housekeeper | 0.29 (2.63) | -5.23 (18.66) | -0.50 (0.71)
  Month 12: chores by family: number analyzed (Participants) | 45 | 40 | 21
  Month 12: chores by family | -0.67 (4.67) | -1.35 (6.69) | -0.24 (3.10)
  Month 18: work done: number analyzed (Participants) | 120 | 116 | 47
  Month 18: work done | 0.17 (4.56) | 0.16 (5.24) | 0.04 (1.37)
  Month 18: missed work due to RA: number analyzed (Participants) | 5 | 1 | 0
  Month 18: missed work due to RA | -5.80 (11.97) | 1.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |
  Month 18: chores by housekeeper: number analyzed (Participants) | 4 | 9 | 1
  Month 18: chores by housekeeper | -2.00 (2.16) | -8.78 (22.26) | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 18: chores by family: number analyzed (Participants) | 33 | 30 | 12
  Month 18: chores by family | 0.03 (3.43) | -1.57 (5.25) | -0.17 (1.19)
  Month 24: work done: number analyzed (Participants) | 111 | 106 | 42
  Month 24: work done | 0.42 (5.37) | -0.04 (2.51) | 0.17 (1.32)
  Month 24: missed work due to RA: number analyzed (Participants) | 3 | 1 | 0
  Month 24: missed work due to RA | -5.33 (7.57) | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint. |
  Month 24: chores by housekeeper: number analyzed (Participants) | 6 | 8 | 1
  Month 24: chores by housekeeper | 0.17 (3.06) | 0.50 (1.51) | 1.00 (NA) — Standard deviation could not be calculated as only 1 participant contributed data for this variable at this timepoint.
  Month 24: chores by family: number analyzed (Participants) | 30 | 27 | 15
  Month 24: chores by family | -0.97 (3.40) | -1.00 (3.00) | -0.47 (1.36)

79. Secondary Outcome: Change From Baseline in Work Performance in Past 3 Months on Days Bothered as Assessed Using RA-HCRU
Description: as for outcome 70
Time Frame: Months 3, 6, 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 242 | 258 | 113
units on a scale
  Month 3 | -1.40 (2.88) | -1.45 (3.90) | -0.81 (2.94)
  Month 6: number analyzed (Participants) | 233 | 243 | 104
  Month 6 | -2.11 (2.92) | -2.44 (2.97) | -1.22 (3.39)
  Month 12: number analyzed (Participants) | 210 | 210 | 88
  Month 12 | -2.15 (3.22) | -2.68 (3.17) | -1.51 (2.93)
  Month 18: number analyzed (Participants) | 195 | 186 | 72
  Month 18 | -2.28 (3.25) | -2.62 (3.15) | -2.22 (3.33)
  Month 24: number analyzed (Participants) | 173 | 174 | 64
  Month 24 | -2.24 (3.36) | -2.38 (3.11) | -1.88 (3.24)

80. Secondary Outcome: Medical Outcomes Study Sleep Scale (MOS-SS) at Baseline and Months 1, 2, and 3
Description: Participant-rated 12 item questionnaire to assess constructs of sleep over past week. 7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence (range: 0-100); sleep quantity (range: 0-24), optimal sleep (yes or no). 9-item index measures of sleep disturbance provide composite scores: sleep problem summary, overall sleep problem. Except Adequacy, Optimal, Quantity of sleep, higher cores=more impairment. Scores transformed (actual raw score [RS] minus lowest possible score divided by possible RS range*100); total score range: 0-100, higher score=more intensity of attribute.
Time Frame: Baseline and Months 1, 2, and 3
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 372 | 397 | 186
units on a scale
  BL: overall sleep problem | 42.65 (19.48) | 42.82 (20.51) | 42.84 (18.07)
  BL: sleep problem summary | 40.66 (19.84) | 41.43 (20.77) | 41.13 (18.20)
  BL: somnolence | 35.77 (21.68) | 36.68 (22.28) | 38.21 (21.19)
  BL: snoring | 34.30 (32.90) | 31.99 (32.37) | 32.58 (32.13)
  BL: sleep disturbance | 45.61 (25.91) | 44.77 (26.54) | 44.30 (25.52)
  BL: awaken short of breath | 20.43 (25.52) | 19.35 (24.42) | 18.71 (23.40)
  BL: adequacy | 46.29 (26.63) | 44.41 (26.95) | 44.65 (26.22)
  Month 1: overall sleep problem: number analyzed (Participants) | 365 | 392 | 184
  Month 1: overall sleep problem | 33.74 (18.23) | 33.60 (20.19) | 38.15 (17.57)
  Month 1: sleep problem summary: number analyzed (Participants) | 365 | 392 | 184
  Month 1: sleep problem summary | 33.11 (18.84) | 33.21 (20.83) | 37.28 (18.17)
  Month 1: somnolence: number analyzed (Participants) | 365 | 392 | 184
  Month 1: somnolence | 29.75 (19.71) | 29.15 (19.65) | 35.11 (19.21)
  Month 1: snoring: number analyzed (Participants) | 365 | 392 | 184
  Month 1: snoring | 30.30 (29.30) | 28.21 (30.26) | 30.76 (31.63)
  Month 1: sleep disturbance: number analyzed (Participants) | 365 | 392 | 184
  Month 1: sleep disturbance | 33.81 (22.52) | 33.58 (24.94) | 37.09 (23.70)
  Month 1: awaken short of breath: number analyzed (Participants) | 365 | 392 | 184
  Month 1: awaken short of breath | 16.66 (22.84) | 17.40 (23.90) | 17.07 (22.76)
  Month 1: adequacy: number analyzed (Participants) | 365 | 392 | 184
  Month 1: adequacy | 53.64 (26.20) | 54.08 (27.32) | 47.23 (24.62)
  Month 2: overall sleep problem: number analyzed (Participants) | 359 | 388 | 178
  Month 2: overall sleep problem | 31.73 (18.37) | 32.76 (20.25) | 35.25 (17.24)
  Month 2: sleep problem summary: number analyzed (Participants) | 360 | 388 | 178
  Month 2: sleep problem summary | 31.26 (18.68) | 32.71 (20.63) | 34.66 (17.19)
  Month 2: somnolence: number analyzed (Participants) | 260 | 388 | 178
  Month 2: somnolence | 27.96 (19.32) | 29.02 (21.10) | 31.65 (19.75)
  Month 2: snoring: number analyzed (Participants) | 359 | 388 | 178
  Month 2: snoring | 31.09 (28.38) | 28.92 (30.40) | 28.20 (28.56)
  Month 2: sleep disturbance: number analyzed (Participants) | 359 | 388 | 178
  Month 2: sleep disturbance | 30.93 (23.06) | 32.31 (24.56) | 34.56 (22.32)
  Month 2: awaken short of breath: number analyzed (Participants) | 360 | 388 | 178
  Month 2: awaken short of breath | 15.44 (21.04) | 17.16 (22.07) | 15.96 (20.21)
  Month 2: adequacy: number analyzed (Participants) | 360 | 388 | 178
  Month 2: adequacy | 54.83 (26.71) | 55.08 (27.81) | 50.84 (25.73)
  Month 3: overall sleep problem: number analyzed (Participants) | 352 | 382 | 172
  Month 3: overall sleep problem | 30.07 (18.59) | 31.55 (19.86) | 33.93 (18.86)
  Month 3: sleep problem summary: number analyzed (Participants) | 352 | 382 | 172
  Month 3: sleep problem summary | 29.87 (19.22) | 31.76 (20.55) | 33.66 (19.82)
  Month 3: somnolence: number analyzed (Participants) | 352 | 383 | 172
  Month 3: somnolence | 27.18 (18.34) | 29.16 (20.99) | 30.39 (19.13)
  Month 3: snoring: number analyzed (Participants) | 352 | 383 | 172
  Month 3: snoring | 30.06 (30.12) | 27.94 (30.11) | 28.60 (28.46)
  Month 3: sleep disturbance: number analyzed (Participants) | 352 | 382 | 172
  Month 3: sleep disturbance | 29.24 (22.54) | 29.83 (24.10) | 32.76 (23.87)
  Month 3: awaken short of breath: number analyzed (Participants) | 352 | 383 | 172
  Month 3: awaken short of breath | 16.76 (22.64) | 16.87 (22.25) | 16.74 (21.71)
  Month 3: adequacy: number analyzed (Participants) | 352 | 383 | 172
  Month 3: adequacy | 58.55 (27.53) | 55.27 (27.60) | 51.74 (26.72)

81. Secondary Outcome: Percentage of Participants With Optimal Sleep Assessed Using MOS-SS
Description: MOS-SS: participant-rated 12 item questionnaire to assess constructs of sleep over past week. It included 7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence, sleep quantity and optimal sleep. Participants responded whether their sleep was optimal or not by choosing yes or no. Number of participants with optimal sleep are reported
Time Frame: Months 1, 2, 3, 6, 12, 18, and 24
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 367 | 393 | 184
percentage of participants
  Month 1 | 55.31 | 55.22 | 51.09
  Month 2: number analyzed (Participants) | 361 | 388 | 178
  Month 2 | 57.06 | 55.41 | 48.88
  Month 3: number analyzed (Participants) | 356 | 383 | 172
  Month 3 | 58.71 | 60.05 | 51.74
  Month 6: number analyzed (Participants) | 340 | 367 | 158
  Month 6 | 61.76 | 58.04 | 58.23
  Month 12: number analyzed (Participants) | 315 | 332 | 136
  Month 12 | 58.10 | 58.43 | 50.00
  Month 18: number analyzed (Participants) | 284 | 295 | 116
  Month 18 | 63.03 | 62.37 | 52.59
  Month 24: number analyzed (Participants) | 264 | 281 | 106
  Month 24 | 61.74 | 55.87 | 55.66

82. Secondary Outcome: Medical Outcomes Study Sleep Scale (MOS-SS) at Months 6, 12, 18, and 24
Description: as for outcome 80
Time Frame: Months 6, 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 340 | 366 | 158
units on a scale
  Month 6: overall sleep problem | 30.73 (18.51) | 30.05 (20.09) | 32.71 (19.54)
  Month 6: sleep problem summary | 30.59 (19.02) | 29.81 (20.75) | 32.17 (19.47)
  Month 6: somnolence | 26.82 (18.62) | 27.34 (20.69) | 29.79 (19.76)
  Month 6: snoring: number analyzed (Participants) | 340 | 365 | 157
  Month 6: snoring | 30.12 (29.49) | 31.01 (30.68) | 27.39 (29.11)
  Month 6: sleep disturbance | 29.26 (22.20) | 28.61 (24.64) | 31.76 (25.72)
  Month 6: awaken short of breath | 17.00 (22.24) | 14.70 (21.28) | 14.68 (20.98)
  Month 6: adequacy | 56.09 (26.92) | 56.45 (27.84) | 53.61 (26.74)
  Month 12: overall sleep problem: number analyzed (Participants) | 315 | 330 | 135
  Month 12: overall sleep problem | 30.01 (17.75) | 29.30 (18.50) | 33.49 (18.56)
  Month 12: sleep problem summary: number analyzed (Participants) | 315 | 330 | 135
  Month 12: sleep problem summary | 29.89 (18.87) | 29.10 (18.99) | 33.70 (19.36)
  Month 12: somnolence: number analyzed (Participants) | 315 | 330 | 135
  Month 12: somnolence | 26.62 (18.29) | 27.17 (20.09) | 31.11 (18.47)
  Month 12: snoring: number analyzed (Participants) | 315 | 330 | 135
  Month 12: snoring | 32.13 (28.80) | 31.76 (31.54) | 30.67 (27.84)
  Month 12: sleep disturbance: number analyzed (Participants) | 315 | 330 | 135
  Month 12: sleep disturbance | 28.73 (20.85) | 27.75 (22.73) | 32.44 (23.52)
  Month 12: awaken short of breath: number analyzed (Participants) | 315 | 330 | 135
  Month 12: awaken short of breath | 15.81 (22.01) | 14.73 (21.89) | 16.59 (21.10)
  Month 12: adequacy: number analyzed (Participants) | 315 | 330 | 135
  Month 12: adequacy | 56.98 (27.00) | 58.18 (27.13) | 54.15 (26.80)
  Month 18: overall sleep problem: number analyzed (Participants) | 284 | 293 | 116
  Month 18: overall sleep problem | 29.99 (17.44) | 28.54 (17.92) | 31.93 (19.62)
  Month 18: sleep problem summary: number analyzed (Participants) | 284 | 293 | 116
  Month 18: sleep problem summary | 29.94 (17.82) | 28.15 (18.38) | 32.24 (20.72)
  Month 18: somnolence: number analyzed (Participants) | 284 | 293 | 116
  Month 18: somnolence | 25.77 (17.62) | 26.73 (18.78) | 28.68 (19.90)
  Month 18:snoring: number analyzed (Participants) | 283 | 293 | 115
  Month 18:snoring | 33.07 (28.88) | 31.13 (29.89) | 29.74 (29.90)
  Month 18: sleep disturbance: number analyzed (Participants) | 284 | 293 | 116
  Month 18: sleep disturbance | 29.04 (21.28) | 27.30 (21.32) | 29.31 (22.59)
  Month 18: awaken short of breath: number analyzed (Participants) | 284 | 293 | 116
  Month 18: awaken short of breath | 15.42 (20.11) | 13.38 (19.82) | 16.55 (21.47)
  Month 18: adequacy: number analyzed (Participants) | 284 | 293 | 116
  Month 18: adequacy | 57.11 (26.35) | 59.01 (27.11) | 53.62 (29.50)
  Month 24: overall sleep problem: number analyzed (Participants) | 264 | 278 | 106
  Month 24: overall sleep problem | 29.78 (17.64) | 29.55 (19.26) | 32.25 (19.17)
  Month 24: sleep problem summary: number analyzed (Participants) | 264 | 278 | 106
  Month 24: sleep problem summary | 30.01 (18.21) | 29.57 (19.80) | 31.79 (19.69)
  Month 24: somnolence: number analyzed (Participants) | 264 | 278 | 106
  Month 24: somnolence | 25.71 (18.41) | 26.98 (20.53) | 28.36 (18.36)
  Month 24: snoring: number analyzed (Participants) | 262 | 278 | 106
  Month 24: snoring | 32.44 (29.18) | 30.22 (30.53) | 30.00 (28.32)
  Month 24: sleep disturbance: number analyzed (Participants) | 264 | 278 | 106
  Month 24: sleep disturbance | 29.03 (21.00) | 27.74 (23.40) | 31.43 (23.59)
  Month 24: awaken short of breath: number analyzed (Participants) | 264 | 278 | 106
  Month 24: awaken short of breath | 15.45 (21.23) | 15.90 (20.86) | 16.60 (19.99)
  Month 24: adequacy: number analyzed (Participants) | 264 | 278 | 106
  Month 24: adequacy | 57.46 (28.15) | 57.52 (27.70) | 56.42 (26.66)

83. Secondary Outcome: Change From Baseline in MOS-SS at Months 1, 2, and 3
Description: as for outcome 80
Time Frame: Months 1, 2, and 3
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 364 | 392 | 184
units on a scale
  Month 1: overall sleep problem | -8.95 (0.86) | -9.14 (0.83) | -4.72 (1.19)
  Month 1: sleep problem summary | -7.85 (0.90) | -8.12 (0.86) | -3.98 (1.24)
  Month 1: somnolence | -6.35 (0.95) | -7.31 (0.91) | -2.15 (1.31)
  Month 1: snoring | -3.12 (1.19) | -3.72 (1.14) | -1.66 (1.65)
  Month 1: quantity: number analyzed (Participants) | 364 | 391 | 183
  Month 1: quantity | 0.41 (0.06) | 0.38 (0.06) | 0.26 (0.09)
  Month 1: sleep disturbance | -11.28 (1.07) | -11.06 (1.03) | -7.36 (1.48)
  Month 1: awaken short of breath | -2.81 (1.04) | -1.92 (1.00) | -2.00 (1.44)
  Month 1: adequacy | 8.56 (1.33) | 9.73 (1.28) | 2.83 (1.84)
  Month 2: overall sleep problem: number analyzed (Participants) | 360 | 388 | 178
  Month 2: overall sleep problem | -11.08 (0.87) | -10.15 (0.83) | -7.62 (1.20)
  Month 2: sleep problem summary: number analyzed (Participants) | 324 | 345 | 164
  Month 2: sleep problem summary | -9.81 (0.90) | -8.75 (0.86) | -6.54 (1.25)
  Month 2: somnolence: number analyzed (Participants) | 360 | 388 | 178
  Month 2: somnolence | -8.11 (0.95) | -7.56 (0.91) | -5.45 (1.33)
  Month 2: snoring: number analyzed (Participants) | 359 | 388 | 178
  Month 2: snoring | -2.31 (1.20) | -3.16 (1.14) | -4.54 (1.67)
  Month 2: quantity: number analyzed (Participants) | 359 | 388 | 177
  Month 2: quantity | 0.42 (0.06) | 0.43 (0.06) | 0.31 (0.09)
  Month 2: sleep disturbance: number analyzed (Participants) | 359 | 388 | 178
  Month 2: sleep disturbance | -14.27 (1.08) | -12.53 (1.03) | -9.97 (1.50)
  Month 2: awaken short of breath: number analyzed (Participants) | 360 | 388 | 178
  Month 2: awaken short of breath | -4.12 (1.05) | -2.15 (1.00) | -3.32 (1.46)
  Month 2: adequacy: number analyzed (Participants) | 360 | 388 | 178
  Month 2: adequacy | 9.90 (1.34) | 10.84 (1.28) | 6.24 (1.87)
  Month 3: overall sleep problem: number analyzed (Participants) | 352 | 382 | 172
  Month 3: overall sleep problem | -12.46 (0.87) | -11.16 (0.83) | -8.99 (1.22)
  Month 3: sleep problem summary: number analyzed (Participants) | 352 | 382 | 172
  Month 3: sleep problem summary | -10.98 (0.90) | -9.58 (0.86) | -7.65 (1.26)
  Month 3: somnolence: number analyzed (Participants) | 352 | 383 | 172
  Month 3: somnolence | -8.71 (0.96) | -7.35 (0.91) | -6.39 (1.34)
  Month 3: snoring: number analyzed (Participants) | 352 | 383 | 172
  Month 3: snoring | -3.36 (1.21) | -4.25 (1.15) | -3.36 (1.69)
  Month 3: quantity: number analyzed (Participants) | 352 | 383 | 171
  Month 3: quantity | 0.45 (0.06) | 0.46 (0.06) | 0.40 (0.09)
  Month 3: sleep disturbance: number analyzed (Participants) | 352 | 382 | 172
  Month 3: sleep disturbance | -15.67 (1.08) | -14.67 (1.03) | -11.90 (1.52)
  Month 3: awaken short of breath: number analyzed (Participants) | 352 | 383 | 172
  Month 3: awaken short of breath | -2.60 (1.06) | -2.48 (1.01) | -2.67 (1.48)
  Month 3: adequacy: number analyzed (Participants) | 352 | 383 | 172
  Month 3: adequacy | 13.46 (1.35) | 11.00 (1.29) | 7.14 (1.89)

84. Secondary Outcome: Change From Baseline in MOS-SS at Months 6, 12, 18, and 24
Description: as for outcome 80
Time Frame: Months 6, 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 339 | 366 | 158
units on a scale
  Month 6: overall sleep problem | -11.62 (0.88) | -12.24 (0.84) | -9.77 (1.24)
  Month 6: sleep problem summary | -10.13 (0.91) | -11.12 (0.87) | -8.64 (1.29)
  Month 6: somnolence | -8.86 (0.97) | -8.83 (0.93) | -6.60 (1.37)
  Month 6: snoring: number analyzed (Participants) | 339 | 365 | 157
  Month 6: snoring | -3.21 (1.22) | -1.11 (1.17) | -4.00 (1.74)
  Month 6: quantity: number analyzed (Participants) | 339 | 366 | 157
  Month 6: quantity | 0.47 (0.07) | 0.44 (0.06) | 0.44 (0.09)
  Month 6: sleep disturbance | -15.44 (1.10) | -15.60 (1.05) | -12.69 (1.55)
  Month 6: awaken short of breath | -2.54 (1.07) | -4.33 (1.02) | -4.23 (1.53)
  Month 6: adequacy | 10.76 (1.36) | 11.57 (1.30) | 8.41 (1.94)
  Month 12: overall sleep problem: number analyzed (Participants) | 314 | 330 | 135
  Month 12: overall sleep problem | -12.21 (0.90) | -11.94 (0.86) | -9.10 (1.30)
  Month 12: sleep problem summary: number analyzed (Participants) | 314 | 330 | 135
  Month 12: sleep problem summary | -10.61 (0.93) | -10.76 (0.90) | -7.41 (1.35)
  Month 12: somnolence: number analyzed (Participants) | 314 | 330 | 135
  Month 12: somnolence | -8.85 (0.99) | -8.24 (0.95) | -5.46 (1.44)
  Month 12: snoring: number analyzed (Participants) | 314 | 330 | 135
  Month 12: snoring | -1.44 (1.25) | 0.20 (1.20) | -1.49 (1.82)
  Month 12: quantity: number analyzed (Participants) | 314 | 329 | 134
  Month 12: quantity | 0.49 (0.07) | 0.37 (0.06) | 0.20 (0.10)
  Month 12: sleep disturbance: number analyzed (Participants) | 314 | 330 | 135
  Month 12: sleep disturbance | -15.94 (1.12) | -15.24 (1.08) | -12.00 (1.63)
  Month 12: awaken short of breath: number analyzed (Participants) | 314 | 330 | 135
  Month 12: awaken short of breath | -3.65 (1.10) | -4.04 (1.06) | -2.12 (1.62)
  Month 12: adequacy: number analyzed (Participants) | 314 | 330 | 135
  Month 12: adequacy | 11.41 (1.40) | 12.15 (1.35) | 9.30 (2.05)
  Month 18: overall sleep problem: number analyzed (Participants) | 284 | 293 | 116
  Month 18: overall sleep problem | -11.55 (0.92) | -12.82 (0.89) | -11.27 (1.36)
  Month 18: sleep problem summary: number analyzed (Participants) | 284 | 293 | 116
  Month 18: sleep problem summary | -10.02 (0.96) | -11.88 (0.93) | -9.41 (1.41)
  Month 18: somnolence: number analyzed (Participants) | 284 | 293 | 116
  Month 18: somnolence | -9.19 (1.02) | -8.70 (0.99) | -7.88 (1.51)
  Month 18:snoring: number analyzed (Participants) | 283 | 293 | 115
  Month 18:snoring | -0.45 (1.29) | -0.59 (1.25) | -3.61 (1.92)
  Month 18: quantity: number analyzed (Participants) | 284 | 293 | 115
  Month 18: quantity | 0.47 (0.07) | 0.38 (0.07) | 0.44 (0.10)
  Month 18: sleep disturbance: number analyzed (Participants) | 284 | 293 | 116
  Month 18: sleep disturbance | -14.89 (1.15) | -15.77 (1.12) | -15.97 (1.71)
  Month 18: awaken short of breath: number analyzed (Participants) | 284 | 293 | 116
  Month 18: awaken short of breath | -3.69 (1.14) | -5.50 (1.11) | -1.55 (1.71)
  Month 18: adequacy: number analyzed (Participants) | 284 | 293 | 116
  Month 18: adequacy | 10.91 (1.44) | 13.26 (1.40) | 9.71 (2.15)
  Month 24: overall sleep problem: number analyzed (Participants) | 264 | 278 | 106
  Month 24: overall sleep problem | -11.64 (0.94) | -11.93 (0.90) | -10.84 (1.39)
  Month 24: sleep problem summary: number analyzed (Participants) | 264 | 278 | 106
  Month 24: sleep problem summary | -9.83 (0.98) | -10.59 (0.94) | -9.64 (1.45)
  Month 24: somnolence: number analyzed (Participants) | 264 | 278 | 106
  Month 24: somnolence | -9.29 (1.04) | -8.63 (1.00) | -8.24 (1.55)
  Month 24: snoring: number analyzed (Participants) | 262 | 278 | 106
  Month 24: snoring | -1.00 (1.32) | -1.22 (1.27) | -3.49 (1.97)
  Month 24: quantity: number analyzed (Participants) | 264 | 278 | 104
  Month 24: quantity | 0.41 (0.07) | 0.31 (0.07) | 0.42 (0.11)
  Month 24: sleep disturbance: number analyzed (Participants) | 264 | 278 | 106
  Month 24: sleep disturbance | -14.67 (1.18) | -15.43 (1.13) | -14.20 (1.76)
  Month 24: awaken short of breath: number analyzed (Participants) | 264 | 278 | 106
  Month 24: awaken short of breath | -3.77 (1.17) | -3.16 (1.13) | -1.69 (1.77)
  Month 24: adequacy: number analyzed (Participants) | 264 | 278 | 106
  Month 24: adequacy | 11.02 (1.47) | 11.87 (1.43) | 11.35 (2.22)

85. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale
Description: FACIT-Fatigue is a 13-item questionnaire. Participant scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status
Time Frame: Baseline and Months 1, 2, 3, 6, 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 373 | 396 | 185
units on a scale
  Baseline | 28.47 (10.90) | 29.06 (10.72) | 28.55 (10.54)
  Month 1: number analyzed (Participants) | 365 | 392 | 184
  Month 1 | 34.39 (10.06) | 36.03 (10.25) | 31.70 (10.20)
  Month 2: number analyzed (Participants) | 358 | 387 | 178
  Month 2 | 36.08 (10.16) | 36.76 (10.20) | 32.83 (10.20)
  Month 3: number analyzed (Participants) | 352 | 383 | 171
  Month 3 | 36.93 (10.09) | 37.63 (10.30) | 34.09 (9.56)
  Month 6: number analyzed (Participants) | 340 | 366 | 158
  Month 6 | 37.55 (9.96) | 38.38 (9.93) | 35.38 (10.15)
  Month 12: number analyzed (Participants) | 315 | 330 | 135
  Month 12 | 37.85 (10.00) | 38.95 (9.73) | 35.99 (9.40)
  Month 18: number analyzed (Participants) | 284 | 293 | 116
  Month 18 | 38.45 (9.20) | 39.22 (9.39) | 35.97 (10.12)
  Month 24: number analyzed (Participants) | 264 | 279 | 106
  Month 24 | 38.52 (9.37) | 39.38 (9.91) | 35.16 (10.65)

86. Secondary Outcome: Change From Baseline in FACIT-Fatigue Scale
Description: as for outcome 85
Time Frame: Months 1, 2, 3, 6, 12, 18, and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 365 | 391 | 183
units on a scale
  Month 1 | 5.79 (0.47) | 7.14 (0.45) | 3.15 (0.66)
  Month 2: number analyzed (Participants) | 358 | 386 | 177
  Month 2 | 7.44 (0.48) | 7.86 (0.45) | 4.22 (0.66)
  Month 3: number analyzed (Participants) | 352 | 382 | 170
  Month 3 | 8.12 (0.48) | 8.70 (0.46) | 5.25 (0.67)
  Month 6: number analyzed (Participants) | 340 | 365 | 158
  Month 6 | 8.71 (0.48) | 9.12 (0.46) | 6.33 (0.68)
  Month 12: number analyzed (Participants) | 315 | 329 | 135
  Month 12 | 8.75 (0.49) | 9.18 (0.47) | 6.89 (0.71)
  Month 18: number analyzed (Participants) | 284 | 292 | 116
  Month 18 | 8.98 (0.50) | 9.41 (0.49) | 7.14 (0.74)
  Month 24: number analyzed (Participants) | 264 | 279 | 106
  Month 24 | 8.97 (0.51) | 9.57 (0.49) | 6.24 (0.75)

87. Secondary Outcome: Change From Baseline in Heart Rate
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: Heart rate was measured at every study visit to determine the overall health of the participants. Any abnormalities were recorded as adverse events. Change from baseline will be analyzed as part of the wider clinical program.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 362 | 390 | 182
beats per minute
  Month 1 | -1.64 (8.15) | -1.83 (8.34) | -0.73 (7.96)
  Month 2: number analyzed (Participants) | 358 | 385 | 176
  Month 2 | -1.37 (8.48) | -1.02 (9.33) | -2.19 (7.72)
  Month 3: number analyzed (Participants) | 352 | 380 | 170
  Month 3 | -1.91 (9.27) | -1.76 (9.40) | -2.37 (8.48)
  Month 6: number analyzed (Participants) | 337 | 363 | 156
  Month 6 | -1.62 (8.64) | -1.70 (9.13) | -2.24 (8.65)
  Month 9: number analyzed (Participants) | 325 | 346 | 142
  Month 9 | -1.31 (9.07) | -1.66 (9.23) | -3.50 (9.36)
  Month 12: number analyzed (Participants) | 312 | 328 | 133
  Month 12 | -2.36 (9.69) | -2.88 (9.12) | -4.08 (10.42)
  Month 15: number analyzed (Participants) | 290 | 308 | 126
  Month 15 | -1.60 (9.22) | -2.12 (10.24) | -3.78 (9.66)
  Month 18: number analyzed (Participants) | 281 | 292 | 113
  Month 18 | -2.45 (9.38) | -2.03 (8.78) | -2.23 (8.47)
  Month 21: number analyzed (Participants) | 269 | 288 | 110
  Month 21 | -1.77 (9.97) | -2.25 (8.71) | -3.34 (9.24)
  Month 24: number analyzed (Participants) | 261 | 278 | 105
  Month 24 | -3.08 (10.16) | -3.31 (9.69) | -4.26 (10.17)

88. Secondary Outcome: Change From Baseline in Temperature
Time Frame: Months 1, 2, 3, 6, 9, 12, 15, 18, 21, and 24
Population: Temperature was measured at every study visit to determine the overall health of the participants. Any abnormalities were recorded as adverse events. Change from baseline in temperature will be analyzed as part of the wider clinical program.
Measure: Mean (Standard Deviation); unit: degrees centigrade
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Number analyzed (Participants) | 362 | 390 | 181
degrees centigrade
  Month 1 | -0.07 (0.30) | -0.05 (0.31) | -0.05 (0.32)
  Month 2: number analyzed (Participants) | 358 | 385 | 175
  Month 2 | -0.07 (0.32) | -0.03 (0.37) | -0.04 (0.35)
  Month 3: number analyzed (Participants) | 352 | 379 | 169
  Month 3 | -0.08 (0.34) | -0.04 (0.34) | -0.05 (0.36)
  Month 6: number analyzed (Participants) | 337 | 363 | 155
  Month 6 | -0.07 (0.35) | -0.04 (0.36) | -0.09 (0.38)
  Month 9: number analyzed (Participants) | 325 | 347 | 141
  Month 9 | -0.07 (0.37) | -0.06 (0.39) | -0.08 (0.36)
  Month 12: number analyzed (Participants) | 312 | 328 | 132
  Month 12 | -0.10 (0.34) | -0.03 (0.39) | -0.12 (0.37)
  Month 15: number analyzed (Participants) | 290 | 308 | 125
  Month 15 | -0.08 (0.35) | -0.05 (0.42) | -0.10 (0.35)
  Month 18: number analyzed (Participants) | 280 | 292 | 112
  Month 18 | -0.07 (0.41) | -0.03 (0.42) | -0.11 (0.38)
  Month 21: number analyzed (Participants) | 269 | 286 | 108
  Month 21 | -0.09 (0.36) | -0.07 (0.40) | -0.13 (0.40)
  Month 24: number analyzed (Participants) | 261 | 278 | 104
  Month 24 | -0.10 (0.37) | -0.07 (0.40) | -0.12 (0.37)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last administration of investigational product.
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | MTX 10, 15, or 20 mg, Weekly
Serious Adverse Events (participants affected / at risk) | 40/373 | 43/397 | 22/186
Other Adverse Events (participants affected / at risk) | 252/373 | 279/397 | 122/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg BID (N=373) | CP-690,550 10 mg BID (N=397) | MTX 10, 15, or 20 mg, Weekly (N=186)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Atrioventicular block first degree (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0
Cataract (Eye disorders) | 2 | 0 | 0
Scleritis (Eye disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Colonic stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0
Salivary gland calculus (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Bone tuberculosis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Chronic hepatitis C (Infections and infestations) | 0 | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Pleural infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tonsillitis bacterial (Infections and infestations) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Varicella (Infections and infestations) | 0 | 0 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foetal exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
High grade B-cell lymphoma Burkitt-like lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 0
Demyelinating polyeuropathy (Nervous system disorders) | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Erythema annulare (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 1
Rheumatoid vasculitis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg BID (N=373) | CP-690,550 10 mg BID (N=397) | MTX 10, 15, or 20 mg, Weekly (N=186)
Anaemia (Blood and lymphatic system disorders) | 15 | 12 | 7
Abdominal pain (Gastrointestinal disorders) | 8 | 15 | 2
Abdominal pain upper (Gastrointestinal disorders) | 12 | 13 | 5
Constipation (Gastrointestinal disorders) | 7 | 9 | 7
Diarrhoea (Gastrointestinal disorders) | 15 | 24 | 15
Dyspepsia (Gastrointestinal disorders) | 13 | 18 | 9
Gastritis (Gastrointestinal disorders) | 13 | 8 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 6 | 5
Nausea (Gastrointestinal disorders) | 27 | 30 | 40
Vomiting (Gastrointestinal disorders) | 11 | 13 | 11
Asthenia (General disorders) | 1 | 7 | 5
Fatigue (General disorders) | 8 | 10 | 7
Oedema peripheral (General disorders) | 11 | 17 | 5
Pyrexia (General disorders) | 4 | 3 | 6
Bronchitis (Infections and infestations) | 20 | 27 | 4
Cystitis (Infections and infestations) | 8 | 3 | 1
Gastroenteritis (Infections and infestations) | 10 | 14 | 6
Herpes zoster (Infections and infestations) | 12 | 17 | 2
Influenza (Infections and infestations) | 10 | 11 | 3
Nasopharyngitis (Infections and infestations) | 28 | 39 | 12
Oral herpes (Infections and infestations) | 7 | 8 | 5
Pharyngitis (Infections and infestations) | 9 | 12 | 4
Respiratory tract infection viral (Infections and infestations) | 12 | 6 | 4
Sinusitis (Infections and infestations) | 9 | 9 | 5
Upper respiratory tract infection (Infections and infestations) | 30 | 36 | 15
Urinary tract infection (Infections and infestations) | 17 | 26 | 7
Alanine aminotransferase increased (Investigations) | 8 | 15 | 11
Aspartate aminotransferase increased (Investigations) | 3 | 11 | 7
Blood creatine Phosphokinase increased (Investigations) | 16 | 36 | 2
Gamma-glutamyltransferase increased (Investigations) | 8 | 14 | 2
Haemoglobin decreased (Investigations) | 5 | 3 | 4
Weight increased (Investigations) | 13 | 17 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 8 | 10 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 | 15 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 8 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 16 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 8 | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 18 | 4
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 7 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 10 | 7 | 4
Dizziness (Nervous system disorders) | 7 | 9 | 4
Headache (Nervous system disorders) | 26 | 34 | 12
Anxiety (Psychiatric disorders) | 4 | 3 | 5
Insomnia (Psychiatric disorders) | 4 | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 4
Acne (Skin and subcutaneous tissue disorders) | 8 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 8 | 5
Rash (Skin and subcutaneous tissue disorders) | 3 | 12 | 3
Hypertension (Vascular disorders) | 26 | 29 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.